

# STATISTICAL ANALYSIS PLAN ALX0061-C203

A Phase II Multicenter, Open-Label Extension Study Assessing the Long-Term Efficacy and Safety of Subcutaneous ALX-0061 in Subjects with Moderate to Severe Rheumatoid Arthritis who Have Completed One of the Preceding Phase IIb Studies with ALX-0061

Version: Final 1.0

Date: 4 OCT 2018

Protocol: 2014-003034-42

ALX0061-C203

## SIGNATURE PAGE





## TABLE OF CONTENTS

| T | ABLE O | F CONTENTS | 3 |
|----|--------|-------------------------------------------------------|----|
| LI | ST OF | ABBREVIATIONS | 6 |
| 1 | INT | RODUCTION | 9 |
| 2 | STU | JDY OBJECTIVES | 9 |
| 3 | STU | JDY DESIGN | 9 |
| | 3.1 | OVERALL STUDY DESIGN | 9 |
| | 3.2 | SAMPLE SIZE | 10 |
| | 3.3 | STUDY ENDPOINTS | 10 |
| 4 | GEI | NERAL ASPECTS FOR STATISTICAL ANALYSIS | 12 |
| | 4.1 | ANALYSIS POPULATIONS | 12 |
| | 4.1.1 | All screened population | 12 |
| | 4.1.2 | 2 Intent-to-observe (ITO) population | 12 |
| | 4.1.3 | Safety population | 12 |
| | 4.1.4 | PK population | 12 |
| | 4.2 | KEY DEFINITIONS AND LABELS | 12 |
| | 4.2.1 | Definition of baseline and change from baseline | 12 |
| | 4.2.2 | Presentation of treatment groups | 13 |
| | 4.2.3 | 3 Totals over groups | 13 |
| | 4.2.4 | General presentation of results | 13 |
| | 4.2.5 | 5 Visit Windows | 13 |
| | 4.3 | GENERAL METHODS | 13 |
| | 4.3.1 | • | |
| | 4.3.2 | 2 Handling of values below (or above) a threshold | 14 |
| | 4.3.3 | B Handling of outliers | 14 |
| | 4.4 | SOFTWARE AND VALIDATION MODEL | 14 |
| 5 | GEI | NERAL CHARACTERISTICS | 15 |
| | 5.1 | SUBJECT DISPOSITION | 15 |
| | 5.2 | PROTOCOL DEVIATIONS AND ELIGIBILITY CRITERIA | 15 |
| | 5.3 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 16 |
| | 5.4 | EXPOSURE TO STUDY MEDICATION AND TREATMENT COMPLIANCE | |
| | 5.5 | MEDICAL HISTORY | 18 |
| | 5.6 | CONCOMITANT THERAPIES | 18 |
| 6 | EFF | ICACY | 19 |
| | 6.1 | MAIN EFFICACY ANALYSIS | 19 |
| | 6.2 | OTHER EFFICACY ANALYSES | 20 |
| 7 | SAF | FETY | 20 |
| | 7.1 | ADVERSE EVENTS | 20 |



| • | 7.2 | LABORATORY EVALUATIONS | 23 |
|---|---|---|---|
| | 7.3 | PHYSICAL EXAMINATION | 24 |
| | 7.4 | VITAL SIGNS | 24 |
| 8 | ANA | ALYSIS OF PHARMACOKINETICS | 24 |
| 9 | ANA | ALYSIS OF IMMUNOGENICITY | 25 |
| 9 | 9.1 | AVAILABLE PARAMETERS | 25 |
| | 9.2 | MISSING RESULTS AND DATA IMPUTATION | 27 |
| | 9.3 | SUBJECT CLASSIFICATIONS (DERIVED PARAMETERS) | 27 |
| | 9.3.1 | ADA subject classification | 27 |
| | 9.3.2 | 2 mADA subject classification | 28 |
| | 9.3.3 | 3 Overall subject classification | 29 |
| | 9.3.4 | NAb subject class | 30 |
| | 9.4 | PRE-AB PREVALENCE AND TE ADA INCIDENCE CALCULATIONS. | 30 |
| | 9.4.1 | Incidence of ADA and derived sets | 30 |
| | 9.4.2 | 2 Incidence of mADA subject classes and derived sets | 31 |
| | 9.4.3 | Incidence of overall subject classification (ADA, mADA results) and derived sets | 31 |
| | 9.4.4 | Incidence of NAb subject classes and derived sets | 32 |
| | 9.4.5 | 5 Safety subgroup analysis | 32 |
| | 9.4.6 | S ADA and NAb incidence over time | 33 |
| 10 | INT | ERIM ANALYSES | 33 |
| 11 | CHA | ANGE FROM ANALYSIS PLANNED IN PROTOCOL | 33 |
| 12 | COI | NVENTIONS | 33 |
| | 12.1 | ANALYSIS PHASES AND VISIT WINDOWS | 33 |
| | 12.1 | .1 Algorithm of allocating visits to time windows | 33 |
| | 12.1 | 2 Selection of visits | 34 |
| | 12.2 | GENERAL CHARACTERISTICS | 35 |
| | 12.2 | .1 Derivation of exposure parameters | 35 |
| | 12.3 | EFFICACY | 35 |
| | 12.4 | SAFETY | 38 |
| | 12.4 | .1 Adverse events | 38 |
| | 12.4 | 2 Laboratory | 39 |
| 13 | IND | EX OF TABLES | 39 |
| | 13.1 | GENERAL | 39 |
| | 13.2 | EFFICACY | 41 |
| | 13.3 | PHARMACOKINETICS | 47 |
| | 13.4 | SAFETY | 47 |
| | 13.5 | IMMUNOGENICITY | 50 |
| 14 | IND | EX OF FIGURES | 51 |
| 15 | | EX OF LISTINGS | |
| AL | X0061 | -C203 – Statistical Analysis Plan – Final 1.0 – 4 OCT 2018 Page | e 4/111 |



| 15.1 | GENERAL | 54 |
|---|---|---|
| 15.2 | Efficacy | 55 |
| 15.3 | PHARMACOKINETICS | 56 |
| 15.4 | SAFETY | 57 |
| 15.5 | IMMUNOGENICITY | 59 |
| 16 AP | PENDICES | 60 |
| 16.1 | APPENDIX 1: SCHEDULE OF ASSESSMENTS | 60 |
| 16.2 | APPENDIX 2: PREDNISOLONE EQUIVALENT DOSE CHART | 64 |
| 16.3 | APPENDIX 3: CTCAE GRADES (VERSION 4.03 14JUN2010) | 65 |
| 16.4 | APPENDIX 4: FACIT-F SCORING GUIDELINES (VERSION 4) | 68 |
| 16.5 | APPENDIX 5: SEARCH CRITERIA FOR ADVERSE EVENTS OF SPECIAL INTEREST | 72 |
| 16.6 | APPENDIX 6: SF-36 QUESTIONNAIRE VERSION 2 | 106 |



## LIST OF ABBREVIATIONS

ADaM Analysis data model

ACR American college of rheumatology

ADA Anti-drug antibody

AE Adverse event

AIDS Acquired immune deficiency syndrome

ALP Alkaline phosphatase
ALT Alanine transaminase
ANCOVA Analysis of covariance
AST Aspartate transaminase

CI Confidence interval

CDAI Clinical disease activity index

CRF Case report form CRP C-reactive protein

CTCAE Common terminology criteria for adverse events

CV Coefficient of variation

CXCL Chemokine (C-X-C motif) ligand

DAS28 Disease activity score using 28 joint counts

DBP Diastolic blood pressure

DSMB Data safety monitoring board

DT Drug Tolerance (immunogenicity assay characteristic)

DY Relative day

ESR Erythrocyte sedimentation rate

EULAR European league against rheumatism

FACIT Functional assessment of chronic illness therapy

GGT Gamma-glutamyl transferase

HAQ-DI Health assessment questionnaire – disability index

ICF Informed consent form

ICH International Council for Harmonisation

IGRA Interferon-gamma release assay

IL-6 Interleukin-6

ITO Intent-to-observe



IWRS Interactive web response system

LDA Low disease activity

LDH Lactate dehydrogenase

LOCF Last observation carried forward

LS Least squares

MedDRA Medical Dictionary for Regulatory Activities

MMP Matrix metalloproteinase

MTX Methotrexate NA Not Analyzed

NAb Neutralizing antibody

NR No Result

NRI Non-responder imputation

OC Observed cases

OLE Open-label extension

PD Pharmacodynamic

PK Pharmacokinetic

q2w Every two weeks

q4w Every four weeks

RA Rheumatoid arthritis

SAP Statistical analysis plan

SBP Systolic blood pressure

s.c. Subcutaneously

SD Standard deviation

SDAI Simplified disease activity index

SDTM Study data tabulation model

SE Standard error

SF-36 Short form (36) health form

SGS-LS SGS-Life Sciences – Clinical Research

SOP Standard operating procedure

STAT Statistics

SJC Swollen joint count

TB Tuberculosis

TEAE Treatment-emergent adverse event



TJC Tender joint count

VAS Visual analogue scale

WHO World Health Organisation



#### 1 INTRODUCTION

ALX-0061 (vobarilizumab) has been developed by the sponsor as a new therapeutic protein neutralizing pro-inflammatory activity in the interleukin-6 (IL-6) pathway. ALX-0061 is a therapeutic protein called nanobody which inhibits the interaction between the IL-6 ligand and the receptor subunit, thereby preventing receptor signaling hence pro-inflammatory activity of IL-6. The investigator's brochure contains more detailed background information. This clinical study (ALX0061-C203) is an open-label extension of Phase IIb studies ALX0061-C201 and ALX0061-C202 and is intended to evaluate the long-term efficacy and safety of ALX-0061 administered subcutaneously (s.c.) to subjects with active rheumatoid arthritis (RA), a chronic systemic inflammatory autoimmune disease.

This statistical analysis plan (SAP) describes the final statistical analysis to be performed for the ALX0061-C203 study. This SAP covers the efficacy, safety, pharmacokinetic, and general characteristics parts of the statistical analysis. It specifies the analysis displays to be presented and describes the methods and procedures in a more elaborated way than in the statistical methods section of the protocol. The statistical analysis will process and present the results following the International Council for Harmonisation (ICH) standards, in particular the ICH-E3, ICH-E6, and ICH-E9 guidelines.

## 2 STUDY OBJECTIVES

The objective of this study is to evaluate the long-term efficacy and safety of ALX-0061 administered s.c. to subjects with active RA.

## 3 STUDY DESIGN

## 3.1 Overall Study Design

This is a multicenter, open-label extension (OLE) phase II study of ALX-0061 administered s.c.in subjects with active RA who have completed the ALX-0061 treatment and assessment period of one of the preceding Phase IIb studies with ALX-0061 (C201 or C202) and who achieved at least 20% improvement in swollen joint count (SJC) and/or tender joint count (TJC) (66/68 counts) compared to baseline at the final visit of the preceding study and for the countries where there was approval for the study.

Eligible subjects will receive ALX-0061 150 mg s.c. injections, beginning at Day 1 (Week 0) of the OLE and every 2 weeks (q2w) thereafter up to and including Week 102. Eligible subjects from study ALX0061-C201 will also continue their methotrexate (MTX) treatment. Subjects will return for 12 ambulatory visits planned at Day 1 (Week 0), and Weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96 and 104. Subjects who received study drug up to and including Week 102, should return for the End of Treatment Visit at Week 104 and for the Follow-up Visit 12 weeks after the last study drug administration at Week 102.

In the current OLE study, maintenance of the response will be reassessed at the study visits every 12 weeks from Week 12 until Week 96. Subjects who fail to maintain response and meet efficacy discontinuation criteria (< 20% improvement in both SJC and TJC



compared to baseline of the preceding Phase IIb study) will be discontinued from the study.

The schedule of assessments can be found in Appendix 1: Schedule of assessments. As this is an OLE study, blinding is not required.

## 3.2 Sample Size

This is an extension study and is not set by statistical power. Subjects who have completed the Week 24 (study ALX0061-C201) or Week 12 (study ALX0061-C202) assessment visit in one of the preceding Phase IIb studies with ALX-0061, and who are qualified for this study per inclusion/exclusion criteria, will be invited to participate in the extension study. Up to a maximum of approximately 501 subjects are planned to participate in this OLE study.

## 3.3 Study Endpoints

The protocol does not define primary or secondary study endpoints. The following endpoints will be analyzed:

## **Efficacy endpoints:**

- American College of Rheumatology (ACR) ACR20, ACR50, and ACR70 response rate over time (Week 0, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96 and Week 104).
- Actual values in ACR-N index improvement over time (Week 0, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96 and Week 104).
- Actual values and change from baseline values in Disease Activity Score using 28 joint counts (DAS28) using CRP and ESR, simplified disease activity index (SDAI) and clinical disease activity index (CDAI) over time (Week 0, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96 and Week 104).
- Disease activity: response rate of remission and response rate of low disease activity (LDA) based on DAS28(ESR), SDAI, CDAI, Boolean (only remission) over time (Week 0, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96 and Week 104).
- Disease activity: response rate of DAS28(CRP) < 2.6 and response rate of low disease activity (LDA) based on DAS28(CRP) over time (Week 0, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96 and Week 104).
- Disease activity: rate of maintained remission at consecutive time points based on DAS28(ESR), SDAI, CDAI, Boolean and rate of maintained LDA at consecutive time points based on DAS28(ESR) over time (Week 0, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96 and Week 104).
- Disease activity: rate of maintained DAS28(CRP) < 2.6 at consecutive time points and rate of maintained LDA at consecutive time points based on DAS28(CRP) over time (Week 0, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96 and Week 104).



- European league against rheumatism (EULAR) DAS28 response rate (good, moderate, or no response) over time (Week 0, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96 and Week 104).
- Actual values and change from baseline values in HAQ-DI over time (Week 0, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96 and Week 104).
- HAQ-DI response rate (i.e., those who have a clinically meaningful improvement from baseline of ≥ 0.25 in HAQ-DI) and HAQ-DI normal physical function response rate (i.e., those who have a score of ≤ 0.5) over time (Week 0, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96 and Week 104).
- Actual values and change from baseline values in Physical and mental component scores of SF-36 over time (Week 0, Week 24, Week 48, Week 72 and Week 104).
- Actual values and change from baseline values in FACIT-Fatigue over time (Week 0, Week 24, Week 48, Week 72 and Week 104).
- Actual values and change from baseline values in duration of morning stiffness at Week 0 and Week 104.

#### Pharmacokinetic (PK) endpoints:

ALX-0061 serum concentration over time (Week 0, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96 and Week 104).

## Immunogenicity endpoints:

- Overall subject classification based on ADA/mADA assays results.
- Overall subject classification based on NAb assay results.

## Safety endpoints:

- Number of events as well as number and percentage of subjects with treatmentemergent Adverse Events (TEAEs), treatment-related AEs, Serious Adverse Events (SAEs), non-serious AEs, treatment-related SAEs, SAEs leading to treatment discontinuation and Adverse Events of Special Interest (AESI), categorized by System Organ Class (SOC) and Preferred Term (PT) and Maximum Severity (where applicable). Note that all adverse events reported in this study are considered treatment-emergent.
- Actual values and change from baseline in clinical laboratory parameters, including blood chemistry, hematology, urinalysis, coagulation and the acute phase proteins (CRP, ESR, and fibrinogen) at Week 0, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96, Week 104 and Followup (Week 0, Week 24, Week 48, Week 72 and Week 104 only for extended clinical laboratory analyses).
- Shift from baseline in clinical laboratory parameters with normal ranges or CTCAE grades at Week 0, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96, Week 104 and Follow-up.
- Actual values and change from baseline values in vital signs measurements at Week 0, Week 4, Week 8, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96, Week 104 and Follow-up.
- Physical examination abnormal findings at Week 0, Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96, Week 104 and Follow-up.



## 4 GENERAL ASPECTS FOR STATISTICAL ANALYSIS

## 4.1 Analysis Populations

The following populations will be considered for analysis:

## 4.1.1 All screened population

The all screened population includes all subjects who signed an informed consent for participation in the ALX0061-C203 study.

## 4.1.2 Intent-to-observe (ITO) population

The ITO population includes all subjects who enrolled in study ALX0061-C203 and is thus equal to the all screened population. General characteristics and efficacy will be analyzed on the ITO population.

## 4.1.3 Safety population

The safety population includes all subjects who received at least 1 administration of study drug, as treated. The safety population will be used for the analysis of exposure and safety data.

## 4.1.4 PK population

The PK population is a subset of the safety population and consists of all subjects who received at least 1 administration of ALX-0061 and for whom at least one ALX-0061 serum concentration has been determined.

The PK population will be used for the analysis of ALX-0061 serum concentrations.

## 4.2 Key Definitions and Labels

## 4.2.1 Definition of baseline and change from baseline

The baseline value will be the baseline value of the parent study.

The absolute change from baseline will be calculated for all post-baseline time points as: Change from baseline at time point t = value at time point t – baseline value

For selected efficacy endpoints, the percentage change from baseline will be calculated for all post-baseline time points as: Percentage change from baseline at time point t=100 \* (value at time point t — baseline value) / baseline value. As percentage change can not be calculated for subjects with a baseline value of 0, these subjects will not be included for the corresponding summary analysis (if planned) and the respective column(s) will be kept blank for the corresponding listing.

For the changes from baseline, only subjects with both a baseline value and a value at the post-baseline time point will be included.



Wherever in the document 'change from baseline' is mentioned, it concerns the absolute change from baseline.

## 4.2.2 Presentation of treatment groups

The following treatment group labels will be used in the tables, listings and figures, unless specified otherwise:

- ALX-0061 150 mg q2w + MTX (C201 PBO + MTX)
- ALX-0061 150 mg q2w + MTX (C201 75 mg q4w + MTX)
- ALX-0061 150 mg q2w + MTX (C201 150 mg q4w + MTX)
- ALX-0061 150 mg q2w + MTX (C201 150 mg q2w + MTX)
- ALX-0061 150 mg q2w + MTX (C201 225 mg q2w + MTX)
- ALX-0061 150 mg q2w + MTX (C201 all subjects)
- ALX-0061 150 mg q2w (C202 150 mg q4w)
- ALX-0061 150 mg q2w (C202 150 mg q2w)
- ALX-0061 150 mg q2w (C202 225 mg q2w)
- ALX-0061 150 mg q2w (C202 all subjects)
- All subjects

## 4.2.3 Totals over groups

Grand total, pooling all subjects, will be displayed in all tables.

## 4.2.4 General presentation of results

All results will be presented per treatment group, unless specified otherwise. All listings will be ordered by treatment group, subject, and time point, unless specified otherwise.

The analysis population will always be indicated in a subtitle in the table, listing or figure.

#### 4.2.5 Visit Windows

The visit windows as defined in Section 12.1 will be applied to all parameters.

#### 4.3 General Methods

#### 4.3.1 Calculation of descriptive statistics

Continuous variables will be summarized using descriptive statistics including the number of non-missing observations (n), the arithmetic mean, the standard deviation (SD) for general characteristics and for PK summaries or standard error (SE) for efficacy, safety and immunogenicity, the median, minimum and maximum.

Descriptive statistics of efficacy will additionally include a 95% confidence interval (CI) of the mean, calculated based on the large sample normal approximation. For changes from



baseline of efficacy parameters, the least squares (LS) mean and 95% CI derived from an ANCOVA model with treatment group as factor and baseline as covariate will be shown.

Descriptive statistics of PK concentrations will additionally include 5% and 95% percentiles, coefficient of variation (CV)% of arithmetic mean, geometric mean and geometric SD.

Descriptive statistics of continuous variables will be presented when n≥2. When n=1, only sample size (n) and mean are shown.

Categorical variables will be summarized using frequency counts and percentages. For efficacy, a Wilson score 95% CI on the percentage in each treatment group will also be shown. When count data are presented, the percentage will be suppressed when the count is zero. Missing values will not be included in the denominator count when computing percentages. For demographics and baseline disease characteristics a 'missing' row will be included to indicate the number of missing values, without percentages.

For the graphs showing mean values of continuous variables, an SE flag will be shown, while for graphs showing percentages, this will be the Wilson score asymptotic SE on the binomial proportions.

Calculated parameters will not be rounded in the derived datasets. The rounding will be done at the reporting level. Mean, median, 95% CI limits will be presented with one decimal more than data collected. Minimum and maximum will be reported with the same precision as data collected and SD and SE with two decimals more than data collected. Percentages will be tabulated with 1 decimal.

## 4.3.2 Handling of values below (or above) a threshold

Values below (above) the detection limit will be imputed by the value of the detection limit itself, unless indicated otherwise. Listings will always present the original value. Example: if the database contains values like "<0.04", then for the descriptive statistics the value of the detection limit (0.04) shall be used. A value like ">1000" will be imputed by "1000".

Individual pharmacokinetic concentrations below the limit of detection or below the quantification limit (BQL) will be reported as BQL. To compute descriptive statistics (i.e. mean (or median or geomean), SD, CV%, minimum and maximum), all BQL values will be treated as missing. When the total number of BQL values exceeds 1/3 of the total number of values at that time point, descriptive statistics will not be computed. Descriptive statistics not calculated for the above reasons will be reported as not calculated (NC).

For handling of titer values from immunogenicity analysis, see section 9.

## 4.3.3 Handling of outliers

There will be no outlier detection. All measured values will be included in the analyses.

## 4.4 Software and Validation Model

SAS version 9.4 or higher will be used for programming.

Currently valid standard operating procedures (SOPs) will be followed.

ALX0061-C203 – Statistical Analysis Plan – Final 1.0 – 4 OCT 2018



ACR20 response will be validated following Model C, other efficacy endpoints, general and safety parts following validation model B:

Model B: review of the output, source code and program log by an independent person (i.e., somebody different from the developer).

Model C: review of the output, source code and program log by an independent person, plus independent programming of the parameters indicated in this SAP.

## 5 GENERAL CHARACTERISTICS

All analyses on general characteristics will be run on the ITO population, unless specified otherwise.

## 5.1 Subject Disposition

Subject disposition will be presented descriptively for the all screened population. This includes the number and percentage of subjects in each of the analysis populations defined in section 4.1. Percentages will be calculated relative to the all screening population. A disposition summary by region and country and a summary by time point will be given for the ITO population. The number and percentage of subjects who completed the study and those who prematurely discontinued from the study will be summarized, along with the primary reasons for discontinuation.

A detailed list of tables and listings can be found in section 13.1 and section 15.1, respectively.

## 5.2 Protocol Deviations and Eligibility Criteria

A protocol deviation is any change, divergence, or departure from the study design or procedures defined in the protocol. Protocol deviations are considered as major if they concern criteria and disease characteristics that are critical to define the study population and criteria that determine or influence clinical endpoints or criteria that may cause immediate hazard to the subjects (impact on subjects' rights, safety or well-being) or increase the safety risk to subjects.

The list of (potentially) major protocol deviations will be reviewed by the sponsor and finalized prior to database lock. Detailed information can be found in the trial protocol deviation criteria list.



Major protocol deviations will be tabulated according to their category. The following categories are considered:

- Selection criteria not met
- Subject not withdrawn as per protocol
- Prohibited concomitant medication
- Treatment non-compliance
- Safety assessment deviation
- Efficacy assessment deviation
- Other

Additionally, major protocol deviations will be listed including categorization and description.

A detailed list of tables and listings can be found in section 13.1 and section 15.1, respectively.

## 5.3 Demographic and Other Baseline Characteristics

Demographic data and baseline disease characteristics will be summarized descriptively by treatment group and overall on the ITO population. The following demographic parameters and baseline disease characteristics will be included in the tables and/or listings:

## **Demographic parameters:**

- Sex at birth (male, female)
- Women of childbearing potential (yes, no), only listed
- Age (years): the age at baseline of the parent trial is used.
- Age categories (<65 years, ≥65 years)</li>
- Year of birth: only listed
- Date of signing the ICF: only listed
- Race (white, black or African American, Asian, American Indian or Alaska native, native Hawaiian or other Pacific islander, other, not allowed to ask). Specification for Asian and other race will only be listed.
- Ethnicity (Hispanic or Latino, non-Hispanic or non-Latino, not allowed to ask)
- Geographic region (Latin America, Europe):
  - o Latin America: Mexico
  - Europe: Spain, Germany, Poland, Belgium, Bulgaria, Republic of Moldova, Georgia, Hungary, Romania, Macedonia and Serbia
- Height (cm)
- Weight (kg)
- Weight categories (≤100 kg, >100 kg; ≤median, >median)
- Body mass index BMI = (weight in kg) / (height in m)<sup>2</sup> (kg/m<sup>2</sup>)

Age, height, weight and their derived parameters will be extracted from the parent study. Previously calculated parameters will not be recalculated.



#### Baseline disease characteristics:

Please refer to the efficacy section 12.3 for detailed definitions of the parameters. Below baseline parameters will be extracted from the parent study and calculated parameters will not be recalculated.

- Swollen joint count (SJC66): number of swollen joints out of 66 assessed joints
- Tender joint count (TJC68): number of tender joints out of 68 assessed joints
- Swollen joint count (SJC28): number of swollen joints out of 28 assessed joints used for DAS28 calculation
- Tender joint count (TJC28): number of tender joints out of 28 assessed joints used for DAS28 calculation
- Tender joint count categories (<10, 10-20, >20)
- Swollen joint count categories (<7, 7-11, >11)
- CRP (mg/dL)
- CRP categories (<= upper limit of normal range [ULN], >ULN and <=1.2xULN, >1.2xULN and <=3xULN, >3xULN)
- ESR (mm/h)
- Physician's global assessment of the disease (VAS; 0-100 mm)
- Patient's global assessment of the disease (VAS; 0-100 mm)
- Patient's assessment of pain (VAS; 0-100 mm)
- HAQ-DI (0-3)
- SF-36 Physical component summary
- SF-36 Mental component summary
- Time since first RA symptoms (years)
- Time since RA diagnosis (years)
- ACR functional class at screening (of parent trial): class I / class II / class III / class IV
- Extra-articular symptom location: any of the following: skin, eyes, gastrointestinal, heart, lung, renal, nervous system, other
- Extra-articular symptoms: only listed
- Rheumatoid factor (RF) concentration (kIU/L)
- RF category (positive [>ULN], negative [<=ULN])</li>
- Anti-CCP category (positive [>ULN], negative [<=ULN])</li>
- Combined RF and anti-CCP category (double positive, double negative, mixed negative and positive)
- DAS28 Score (ESR)
- DAS28 Score (CRP)
- DAS28(ESR) and DAS28(CRP) categories (<=3.2, >3.2 and <=5.1, >5.1)
- Clinical Disease Activity Index (CDAI)
- Simplified Disease Activity Index (SDAI)
- MTX use (dose)



- Corticosteroid use (prednisone equivalent dose)
- Duration of morning stiffness (minutes)
- FACIT

A detailed list of tables and listings can be found in section 13.1 and section 15.1, respectively.

## 5.4 Exposure to Study Medication and Treatment Compliance

Extent of exposure will be analyzed descriptively by treatment group and overall based on the safety population. Note that only exposure during the OLE will be analyzed, so this will not reflect the total exposure of a subject to ALX-0061.

The following parameters will be summarized: total treatment duration, total number of study drug doses received, cumulative dose of study drug received, compliance and home administration. The derivation of these parameters can be found in section 12.2.1. A detailed list of tables and listings can be found in section 13.1 and section 15.1, respectively.

## 5.5 Medical history

Medical history was listed in the parent trials.

## 5.6 Concomitant Therapies

Any concomitant therapy taken during the study will be recorded in the eCRF, including ongoing concomitant therapies from the parent trial. Concomitant therapies are defined as therapies with a stop date on or after date of first dose of study drug in the C203 study. Therapies stopped before the study are not recorded. Analysis of prior medications is available in the parent trials.

All therapies are coded using the latest WHO-DRUG version. No anatomical therapeutic chemical classification system (ATC) selection is performed.

Concomitant therapies will be tabulated by generic term, for RA and non-RA medications separately, by treatment group and overall using the ITO population. Multiple records of the same generic term for the same subject will be counted only once. The table will therefore present subjects, not occurrences. The tables are sorted by decreasing frequency based on all subjects.

Systemic corticosteroids are selected as steroid RA-therapy with intravenous or intramuscular administration (not intra articular)

A detailed list of tables and listings can be found in section 13.1 and section 15.1, respectively.



## 6 EFFICACY

## 6.1 Main Efficacy Analysis

No inferential statistical analyses will be performed. All tables will be presented by treatment group and overall, including treatment groups defined by previous dosing regimen of the parent trial (cfr. section 4.2.2). All analyses will be run on the ITO. The main analysis will be on observed cases (OC).

Continuous efficacy endpoints will be summarized as follows:

- Actual values: descriptive statistics (mean, 95% CI on the mean [normal approximation], SE, median, minimum, and maximum) per endpoint and time point. The baseline value from the parent trial will be included to the summary, if applicable.
- Changes from baseline: baseline adjusted LS means and 95% CI from an ANCOVA model with treatment as factor and baseline as covariate, median, minimum and maximum per endpoint and post-baseline time point.

This will be done for the following parameters: ACR-N, DAS28(CRP), DAS28(ESR), SDAI, CDAI, HAQ-DI, SF-36 physical and mental component scores, FACIT-Fatigue, duration of morning stiffness, patient's assessment of pain (VAS-scale), patient's global assessment of disease activity (VAS-scale), physician's global assessment of disease activity (VAS-scale), CRP, ESR, TJC68, TJC28, SJC68, SJC28, MTX dose, corticosteroids dose. Different types of sytemic corticosteroids will be converted to Prednisolone equivalent doses before calculating the cumulative dose of corticosteroids. The cumulative dose will be given in mg/day (Please refer to Appendix 2 section 16.2 for more details).

Categorical efficacy endpoints will be presented using a frequency tabulation of the parameter at each time point, including a Wilson score 95% CI on the percentage of subjects in the category of interest. The baseline value from the parent trial will be included to the summary, if applicable. This wil be done for the following parameters: ACR20, ACR50, ACR70, EULAR response (including EULAR good response), DAS28(ESR) low disease activity / remission / maintained low disease activity, DAS28(CRP) low disease activity / DAS(CRP) < 2.6 / maintained DAS(CRP) < 2.6 / maintained low disease activity, SDAI low disease activity / remission / maintained remission, CDAI low disease activity / remission / maintained remission, Boolean remission / maintained remission, HAQ-DI clinically meaningful improvement, HAQ-DI normal physical function, MTX dose reduction rate, MTX discontinuation rate.

All 95% Cls will be two-sided.

In addition, line plots of the mean actual values per time point, including SE bars, for continuous endpoints, and line plots of the response rates (in percentage) per time point, including SE bars, for categorical endpoints, will be provided.

Definitions and calculation of efficacy parameters are detailed in section 12.3.

A detailed list of tables, figures and listings can be found in section 13.2, section 14 and section 15.2, respectively.



## 6.2 Other Efficacy Analyses

The sensitivity of results to missing data will be assessed by conducting a sensitivity analysis using LOCF imputed cases. Missing post-baseline values are imputed by the last non-missing preceding post-baseline value. Baseline itself is not imputed.

The sensitivity analysis will be done for the following efficacy endpoints:

- ACR20/50/70
- DAS28(ESR) actual values and changes from baseline
- DAS28(ESR) remission/low disease activity
- DAS28(CRP) actual values and changes from baseline
- DAS28(CRP) < 2.6/low disease activity

A second sensitivity analysis will be done using NRI imputed cases. Missing post-baseline ACR values are imputed with the value corresponding to that of non-responders.

This sensitivity analysis will be done for the following efficacy endpoints:

- ACR20/50/70
- DAS28(ESR) remission/low disease activity
- DAS28(CRP) < 2.6/low disease activity

In addition, for the same efficacy endpoints, a subgroup analysis will be conducted on the observed cases.

The following subgroups will be considered:

- Age category (<65 yrs at baseline, >= 65 yrs at baseline)
- Geographic region
- If any subcategory has less than 10% of the total number of patients then the subgroup analysis will not be produced.

A detailed list of tables can be found in section 13.2.

#### 7 SAFETY

#### 7.1 Adverse Events

All safety summaries will be based on the safety population and presented by treatment group (see section 4.2.2). As study drug treatment is not interrupted between the parent study and this study, all adverse events reported in this study are considered treatment-emergent. However, unless specified otherwise, only adverse events that started after the first dose of C203 will be considered in the tables.

All adverse events will be coded and classified by System Organ Class (SOC) and Preferred Term (PT) using the medical dictionary for regulatory activity (MedDRA) that is current at the time of database lock.

A TEAE will be categorized as study drug-related if the relationship to study drug is reported to be 'possibly related' or 'related', or missing. In tabulations this categorization

## Ablynx


will be used, but in the listings the original reported relationship will be presented. If the relationship is reported to be 'not applicable', it will not be considered in the tabulations.

A TEAE is reported as related to study procedure or not related to study procedure. Missing study procedure relationship will be considered as related.

A general summary table with AE events starting after first dose of C203 only will be produced to report the number and percentage of subjects with at least one event, the number of events and the incidence per 100 patient years, which will be calculated as: 100 x (Number of subjects with AE)/(Total number of years observed while on C203, summed for all subjects). Percentages will be calculated out of the number of subjects in the relevant treatment group.

The following categories will be included in the summary table:

- TEAE
- serious TEAE
- TEAE leading to death
- severe TEAE as classified by the investigator
- TEAE for which the study drug was interrupted
- TEAE for which the study drug was discontinued
- study drug-related TEAE
- serious study drug-related TEAE
- injection-site reaction.

Note that the TEAE here refers to the AEs starting after first dose of study drug in C203 study.

A similar summary table will be produced for all TEAEs including those of the parent trials (C201 and C202). Any event happening either on parent trial or on the current trial will be considererd for deriving the number and percentage of subjects with at least one event, and the number of events. The incidence per 100 patient years will be calculated as: 100 x (Number of subjects with AE)/(Total number of years observed starting from the first dose in parent trial, summed for all subjects).

Another summary table will be presented selecting adverse events of special interest. Search criteria for these adverse events can be found in section 16.5.



The following categories will be included in the summary table:

- infection
- serious infection (requiring hospitalization or i.v. antimicrobial treatment)
- opportunistic infection, excluding TB
- active TB infection
- latent TB infection
- Herpes zoster infection
- malignancy
- hypersensitivity reaction (including anaphylaxis and angioedema)
- hypersensitivity reaction (including anaphylaxis and angioedema) leading to withdrawal
- GI perforation
- demyelinating disorder
- MACE

This table will represent events which occurs only after the first dose of study drug in C203 study.

One more summary table for AEs of special interest will be produced including events from the parent trials as well. Any event happening either on parent trial or on the current trial will be considererd for deriving the number and percentage of subjects with at least one event, and the number of events. The incidence per 100 patient years will be calculated as: 100 x (Number of AEs)/(Total number of years observed starting from the first dose in parent trial, summed for all subjects).

Tables by SOC and PT will report the number and percentage of subjects with at least one event, occurring only after the first dose of study drug on C203 study. Percentages will be calculated out of the number of subjects in the relevant treatment group.

These tables will be prepared for the following selections of AEs:

- TEAEs
- TEAEs by severity (Mild, Moderate, Severe)
- TEAEs with an incidence of at least 3%
- serious TEAEs
- non-serious TEAEs
- study drug-related TEAEs
- study procedure-related TEAEs
- TEAE for which the study or the study drug were discontinued

The tables by SOC and PT will be sorted in descending order starting from the SOC with the highest incidence in the all subjects group. If the total incidence for any two or more SOCs is equal, the SOCs will be presented in alphabetical order. Within each SOC, the PTs will be presented in the same manner as the SOCs. At each level of subject summarization, a subject is counted once if the subject reported one or more events. In the summary table by severity, if a subject reported multiple occurences of the same TEAE, only the most severe will be presented. TEAEs with missing severity will be presented in a separate 'Missing' category.



The AE onset day and the AE duration will not be presented in the tabulations, but will be listed. Their derivation is provided in section 12.4.1.

A detailed list of tables and listings can be found in section 13.4 and section 15.4, respectively.

## 7.2 Laboratory Evaluations

The following laboratory parameters will be summarized and displayed at the scheduled time points:

- Biochemistry: total bilirubin, alkaline phosphatase, gamma-glutamyltransferase, AST, ALT, lactate dehydrogenase, creatinine, urea, total protein, albumin, glucose, inorganic phosphate, sodium, potassium, calcium, and chloride. In the extended clinical laboratory analysis, fasting serum lipids will be included as well (i.e. total cholesterol, HDL-cholesterol, LDL-cholesterol, LDL/HDL cholesterol ratio (calculated as LDL/HDL) and triglycerides)
- **Hematology**: leukocytes, erythrocytes, hemoglobin, hematocrit, thrombocytes, partial automated differentiation (lymphocytes, monocytes, eosinophils, basophils, neutrophils and neutrophils segmented), mean corpuscular volume, mean corpuscular hemoglobin, and mean corpuscular hemoglobin concentration.
- Acute phase proteins: fibrinogen, CRP, and ESR.
- **Urinalysis**: erythrocytes/blood, urobilinogen, ketones, glucose, protein, pH, and leukocytes.
- **Coagulation**: activated partial prothrombin time, prothrombin time, and INR (the latter for subjects on warfarin only).

For lab tests with numeric values, tables showing descriptive statistics (mean, median, standard error, minimum, and maximum) per lab test category (hematology, biochemistry, acute phase proteins, urinalysis, coagulation), lab test and unit and time point by treatment group and using the safety population will be prepared for:

- actual values
- absolute changes from baseline (definition in section 4.2.1)

Urinalysis results will be presented in a frequency table per lab test and time point.

The statistical summary will only present results in Standard International (SI) units. Other units will not be presented. In the tables, the number of significant digits of the original values will be used to determine the number of decimals that will be printed.

All values will be compared to their matching normal ranges (low, normal, high). For both values and normal ranges the SI units will be considered to determine abnormalities. Additionally, for key hematology and biochemistry parameters, toxicities will be derived according to the common terminology criteria for adverse events (CTCAE, see appendix 16.2) grading, version 4.03 (ALT, AST, total bilirubin, gamma-glutamyltransferase, leukocytes, neutrophils, thrombocytes, fibrinogen and cholesterol). Details for derivation of classification based on normal ranges of laboratory parameters can be found in section 12.4.2.



Cross-tabulations per lab test category (hematology, biochemistry, acute phase proteins, urinalysis, coagulation), lab test and time point will show the shift at each post-baseline time point versus the baseline.

The following types of cross-tabulations will be prepared:

- for all tests with normal ranges: shift in abnormality (L/N/H)
- for ALT, AST, total bilirubin, GGT, leukocytes, neutrophils, thrombocytes, fibrinogen and lipids test results only: shift in CTCAE toxicity grades (grade 1 to 4)

Longitudinal box plots will be prepared for the following variables: neutrophils, platelets, ALT, AST and LDL/HDL ratio.

A detailed list of tables, figures and listings can be found in section 13.4, section 14 and section 15.4, respectively.

## 7.3 Physical Examination

Abnormal physical examination findings will be listed (see section 15.4). No summaries will be provided.

## 7.4 Vital Signs

The following parameters will be analysed: weight, systolic and diastolic blood pressure, pulse rate and body temperature.

Tables showing descriptive statistics (mean, median, standard error, minimum, and maximum) per vital sign test and unit and time point by treatment group and using the safety population will be prepared for:

- actual values
- absolute change from baseline

A detailed list of tables and listings can be found in section 13.4 and section 15.4, respectively.

## 8 ANALYSIS OF PHARMACOKINETICS

All analyses will be run on the PK population.

Drug concentration will be analyzed descriptively (n, arithmetic mean, SD and SE, median, minimum and maximum, 5% and 95% percentiles, CV% of arithmetic mean, geometric mean and geometric SD) by treatment group and timepoint.

Individual pharmacokinetic concentrations will be reported in  $\mu$ g/mL. Concentrations in ng/mL will be converted. Values BQL will be handled as detailed in section 4.3.2.

Pharmacokinetic concentrations and descriptive statistics will be reported to 3 significant digits for values up to, but not including 1000. Values equal to and above 1000 will be reported as the value without decimal signs. In case the actual sampling time deviates more than allowed per study protocol from the nominal time, these samples will not be included in the calculation of descriptive statistics.



A detailed list of tables and listings can be found in section 13.3 and section 15.4, respectively.

## 9 ANALYSIS OF IMMUNOGENICITY

## 9.1 Available parameters

Immunogenicity is assessed via a tiered sample analysis approach (illustrated in Figure 1). In a first step all samples will be analyzed in the conventional anti-drug antibody (ADA) assay and only samples from subjects classified as 'Pre-Ab Pos – Equivocal' will be further analyzed in the mADA assay. This assay is a characterization assay and has been developed to enable detection of TE ADA in presence of (high) pre-existing antibody (pre-Ab) levels. Furthermore, positive ADA samples will be evaluated for their neutralizing potential in the neutralizing antibody (NAb) assay.

As such, the available parameters per sample are:

- ADA log10(titer) (no data imputation)
- mADA log10(titer) (for subset of subjects only, no data imputation)
- NAb normalized response (for subset of samples only, data imputation required for ADA negative samples)

Additional provided information needed for data interpretation is:

- ADA Minimum Significance Ratio (MSR): MSR is an assay parameter reflecting
  precision of titer assessments and is needed to interpret the treatment emergent
  (TE) response for subjects presenting with pre-Ab. In such cases, pre- and postdose titers will be compared. The titer is considered to be significantly increased
  post-dose, if the highest post-dose titer compared to the highest pre-dose titer is
  higher than the MSR value. The increase of the log10(titer) post- versus pre-dose
  should be > log10(MSR).
- mADA MSR: MSR value determined in the mADA assay, similar application as described above, but applied to mADA titers.
- NAb assay cutpoint (CP): cut-off value to determine if a sample is negative or positive. Since the NAb assay is an inhibition assay, samples equal to or below the CP will be considered positive.





Table 1 provides clarification on when the reported value of a sample needs to be categorized as "negative", "positive" or "missing" in each of the respective assays. Samples scoring negative in the ADA or mADA assay are not titrated and the respective log10(titer) is reported as <log10(Minimal required dilution [MRD]) with MRD=100, i.e. log10(titer) <2.00. The latter will not to be included in descriptive statistics on titers; but they will be included in the individual line plot, set arbitrarily to 1.80. Similarly, NAb negative results should not be included in descriptive statistics on response ratios, but will be included in the individual line plot, set arbitrarily to 1.00.

Table 1: Reported values in each assay and corresponding data interpretation

| ADA: mADA: log10(titer) | | NAb data from<br>parent trial:<br>neutralizing<br>response <sup>1</sup> | NAb data C203<br>post-baseline<br>visits <sup>2</sup> :<br>response ratio | Data<br>interpretation |
|---|---|---|---|---|
| "< 2.00" | "< 2.00" | "Υ" | Numeric value > CP <sup>3</sup> | NEGATIVE<br>(NEG)<br>(ISORRES) |
| Numeric value<br>≥ 2.00 | Numeric value ≥<br>2.00 | "N" | Numeric value<br>≤ CP³ | POSITIVE (POS)<br>(ISORRES) |
| "NA" or "NR" | "NA" or "NR" | "NA" or "NR" | "NA" or "NR" | MISSING<br>(COVAL) |

<sup>&</sup>lt;sup>1</sup> Parent trial screening and baseline visit as well as OLE baseline visit (corresponding to w24/w12 for C201/C202 respectively)

The immunogenicity status prior to drug administration will be derived from the parent trial (ALX0061-C201 or ALX0061-202) screening and baseline sample results (see further). The TE/post-dose response will be evaluated based on samples collected within ALX0061-C203 (OLE) at following timepoints according to schedule of assessment: Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96, Week 104 and

<sup>&</sup>lt;sup>2</sup> NAb results reporting strategy has been adapted for study C203 compared to parent trial: NAb data are reported as response ratios, in contrast to C201/C202 results, which were reported as Y/N in the clinical database <sup>3</sup> CP will be reported along with actual sample results



FU or ET visit. In all immunogenicity TFLs organized per timepoint, both parent screening & baseline as well as Week 0 need to be included.

## 9.2 Missing results and data imputation

The mADA assay will only be performed on a subset of samples ('Pre-Ab Pos – Equivocal'). In case no mADA results are reported for a given subject, the corresponding fields in the listing will remain empty and no data imputation is to be done.

The NAb assay will only be performed on a subset of samples (ADA positive samples). In case no NAb results are reported (empty field), the following imputations will be made (imputed values will be followed by "\*" in listings):

- No NAb record and corresponding ADA result NEGATIVE: these samples will be considered NEGATIVE and should appear as "NEG\*" in listings
- No NAb record and corresponding ADA result Not Analyzed (NA): these samples will be considered "NA" and should appear as "NA\*" in listings
- No NAb record and corresponding ADA result POSITIVE or No Result (NR): these samples will be considered "NR" and should appear as "NR\*" in listings

## 9.3 Subject classifications (derived parameters)

Subject classification on immunogenicity results (ADA, mADA and NAb) will be based on the assay results (titers or response ratios outlined in 9.1). Subject classifications will be attributed based on all available data for each subject.

One subject will either have three or four subject classifications:

- an ADA subject classification (mandatory)
- a mADA subject classification (optional, only for subjects with ADA classification "Pre-Ab positive – Equivocal")
- an overall subject classification (combining results of ADA and mADA analysis)
- a NAb subject classification (mandatory, derived from reported and/or imputed results)

Subjects will be classified based on their pre-dose status (i.e. screening and baseline) and treatment-emergent (TE) status (post-dose response). The immunogenicity status prior to drug administration will be derived from the <u>parent trial (ALX0061-C201 or ALX0061-C202) screening and baseline</u> sample results. The TE/post-dose response will be evaluated based on samples collected within ALX0061-C203 at following time points: Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96, Week 104 and FU or ET visit.

#### 9.3.1 ADA subject classification

All available ADA assay results (positive or negative) per subject will be evaluated and subjects will be classified based on a combined statement on pre-Ab status (pre-Ab neg or pre-Ab pos, to be derived from parent trial) and the TE ADA response (TE neg, TE pos, Equivocal (EQ) or inconclusive) as outlined in Table 2.



For each subject, one ADA subject classification will be determined. This implies that in the listing subject classification will be identical for all ADA visits of the given subject.

Table 2: ADA subject classification

| ADA subject class | Evaluation based on all ADA assay results (titer) of the respective subject | |
|---|---|---|
| | Pre-Ab status evaluated on | TE ADA Response evaluated based on Week |
| | screening and baseline sample of | 12, Week 24, Week 36, Week 48, Week 60, |
| | parent trial | Week 72, Week 84, Week 96, Week 104 and |
| | | FU or ET visit |
| PRE-AB NEG - TE ADA NEG | All pre-dose samples negative | All post-dose samples ADA negative |
| PRE-AB NEG - TE ADA POS | All pre-dose samples negative | At least one positive ADA sample(s) post-dose |
| PRE-AB NEG - TE ADA | All pre-dose samples negative | All post-dose samples(/results) are missing |
| INCONCLUSIVE | | |
| PRE-AB POS - TE ADA NEG | One or more of the pre-dose | All post-dose samples are ADA negative |
| | samples is positive | |
| PRE-AB POS - TE ADA POS | One or more of the pre-dose | Significant increase in titer post-dose versus |
| | samples is positive | pre-dose* |
| PRE-AB POS - EQ | One or more of the pre-dose | Positive ADA sample(s) post-dose and no |
| | samples is positive | significant increase in titer post-dose versus |
| | | pre-dose* |
| PRE-AB POS – TE ADA | One or more of the pre-dose | All post-dose samples(/results) are missing |
| INCONCLUSIVE | samples is positive | |
| MISSING | No pre-dose samples are available | N/A |

<sup>\*</sup> The titer is considered to be significantly increased post-dose, if the highest post-dose titer compared to the highest pre-dose titer is higher than the ADA MSR value: the increase of the log10(titer) post- versus pre-dose should be > log10(MSR).

## 9.3.2 mADA subject classification

All available mADA assay results (positive or negative) per subject will be evaluated and subjects will be classified based on a combined statement on pre-Ab status (pre-Ab neg or pre-Ab pos, to be derived from parent trial) and the TE ADA response (TE neg, TE pos, EQ or inconclusive) as outlined in Table 3.

For each subject tested in the mADA assay (i.e. "PRE-AB POS – EQ" subjects based on ADA assessment), one mADA subject classification will be determined. This implies that in the listing this will be identical for all ADA visits of the given subject. In case the subject was not tested in the mADA assay, corresponding fields in the listing will remain empty.

Table 3: mADA subject classification

| mADA subject class | Evaluation based on all mADA assay results (titer) of the respective subject | |
|---|---|---|
| | Pre-Ab status evaluated on screening and baseline of parent trial | TE ADA Response evaluated based on<br>Week 12, Week 24, Week 36, Week 48,<br>Week 60, Week 72, Week 84, Week 96, |
| | | Week 104 and FU or ET visit |
| PRE-AB NEG - TE ADA NEG | All pre-dose samples negative | All post-dose samples ADA negative |
| PRE-AB NEG - TE ADA POS | All pre-dose samples negative | At least one positive ADA sample(s) post- |
| | | dose |
| PRE-AB NEG - TE ADA INCONCLUSIVE | All pre-dose samples negative | All post-dose samples(/results) are missing |

| PRE-AB POS - TE ADA NEG | One or more of the pre-dose samples is | All post-dose samples ADA negative |
|---|---|---|
| | positive | |
| PRE-AB POS - TE ADA POS | One or more of the pre-dose samples is | Significant increase in titer post-dose |
| | positive | versus pre-dose* |
| PRE-AB POS - EQ | One or more of the pre-dose samples is | Positive ADA sample(s) post-dose and no |
| | positive | significant increase in titer post-dose versus |
| | | pre-dose* |
| PRE-AB POS – TE ADA | One or more of the pre-dose samples is | All post-dose samples(/results) are missing |
| INCONCLUSIVE | positive | |
| MISSING | No pre-dose samples are available | N/A |

<sup>\*</sup> The titer is considered to be significantly increased post-dose, if the highest post-dose titer compared to the highest predose titer is higher than the mADA MSR value: the increase of the log10(titer) post- versus pre-dose should be > log10(MSR).

## 9.3.3 Overall subject classification

Overall subject classification will be determined based on the combined results of ADA and/or mADA analysis. The classification is identical to the ADA subject classification, except for subjects classified as "pre-Ab pos - EQ" based on ADA assay results which are further evaluated in the mADA assay. For those subjects, a re-classification is done based on combined ADA and mADA assay. This is illustrated in Table 4. For each subject, one overall subject classification is to be assigned. This implies that in the listing the overall subject classification will be identical for all ADA visits of the given subject.

Table 4: ADA, mADA and Overall subject classification

| ADA subject classification | mADA subject classification | Overall subject classification |
|---|---|---|
| Missing | - | Missing |
| PRE-AB NEG - TE ADA NEG | -<br>- | PRE-AB NEG - TE ADA NEG |
| PRE-AB NEG - TE ADA POS | <del>-</del> | PRE-AB NEG - TE ADA POS |
| PRE-AB NEG - TE ADA<br>INCONCLUSIVE | - | PRE-AB NEG - TE ADA<br>INCONCLUSIVE |
| PRE-AB POS - TE ADA NEG | - | PRE-AB POS - TE ADA NEG |
| PRE-AB POS - TE ADA POS | -<br>- | PRE-AB POS - TE ADA POS |
| PRE-AB POS - TE ADA<br>INCONCLUSIVE | - | PRE-AB POS - TE ADA<br>INCONCLUSIVE |
| PRE-AB POS - EQ — | Missing | PRE-AB POS - EQ |
| | PRE-AB NEG - TE ADA NEG | PRE-AB POS - EQ |
| | PRE-AB NEG - TE ADA POS | PRE-AB POS - TE ADA POS |
| | PRE-AB NEG - TE ADA INCONCLUSIVE | PRE-AB POS - EQ |
| | PRE-AB POS - TE ADA POS | PRE-AB POS - TE ADA POS |
| | PRE-AB POS - TE ADA<br>INCONCLUSIVE | PRE-AB POS - EQ |
| | PRE-AB POS – TE ADA NEG | PRE-AB POS – EQ |
| | PRE-AB POS – EQ | PRE-AB POS – EQ |



## 9.3.4 NAb subject class

All available NAb assay results (\*) (positive or (imputed) negative) per subject will be evaluated and subjects will be classified based on a combined statement on pre-dose status (pre-dose neg or pre-dose pos, to be derived from parent trial) and the post-dose response (negative, positive or inconclusive) as outlined in Table 5.

(\*) Note that for the pre-dose Nab results (screening and baseline) from the parent trials (ALX0061-C201 or ALX0061-C202) 'Y' (Yes) should be imputed to POS and 'N' (No) should be imputed to NEG.

For each subject, one NAb subject classification is to be determined. This implies that in the listing this will be identical for all NAb visits of the given subject. For subjects with no positive ADA samples, the NAb results were imputed as "NEG\*", and the NAb subject class will be "PRE-DOSE NEG - NEG ON TREATMENT". The latter also has to appear in the Listing.

Table 5: NAb subject classification

| NAb subject class | Evaluation based on all NAb assay results (titer) of the respective subject | |
|---|---|---|
| | Pre-dose status evaluated on screening | Response on treatment evaluated |
| | and baseline of parent trial | based on Week 12, Week 24, Week 36, |
| | | Week 48, Week 60, Week 72, Week 84, |
| | | Week 96, Week 104 and FU or ET visit |
| PRE-DOSE NEG - NEG | All pre-dose samples negative | All post-dose samples are negative |
| ON TREATMENT | (reported or imputed) | (reported or imputed) |
| PRE-DOSE NEG - POS | All pre-dose samples negative | At least one positive sample(s) post-dose |
| ON TREATMENT | (reported or imputed) | |
| PRE-DOSE POS - NEG | One or more of the pre-dose samples is | All post-dose samples are negative |
| ON TREATMENT | positive | (reported or imputed) |
| PRE-DOSE POS - POS | One or more of the pre-dose samples is | At least one positive sample(s) post-dose |
| ON TREATMENT | positive | |
| PRE-DOSE NEG - | All pre-dose samples negative | All post-dose samples(/results) are |
| INCONCLUSIVE | (reported or imputed) | missing |
| PRE-DOSE POS - | One or more of the pre-dose samples is | All post-dose samples(/results) are |
| INCONCLUSIVE | positive | missing |
| MISSING | No pre-dose (and/or post-dose) samples are | No pre-dose (and/or post-dose) sample: |
| | available | are available |

## 9.4 Pre-Ab prevalence and TE ADA Incidence calculations

#### 9.4.1 Incidence of ADA and derived sets

The following subject categories (1-8) and derived sets (9-15) will be used in the ADA incidence tables:

- 1. PRE-AB NEG TE ADA NEG
- 2. PRE-AB NEG TE ADA POS
- 3. PRE-AB NEG TE ADA INCONCLUSIVE
- 4. PRE-AB POS TE ADA NEG
- 5. PRE-AB POS TE ADA POS
- 6. PRE-AB POS EQ
- 7. PRE-AB POS TE ADA INCONCLUSIVE



- 8. MISSING
- 9. TOTAL PRE-AB NEG (equals 1 + 2 + 3)
- 10. TOTAL PRE-AB POS (equals 4 + 5 + 6 + 7)
- 11. TOTAL TE ADA NEG (equals 1 + 4)
- 12. TOTAL TE ADA POS (equals 2 + 5)
- 13. TOTAL TE INCONCLUSIVE (3 + 7)
- 14. TE POS within PRE-AB NEG POPULATION (equals 2/9)
- 15. TE POS within PRE-AB POS POPULATION (equals 5/10)

Incidences will be shown per treatment group. The number of subjects (s) in each subject category or derived set (excluding 14-15) is divided by the number of subjects (n) within each treatment group, excluding the subjects who are classified as missing. Incidences are shown as s/n (%), with the calculated percentage added in between brackets.

## 9.4.2 Incidence of mADA subject classes and derived sets

The same subject categories (1-8) and derived sets (9-15) as shown above in 9.4.1 will be presented in the mADA incidence table, but the denominator to calculate incidences differs.

Incidences will be shown per treatment group. The number of subjects (s) in each subject category or derived set (excluding 14-15) is divided by the number of subjects (n) within each treatment group which were characterized in mADA assay (i.e. "PRE-AB POS – EQ" in ADA assay), excluding the subjects who are classified as missing. Incidences are shown as s/n (%), with the calculated percentage added in between brackets.

## 9.4.3 Incidence of overall subject classification (ADA, mADA results) and derived sets

The following subject categories (1-8) and derived sets (9-13) will be used in the overall incidence tables:

- 1. PRE-AB NEG TE ADA NEG
- 2. PRE-AB NEG TE ADA POS
- 3. PRE-AB NEG TE ADA INCONCLUSIVE
- 4. PRE-AB POS TE ADA NEG
- 5. PRE-AB POS TE ADA POS
- 6. PRE-AB POS EQ
- 7. PRE-AB POS TE ADA INCONCLUSIVE
- 8. MISSING
- 9. TOTAL PRE-AB NEG (equals 1 + 2 + 3)
- 10. TOTAL PRE-AB POS (equals 4 + 5 + 6 + 7)
- 11. TOTAL TE ADA NEG (equals 1 + 4)
- 12. TOTAL TE ADA POS (equals 2 + 5)
- 13. TOTAL TE INCONCLUSIVE (3 + 7)
- 14. TE POS within PRE-AB NEG POPULATION (equals 2/9)
- 15. TE POS within PRE-AB POS POPULATION (equals 5/10)



Incidences will be shown per treatment group. The number of subjects (s) in each subject category or derived set (excluding 14-15) is divided by the number of subjects (n) within each treatment group, excluding the subjects who are classified as missing. Incidences are shown as s/n (%), with the calculated percentage added in between brackets.

## 9.4.4 Incidence of NAb subject classes and derived sets

The following subject categories (1-7) and derived sets (8-14) will be used in the mADA incidence tables:

- 1. PRE-DOSE NEG NEG ON TREATMENT
- 2. PRE-DOSE NEG POS ON TREATMENT
- 3. PRE-DOSE POS NEG ON TREATMENT
- 4. PRE-DOSE POS POS ON TREATMENT
- 5. PRE-DOSE NEG INCONCLUSIVE
- 6. PRE-DOSE POS INCONCLUSIVE
- 7. MISSING
- 8. TOTAL PRE-DOSE NEG (equals 1 + 2 + 5)
- 9. TOTAL PRE-DOSE POS (equals 3 + 4 + 6)
- 10. TOTAL NEG ON TREATMENT (equals 1 + 3)
- 11. TOTAL POS ON TREATMENT (equals 2 + 4)
- 12. TOTAL INCONCLUSIVE (5 + 6)
- 13. POS ON TREATMENT within PRE-DOSE NEG POPULATION (equals 2/8)
- 14. POS ON TREATMENT within PRE-DOSE POS POPULATION (equals 4/9)

Incidences will be shown per treatment group. The number of subjects (s) in each subject category or derived set (excluding 13-14) is divided by the number of subjects (n) within each treatment group, excluding the subjects who are classified as missing. Incidences are shown as s/n (%), with the calculated percentage added in between brackets.

## 9.4.5 Safety subgroup analysis

For the following subgroups, the incidence rates will be determined of the different overall subject classifications (1-8) as listed in 9.4.3.

- Injection-site reaction
  - No injection-site reaction
  - At least 1 injection-site reaction
- Hypersensitivity reaction
  - No hypersensitivity reaction
  - At least 1 hypersensitivity reaction



#### 9.4.6 ADA and NAb incidence over time

For ADA and NAb data, incidence of positive samples over time will be calculated. Positivity needs to be deducted based on reported titer values (ADA) or response ratio (NAb), as clarified in Table 1. Incidence calculation should account for subject drop-out: for each visit, the number of positive samples is divided by the available results for the given visit (positive + negative samples (reported and/or imputed), excluding missing values (NA & NR)). The latter should be clarified in a footnote of the concerning tables.

## 10 INTERIM ANALYSES

No interim analysis are foreseen.

## 11 CHANGE FROM ANALYSIS PLANNED IN PROTOCOL

The subgroup analysis for efficacy according to the protocol included demographics (including weight and region), baseline disease characteristics, and baseline and prior medications, but will be limited to age category and geographic region.

A second sensitivity analysis will be done for efficacy based on NRI for the categorical endpoints analysed in the first sensitivity analysis.

The protocol mentions a subgroup analysis for safety which will not be performed.

The protocol states descriptive statistics will be used to summarize changes from baseline, but model-based, baseline-adjusted LS means and 95% CI will be used for efficacy endpoints.

## 12 CONVENTIONS

## 12.1 Analysis Phases and Visit Windows

## 12.1.1 Algorithm of allocating visits to time windows

All assessments (including unscheduled assessments) will be placed into time windows according to their relative day (DY) in the study, according to the following allocation table:

| Time point label | Target day | Interval lower bound | Interval upper bound |
|------------------|------------|----------------------|----------------------|
| Week 4 | 29 | 1 | 43 |
| Week 8 | 57 | 44 | 71 |
| Week 12 | 85 | 72 | 126 |
| Week 24 | 169 | 141 | 197 |
| Week 36 | 253 | 225 | 281 |

| Time point label | Target day | Interval lower bound | Interval upper bound |
|---|---|---|---|
| Week 48 | 337 | 309 | 365 |
| Week 60 | 421 | 393 | 449 |
| Week 72 | 505 | 477 | 533 |
| Week 84 | 589 | 561 | 617 |
| Week 96 | 673 | 645 | 700 |
| Week 104 | 729 | 701 | Week 102 visit date + 28 days |
| Follow-up | | Last treatment date + 29 days | +INF |

The definition of the time window for "Follow-up" implies that for Week 4 to Week 104 assessments, if the assessment or sample date is more than 28 days after the last dose of treatment, the assessment will be mapped to the Follow-up visit. If the assessment or sample date is less than or equal to 28 days after the last dose of treatment (including for assessments or samples taken at the early termination visit, if this condition holds), the assessment will be mapped to the corresponding analysis visit, in case it falls within the interval lower and upper bound for this analysis visit.

Baseline is defined in section 4.2.1.

Tables, figures and listings will present the time points as defined above, not the case report form (CRF) visits.

#### 12.1.2 Selection of visits

It is possible that more than one visit gets allocated into the same time window. In that case, only one visit will be selected for analysis tables and figures. The nonselected visit(s) will only be listed. In case an assessment gets allocated to a time window at which the assessment was not scheduled as per protocol, this assessment will not be shown in the tables or figures but will only be listed.

The visit with a DY closest to the target day will be selected. In case of ties on the same day with time not available, the assessment linked with the CRF visit will be selected for analysis.

In case more than one parameter is measured per time point (e.g. for lab), the selection is performed per parameter and per time point, not per "sample" and per time point. Missing values are removed before the selection is made.



## 12.2 General characteristics

## 12.2.1 Derivation of exposure parameters

The following exposure parameters will be derived:

- Total treatment duration = date of last study drug administration date of first study drug administration in C203 + 14 days
- Total number of study drug doses received during C203
- Cumulative dose of study drug received: total dose of study drug in mg administered during C203
- Compliance = 100 \* (total number of study drug doses actually received during C203/expected number of study drug doses during C203)

Where the expected number of study drug doses is calculated as follows:

- For subjects completing the study: 52
- For subjects prematurely discontinuing the study: 1 baseline dose + integer of (date of last study drug administration – date of first study drug administration in C203)/14

## 12.3 Efficacy

The following assessments will be used to derive the efficacy parameters:

- Physician's assessment of tender/painful and swollen joint count: 68 joints are assessed for tenderness (TJC) and 66 joints are assessed for swelling (SJC). Joints that underwent intra-articular (IA) corticosteroid injection during the last 4 weeks will be considered as swollen and tender. Only joints that were ticked 'Yes' will be taken into account. Left and right will be summed to obtain one overall joint count.
- Physician's assessment of tender/painful and swollen joint count, selected: a selection of 28 joints are assessed for tenderness (TJC28) and for swelling (SJC28)
- Average duration of morning stiffness
- Patient's assessment of pain (100 mm) (VAS)
- Patient's global assessment of disease activity (100 mm) (VASPA)
- Physician's global assessment of disease activity (100 mm) (VASPHA)
- C-reactive protein concentration (mg/L) (CRP)
- Erythrocyte sedimentation rate (mm/h) (ESR)



- HAQ-DI (/60): 20-question instrument to assess the degree of difficulty to accomplish tasks in 8 functional areas (dressing and grooming, hygiene, arising, reach, eating, grip, walking, common daily activities) over the previous week. Responses for each question range from 0 (no difficulty) to 3 (unable to do). The score is calculated in 3 steps:
  - Derivation of the 8 category scores, by selecting the highest sub-category score
  - Adjusting for use of aids/devices and/or help from another person: scores of 0 or 1 will then be increased to 2
  - Calculating the mean of the category scores. In case less than 6 category scores are available, the HAQ-DI score will not be computed.
- SF-36 questionnaire: 36 item questionnaire that can be summarized into 8 domains (physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, mental health) and into 2 summary measures (physical component and mental component). Version 2 of the questionnaire was used (see Section 16.6. Appendix 6)
- FACIT-F: quality of life (QOL) questionnaire consisting of 40 questions ranging from 0 to 4, grouped in 5 domains (physical well-being, social/family well-being, emotional well-being, functional well-being and fatigue). Scoring guidelines to derive subscores and total scores can be found in section 16.4.

Based on the above assessments, the following parameters will be derived:

- ACR20 response:
  - YES if ALL of the following criteria are fulfilled:
    - % improvement relative to baseline in tender/painful joint count >= 20%
    - % improvement relative to baseline in swollen joint count >= 20%
    - " improvement relative to baseline >= 20% for at least 3 of the following assessments: patient's assessment of pain, patient's global assessment of disease activity, physician's global assessment of disease activity, HAQ-DI, CRP
  - NO if not all of the above criteria are fulfilled
  - Handling of missing values:
    - if TJC or SJC are missing, ACR response will be missing
    - if any of patient's assessment of pain, patient's global assessment of disease activity, physician's global assessment of disease activity, HAQ-DI or CRP are missing, but at least 3 have a change from baseline >= 20% or at least 3 have a change from baseline < 20%, ACR response can be derived, otherwise it will be missing.
- ACR50 response: definition similar to ACR20 response, but using 50% as cut-off
- ACR70 response: definition similar to ACR20 response, but using 70% as cut-off
### Ablynx CONFIDENTIAL



- ACR-N index of improvement: minimum of the following 3 criteria:
  - % improvement relative to baseline in tender/painful joint count
  - % improvement relative to baseline in swollen joint count
  - Median % improvement relative to baseline of the following assessments: patient's assessment of pain, patient's global assessment of disease activity, physician's global assessment of disease activity, HAQ-DI, CRP
- $DAS28(ESR) = (0.56 \times \sqrt{TJC28}) + (0.28 \times \sqrt{SJC28}) + (0.70 \times ln[ESR]) + (0.014 \times VASPA)$ , with VASPA measured in mm
- $DAS28(CRP) = (0.56 \times \sqrt{TJC28}) + (0.28 \times \sqrt{SJC28}) + (0.36 \times ln[CRP + 1]) + (0.014 \times VASPA) + 0.96$ , with VASPA measured in mm and CRP in mg/L
- EULAR response is defined as follows based on the actual value of DAS28 (DAS28) in both ESR and CRP and the change from baseline in DAS28 (ΔDAS28) in both ESR and CRP:
  - Good response:  $\Delta DAS28 > 1.2 \text{ AND } DAS28 \leq 3.2$
  - o Moderate response ( $\Delta DAS28 > 1.2~AND~DAS28 > 3.2$ )  $OR~(0.6 < \Delta DAS28 \le 1.2~AND~DAS28 \le 5.1$ )
  - o No response ( $\Delta DAS28 \le 0.6$ ) OR ( $0.6 < \Delta DAS28 \le 1.2$  AND DAS28 > 5.1)
  - Pooled category Moderate+Good will be shown as well.
- Disease activity is defined as follows based on the actual value of DAS28(ESR):
  - $\circ$  Remission: *DAS*28(*ESR*) < 2.6
  - Low disease activity:  $2.6 \le DAS28(ESR) \le 3.2$
  - Moderate disease activity:  $3.2 < DAS28(ESR) \le 5.1$
  - $\circ$  High disease activity: DAS28(ESR) > 5.1
  - Pooled category Remission + Low disease activity will be shown as well
- Disease activity is defined as follows based on the actual value of DAS28(CRP):
  - $\circ$  DAS28(CRP) < 2.6
  - Low disease activity:  $2.6 \le DAS28(CRP) \le 3.2$
  - Moderate disease activity:  $3.2 < DAS28(CRP) \le 5.1$
  - High disease activity: DAS28(CRP) > 5.1
  - Pooled category DAS28(CRP) < 2.6 + Low disease activity will be shown as well
- Boolean remission is defined as follows:
  - Yes:  $TJC28 \le 1$  AND  $SJC28 \le 1$  AND  $VASPA \le 1$  cm AND  $CRP \le 1$  mg/dL
  - o No: else
- Clinically meaningful improvement in HAQ-DI (clinically meaningful improvement from baseline – absolute change) is defined as follows:
  - Yes:  $\Delta HAQDI \ge 0.25$
  - o No:  $\Delta HAQDI < 0.25$

#### lynx CONFIDENTIAL



- Normal physical function based on HAQ-DI is defined as follows:
  - Yes: *HAQDI* ≤ 0.5No: *HAQDI* > 0.5
- CDAI score = TJC28 + SJC28 + VASPA (cm) + VASPHA (cm)
- CDAI classification:
  - Remission:  $CDAI \le 2.8$
  - Low disease activity:  $2.8 < CDAI \le 10$
  - Moderate disease activity:  $10 < CDAI \le 22$
  - High disease activity: 22 < CDAI
  - o Pooled category Remission+Low disease activity will be shown as well
- SDAI score = TJC28 + SJC28 + VASPA (cm) + VASPHA (cm) + CRP (mg/dL)
- SDAI classification:
  - Remission:  $SDAI \leq 3.3$
  - Low disease activity:  $3.3 < SDAI \le 11$
  - Moderate disease activity:  $11 < SDAI \le 26$
  - High disease activity: 26 < SDAI</li>
  - Pooled category Remission+Low disease activity will be shown as well
- Maintained remission at Week x: remission at Week x and all consecutive time points.

MTX and corticosteroid dose related endpoints will be derived as follows:

- MTX dose decrease from baseline at W0,W48 and W104:
  - Yes: daily dose at Week 0/ Week 48 / Week 104 visit < baseline dose</li>
  - o No: else
- Discontinuation of MTX dose at W0,W48 and W104:
  - Yes: daily dose at Week 0/ Week 48 / Week 104 visit = 0
  - o No: else
- Change from baseline of MTX dose at Week 0/ Week 48 / Week 104
- Change from baseline of corticosteroid dose at Week 0/ Week 48 / Week 104

### 12.4 Safety

#### 12.4.1 Adverse events

AE onset day and AE duration are defined as follows:

AE onset day

- AE start date date of first study drug intake in C203 + 1 day (when the AE start date is completely known)
- missing (when the AE start date is incomplete or unknown).



#### AE duration

- AE stop date AE start date + 1 day (when both dates are completely known)
- trial termination date AE start date + 1 day (when the AE start date is fully known but the AE is not resolved at the end of the trial): in this case the duration will be presented as ">x days" in the listing rather than "x days"
- missing (when the AE start date is incomplete or unknown, or when the AE has resolved but with an incomplete or unknown end date).

### 12.4.2 Laboratory

Values will be scored as abnormally low (L), normal (N) or abnormally high (H). A value is classified as abnormally low when the value < lower limit of the normal range. A value is classified as abnormally high when the value > upper limit of the normal range. Tests without normal ranges will not be scored.

An original value like "<X" where X equals the lower limit of the normal range will be classified as abnormally low (L). An original value like ">X" where X equals the upper limit of the normal range will be classified as abnormally high (H).

Urinalysis tests for which a normal range is available, will also be categorized as L, N, or H. If there is doubt on whether the result is within normal range or not, the worst-case will be taken. E.g., when the test result equals "4 to 6" and the normal range is 0-5, then the test result will be classified as abnormally high (H) if it is a post-baseline visit, and will be classified as normal (N) if it is a baseline visit. In such cases, the original urinalysis test result will not be used for the tables, but will only be listed. Urinalysis tests for which no normal range is available, will be tabulated separately as categorical data.

All nonmissing post-baseline values (including unscheduled measurements and follow-up measurements) will be used to derive the following worst-case abnormalities for each parameter:

- H = abnormally high: at least one postdose measurement is above the normal range, and there are no values below the normal range.
- L = abnormally low: at least one postdose measurement is below the normal range, and there are no values above the normal range.
- H+L = abnormally high and low: at least one postdose measurement is above the normal range, and at least one other postdose measurement is below the normal range.
- N = normal: all postdose measurements are within normal limits.

#### 13 INDEX OF TABLES

#### 13.1 General

#### Table 14.1.1.1: Subject disposition: Tabulation by analysis population

Tabulation of the number of subjects in each of the analysis populations defined in section 4.1.

Population: all screened population.



### Table 14.1.1.2: Subject disposition: Tabulation by region and country

Tabulation of the number of subjects per region and country.

Population: ITO population.

### Table 14.1.1.3: Subject disposition: Tabulation by time point

Tabulation of the number of subjects per time point.

Population: ITO population.

#### Table 14.1.1.4: Trial termination: Tabulation

Tabulation of study completion / study discontinuations and the primary reason for discontinuation.

Population: ITO population.

#### Table 14.1.1.5: Major protocol deviations: Tabulation

Tabulation of the major protocol deviations per category including Selection criteria not met / Subject not withdrawn as per protocol / Prohibited concomitant medication / Treatment non-compliance / Safety assessment deviation / Efficacy assessment deviation / Other.

Population: ITO population.

### Table 14.1.2.1: Demographic data: Tabulation and descriptive statistics

Descriptive statistics for continuous parameters and frequency tabulation for categorical parameters.

Population: ITO population.

# Table 14.1.2.2: Baseline disease characteristics: Tabulation and descriptive statistics

Descriptive statistics for continuous parameters and frequency tabulation for categorical parameters.

Population: ITO population.

### Table 14.1.2.3: Tabulation of RA related concomitant therapies by generic term

Tabulation of the generic terms of RA related concomitant therapies.

Population: safety population.

### Table 14.1.2.4: Tabulation of non-RA related concomitant therapies by generic term

Tabulation of the generic terms of non-RA related concomitant therapies.

Population: safety population.

#### Table 14.1.2.5: Exposure to study medication: Descriptive statistics

Descriptive statistics of exposure parameters except home administration, including compliance.

Population: safety population.

#### Table 14.1.2.6: Exposure to study medication: Home administration

Tabulation of any study drug administration received at home (yes/no) and of all study drug administrations received at home, except those received during a scheduled study visit (yes/no).



### 13.2 Efficacy

### Table 14.2.1.1.1: ACR response - ACR20 response

Frequency tabulation of the ACR20 response at each time point, including a Wilson score 95% CI on the percentage of subjects achieving ACR20 response.

Population: ITO.

### Table 14.2.1.1.2: ACR response - ACR50 response

Frequency tabulation of the ACR50 response at each time point, including a Wilson score 95% CI on the percentage of subjects achieving ACR50 response.

Population: ITO.

## Table 14.2.1.1.3: ACR response - ACR70 response

Frequency tabulation of the ACR70 response at each time point, including a Wilson score 95% CI on the percentage of subjects achieving ACR70 response.

Population: ITO.

#### Table 14.2.1.1.4: ACR response - ACR-N index of improvement

Descriptive statistics of the ACR-N index actual values at each time point.

Population: ITO.

#### Table 14.2.1.2.1: DAS28 Score – Actual values and change from baseline

Descriptive statistics of the DAS28(CRP) and the DAS28(ESR) score actual values and change from baseline at each time point. Additionally, the change from baseline at each time point will be modelled using an ANCOVA model with treatment group and baseline DAS28 score as covariates and the LS means with 95% CI will be reported.

Population: ITO.

#### Table 14.2.1.2.2: DAS28 Score – EULAR (using CRP and using ESR) response

Frequency tabulation of the EULAR response, based on the DAS28(CRP) and the DAS28(ESR) score at each time point, including a Wilson score 95% CI on the percentage of subjects achieving EULAR response.

Population: ITO.

#### Table 14.2.1.2.3: DAS28 Score – Disease activity (ESR)

Frequency tabulation of the disease activity, based on the DAS28(ESR) score at each time point, including a Wilson score 95% CI on the percentage of subjects achieving LDA/remission, remission and maintained remission.

Population: ITO.

#### Table 14.2.1.2.4: DAS28 Score – Disease activity (CRP)

Frequency tabulation of the disease activity, based on the DAS28(CRP) score at each time point, including a Wilson score 95% CI on the percentage of subjects achieving DAS28(CRP) ≤ 3.2, DAS28(CRP) < 2.6 and maintained DAS28(CRP) < 2.6.



#### Table 14.2.1.3.1: Boolean disease remission definition

Frequency tabulation of the disease remission, based on the Boolean definition at each time point, including a Wilson score 95% CI on the percentage of subjects achieving remission and maintained remission.

Population: ITO.

### Table 14.2.1.4.1: CDAI Score – Actual values and change from baseline

Descriptive statistics of the CDAI score actual values and change from baseline at each time point. Additionally, the change from baseline at each time point will be modelled using an ANCOVA model with treatment group and baseline CDAI score as covariates and the LS means with 95% CI will be reported.

Population: ITO.

### Table 14.2.1.4.2: CDAI Score – Disease activity

Frequency tabulation of the disease activity, based on the CDAI score at each time point, including a Wilson score 95% CI on the percentage of subjects achieving LDA/remission, remission and maintained remission.

Population: ITO.

#### Table 14.2.1.5.1: SDAI Score – Actual values and change from baseline

Descriptive statistics of the SDAI score actual values and change from baseline at each time point. Additionally, the change from baseline at each time point will be modelled using an ANCOVA model with treatment group and baseline SDAI score as covariates and the LS means with 95% CI will be reported.

Population: ITO.

#### Table 14.2.1.5.2: SDAI Score – Disease activity

Frequency tabulation of the disease activity, based on the SDAI score at each time point, including a Wilson score 95% CI on the percentage of subjects achieving LDA/remission, remission and maintained remission.

Population: ITO.

#### Table 14.2.1.6.1: HAQ-DI Score – Actual values and change from baseline

Descriptive statistics of the HAQ-DI score actual values and change from baseline at each time point. Additionally, the change from baseline at each time point will be modelled using an ANCOVA model with treatment group and baseline HAQ-DI score as covariates and the LS means with 95% CI will be reported.

Population: ITO.

#### Table 14.2.1.6.2: HAQ-DI Score – Clinically meaningful improvement

Frequency tabulation of the clinically meaningful improvement, based on the HAQ-DI score ( $\Delta HAQDI \geq 0.25$ ) at each time point, including a Wilson score 95% CI on the percentage of subjects with HAQ-DI response.



### Table 14.2.1.6.3: HAQ-DI Score – Normal physical function

Frequency tabulation of normal physical function, based on the HAQ-DI score ( $HAQDI \le 0.5$ ) at each time point, including a Wilson score 95% CI on the percentage of subjects achieving normal physical function.

Population: ITO.

# Table 14.2.1.7.1: SF-36 – Physical and mental component scores - Actual values and change from baseline

Descriptive statistics of the physical and mental component scores actual values and change from baseline at each time point. Additionally, the change from baseline at each time point will be modelled using an ANCOVA model with treatment group and baseline score as covariates and the LS means with 95% CI will be reported.

Population: ITO.

### Table 14.2.1.8.1: FACIT-F – Actual values and change from baseline

Descriptive statistics of the FACIT-F total score and scores of subscales actual values and change from baseline at each time point. Additionally, the change from baseline at each time point will be modelled using an ANCOVA model with treatment group and baseline FACIT-F score as covariates and the LS means with 95% CI will be reported.

Population: ITO.

# Table 14.2.1.9.1: Duration of morning stiffness – Actual values and change from baseline

Descriptive statistics of the duration of morning stiffness actual values and change from baseline at each time point. Additionally, the change from baseline at each time point will be modelled using an ANCOVA model with treatment group and baseline duration as covariates and the LS means with 95% CI will be reported.

Population: ITO.

#### Table 14.2.1.10.1: VAS scales – Actual values and change from baseline

Descriptive statistics of the patient's assessment of pain VAS, patient's global assessment of disease activity VAS and the physician's global assessment of disease activity VAS actual values and change from baseline at each time point. Additionally, the change from baseline at each time point will be modelled using an ANCOVA model with treatment group and baseline VAS as covariates and the LS means with 95% CI will be reported.

Population: ITO.

## Table 14.2.1.11.1: CRP and ESR – Actual values and change from baseline

Descriptive statistics of CRP and ESR concentrations actual values and change from baseline at each time point. Additionally, the change from baseline at each time point will be modelled using an ANCOVA model with treatment group and baseline CRP/ESR as covariates and the LS means with 95% CI will be reported.

Population: ITO.

### Table 14.2.1.12.1: TJC and SJC – Actual values and change from baseline

Descriptive statistics of tender joint counts and swollen joint counts actual values and change from baseline at each time point. Additionally, the change from baseline at each



time point will be modelled using an ANCOVA model with treatment group and baseline TJC/SJC count as covariates and the LS means with 95% CI will be reported.

Population: ITO.

### Table 14.2.1.13.1: RA therapy reduction – MTX dose reduction

Frequency tabulation of MTX dose reduction at 1 and 2 years, including a Wilson score 95% CI on the percentage of subjects achieving MTX dose reduction.

Population: ITO.

#### Table 14.2.1.13.2: RA therapy reduction – MTX discontinuation

Frequency tabulation of MTX discontinuation at 1 and 2 years, including a Wilson score 95% CI on the percentage of subjects discontinuing MTX.

Population: ITO.

# Table 14.2.1.13.3: RA therapy reduction – Actual values and change from baseline in MTX dose

Descriptive statistics of the actual values and change from baseline in MTX dose at 1 and 2 years. Additionally, the change from baseline at each time point will be modelled using an ANCOVA model with treatment group and baseline MTX dose as covariates and the LS means with 95% CI will be reported.

Population: ITO.

# Table 14.2.1.13.4: RA therapy reduction – Actual values and change from baseline in corticosteroids dose

Descriptive statistics of the actual values and change from baseline in prednisolone equivalent corticosteroids dose at 1 and 2 years. Additionally, the change from baseline at each time point will be modelled using an ANCOVA model with treatment group and baseline prednisolone equivalent corticosteroids dose as covariates and the LS means with 95% CI will be reported.

Population: ITO.

# Table 14.2.2.1.1: ACR response - ACR20 response - Last observation carried forward (LOCF)

Frequency tabulation of the ACR20 response at each time point, including a Wilson score 95% CI on the percentage of subjects achieving ACR20 response.

Population: ITO.

# Table 14.2.2.1.2: ACR response - ACR50 response - Last observation carried forward (LOCF)

Frequency tabulation of the ACR50 response at each time point, including a Wilson score 95% CI on the percentage of subjects achieving ACR50 response.

Population: ITO.

# Table 14.2.2.1.3: ACR response - ACR70 response - Last observation carried forward (LOCF)

Frequency tabulation of the ACR70 response at each time point, including a Wilson score 95% CI on the percentage of subjects achieving ACR70 response.



# Table 14.2.2.2.1: DAS28 Score – Actual values and change from baseline – Last observation carried forward (LOCF)

Descriptive statistics of the DAS28(CRP) and the DAS28(ESR) score actual values and change from baseline at each time point. Additionally, the change from baseline at each time point will be modelled using an ANCOVA model with treatment group and baseline DAS28 score as covariates and the LS means with 95% CI will be reported.

Population: ITO.

# Table 14.2.2.2.2: DAS28 Score – Disease activity (ESR) – Last observation carried forward (LOCF)

Frequency tabulation of the disease activity, based on the DAS28(ESR) score at each time point, including a Wilson score 95% CI on the percentage of subjects achieving LDA/remission, remission and maintained remission.

Population: ITO.

# Table 14.2.2.2.3: DAS28 Score – Disease activity (CRP) – Last observation carried forward (LOCF)

Frequency tabulation of the disease activity, based on the DAS28(CRP) score at each time point, including a Wilson score 95% CI on the percentage of subjects achieving DAS28(CRP) ≤ 3.2, DAS28(CRP) < 2.6 and maintained DAS28(CRP) < 2.6.

Population: ITO.

# Table 14.2.3.1.1: ACR response - ACR20 response - Non-responder imputation (NRI)

Frequency tabulation of the ACR20 response at each time point, including a Wilson score 95% CI on the percentage of subjects achieving ACR20 response.

Population: ITO.

# Table 14.2.3.1.2: ACR response - ACR50 response - Non-responder imputation (NRI)

Frequency tabulation of the ACR50 response at each time point, including a Wilson score 95% CI on the percentage of subjects achieving ACR50 response.

Population: ITO.

# Table 14.2.3.1.3: ACR response - ACR70 response - Non-responder imputation (NRI)

Frequency tabulation of the ACR70 response at each time point, including a Wilson score 95% CI on the percentage of subjects achieving ACR70 response.

Population: ITO.

# Table 14.2.3.2.1: DAS28 Score – Disease activity (ESR) – Non-responder imputation (NRI)

Frequency tabulation of the disease activity, based on the DAS28(ESR) score at each time point, including a Wilson score 95% CI on the percentage of subjects achieving LDA/remission, remission and maintained remission.



# Table 14.2.3.2.2: DAS28 Score – Disease activity (CRP) – Non-responder imputation (NRI)

Frequency tabulation of the disease activity, based on the DAS28(CRP) score at each time point, including a Wilson score 95% CI on the percentage of subjects achieving DAS28(CRP)  $\leq$  3.2, DAS28(CRP)  $\leq$  2.6 and maintained DAS28(CRP)  $\leq$  2.6.

Population: ITO.

#### Table 14.2.4.1.1: ACR response - ACR20 response by age category

Frequency tabulation of the ACR20 response by age category, including a Wilson score 95% CI on the percentage of subjects achieving ACR20 response for each treatment group.

Population: ITO.

### Table 14.2.4.1.2: ACR response - ACR50 response by age category

Frequency tabulation of the ACR50 response by age category, including a Wilson score 95% CI on the percentage of subjects achieving ACR50 response for each treatment group.

Population: ITO.

#### Table 14.2.4.1.3: ACR response - ACR70 response by age category

Frequency tabulation of the ACR70 response by age category, including a Wilson score 95% CI on the percentage of subjects achieving ACR70 response for each treatment group.

Population: ITO.

# Table 14.2.4.2.1: DAS28 Score – Actual values and change from baseline by age category

Descriptive statistics of the DAS28(CRP) and the DAS28(ESR) score actual values and change from baseline at each time point by age category.

Population: ITO.

### Table 14.2.4.2.2: DAS28 Score – Disease activity (ESR) by age category

Frequency tabulation of the disease activity, based on the DAS28(ESR) score by age category at each time point, including a Wilson score 95% CI on the percentage of subjects achieving LDA/remission, remission and maintained remission.

Population: ITO.

### Table 14.2.4.2.3: DAS28 Score – Disease activity (CRP) by age category

Frequency tabulation of the disease activity, based on the DAS28(CRP) score by age category at each time point, including a Wilson score 95% CI on the percentage of subjects achieving DAS28(CRP)  $\leq$  3.2, DAS28(CRP)  $\leq$  2.6 and maintained DAS28(CRP)  $\leq$  2.6.

Population: ITO.

### Table 14.2.5.1.1: ACR response - ACR20 response by region

Frequency tabulation of the ACR20 response by region, including a Wilson score 95% CI on the percentage of subjects achieving ACR20 response for each treatment group.



#### Table 14.2.5.1.2: ACR response - ACR50 response by region

Frequency tabulation of the ACR50 response by region, including a Wilson score 95% CI on the percentage of subjects achieving ACR50 response for each treatment group.

Population: ITO.

#### Table 14.2.5.1.3: ACR response - ACR70 response by region

Frequency tabulation of the ACR70 response by region, including a Wilson score 95% CI on the percentage of subjects achieving ACR70 response for each treatment group.

Population: ITO.

### Table 14.2.5.2.1: DAS28 Score – Actual values and change from baseline by region

Descriptive statistics of the DAS28(CRP) and the DAS28(ESR) score actual values and change from baseline at each time point by region.

Population: ITO.

## Table 14.2.5.2.2: DAS28 Score – Disease activity (ESR) by region

Frequency tabulation of the disease activity, based on the DAS28(ESR) score by region at each time point, including a Wilson score 95% CI on the percentage of subjects achieving LDA/remission, remission and maintained remission.

Population: ITO.

#### Table 14.2.5.2.3: DAS28 Score – Disease activity (CRP) by region

Frequency tabulation of the disease activity, based on the DAS28(CRP) score by region at each time point, including a Wilson score 95% CI on the percentage of subjects achieving DAS28(CRP)  $\leq$  3.2, DAS28(CRP) < 2.6 and maintained DAS28(CRP) < 2.6.

Population: ITO.

#### 13.3 Pharmacokinetics

#### Table 14.2.6.1: PK: Descriptive statistics of drug concentrations

Descriptive statistics of drug concentrations by scheduled sampling time and treatment group.

Population: PK population.

### 13.4 Safety

#### Table 14.3.1.1: Treatment-emergent adverse events: Summary table

Summary table of TEAEs presenting the number of events, the number and percentage of subjects and the incidence per 100 patient years.

Population: safety population.

# Table 14.3.1.2: Treatment-emergent adverse events: Summary table including TEAEs from the parent trials

Summary table of TEAEs including TEAEs from the parent trials presenting the number of events, the number and percentage of subjects and the incidence per 100 patient years. Population: safety population.



# Table 14.3.1.3: Treatment-emergent adverse events: Incidence of adverse events of special interest

Summary table of TEAEs of special interest presenting the number and percentage of subjects, the number of events and the incidence per 100 patient years.

Population: safety population.

# Table 14.3.1.4: Treatment-emergent adverse events: Incidence of adverse events of special interest including TEAEs from the parent trials

Summary table of TEAEs of special interest including TEAEs from the parent trials presenting the number and percentage of subjects, the number of events and the incidence per 100 patient years.

Population: safety population.

# Table 14.3.1.5: Treatment-emergent adverse events: Tabulation of all adverse events

Tabulation of TEAE preferred terms per system organ class and preferred term.

Population: safety population.

# Table 14.3.1.6: Treatment-emergent adverse events: Tabulation of all adverse events by severity

Tabulation of TEAE preferred terms per system organ class and preferred term by severity.

Population: safety population.

# Table 14.3.1.7: Treatment-emergent adverse events: Tabulation of adverse events with an incidence of at least 3%

Tabulation of TEAE preferred terms per system organ class. The incidence cut-off of 3% is to be calculated by treatment group.

Population: safety population.

# Table 14.3.1.8: Treatment-emergent adverse events: Tabulation of serious adverse events

Tabulation of serious TEAE preferred terms per system organ class and preferred term.

Population: safety population.

# Table 14.3.1.9: Treatment-emergent adverse events: Tabulation of non-serious adverse events

Tabulation of non-serious TEAE preferred terms per system organ class and preferred term.

Population: safety population.

### Table 14.3.1.10: Treatment-emergent adverse events: Tabulation of study drugrelated adverse events

Tabulation of TEAE preferred terms per system organ class and preferred term, selecting only the TEAEs that were study drug-related (as defined in section 7.1).



# Table 14.3.1.11: Treatment-emergent adverse events: Tabulation of adverse events related to study procedures

Tabulation of TEAE preferred terms per system organ class and preferred term, selecting only the TEAEs that were related to study procedures.

Population: safety population.

# Table 14.3.1.12: Treatment-emergent adverse events: Tabulation of the adverse events for which the trial or the study medication were discontinued

Tabulation of TEAE preferred terms per system organ class. Selecting only the TEAEs for which the study treatment was permanently discontinued, or for which the study was discontinued.

Population: safety population.

# Table 14.3.2.1: Laboratory data: Descriptive statistics of the actual values and change from baseline per time point

Descriptive statistics per lab test category (hematology, biochemistry, acute phase proteins, urinalysis, coagulation), lab test and unit and time point.

Population: safety population.

#### Table 14.3.2.2: Laboratory data: Frequency table of urinalysis results per time point

Frequency-tabulation per lab test and time point. The table will present the categorical results of urinalysis tests without normal range at each time point.

Population: safety population.

#### Table 14.3.2.3: Laboratory data: Cross-tabulation of the abnormalities per time point

Cross-tabulation per lab test category (hematology, biochemistry, acute phase proteins, urinalysis, coagulation), lab test and time point.

Population: safety population.

# Table 14.3.2.4: Laboratory data: Cross-tabulation of the CTCAE toxicity per time point for key hematology and biochemistry parameters

Cross-tabulation per lab test category, lab test and time point.

Population: safety population.

### Table 14.3.2.5: Laboratory data: Cross-tabulation of the worst-case abnormalities

Cross-tabulation per lab test category (hematology, biochemistry, acute phase proteins, urinalysis, coagulation) and lab test.

Population: safety population.

# Table 14.3.2.6: Laboratory data: Cross-tabulation of the worst-case CTCAE toxicity for key hematology and biochemistry parameters

Cross-tabulation per lab category and lab test.

Population: safety population.

# Table 14.3.3.1: Vital signs: Descriptive statistics of the actual values and change from baseline per time point

Descriptive statistics per test and unit and time point.



### 13.5 Immunogenicity

# Table 14.3.4.1: Immunogenicity: Prevalence and incidence table of pre-Ab and treatment-emergent ADA based on ADA assay results

Table sorted by treatment group. The table will present the incidence of different ADA subject categories and derived sets (see 9.4.1)

Population: safety population.

# Table 14.3.4.2: Immunogenicity: Prevalence and incidence table of pre-Ab and treatment-emergent ADA based on mADA assay results

Table sorted by treatment group. The table will present the incidence of different mADA subject categories and derived sets (see 9.4.2).

Population: safety population.

# Table 14.3.4.3: Immunogenicity: Prevalence and incidence table of pre-Ab and treatment-emergent ADA based on ADA and mADA assay results (overall subject classification)

Table sorted by treatment group. The table will present the incidence of different overall subject categories and derived sets (see 9.4.3)

Population: safety population.

# Table 14.3.4.4: Immunogenicity: Prevalence and incidence table of pre-dose and treatment-emergent ADA based on NAb results

Table sorted by treatment group. The table will present the NAb subject classification and derived sets (see 9.4.4).

Population: safety population.

# Table 14.3.4.5: Immunogenicity: Prevalence and incidence table of pre-Ab and treatment-emergent ADA based on ADA and mADA assay results (overall subject classification) by injection-site reaction

Table sorted by injection-site reaction category (see 9.4.5) and treatment group. The table will present the incidence of different overall subject classifications (no derived sets).

Population: safety population.

# Table 14.3.4.6: Immunogenicity: Prevalence and incidence table of pre-Ab and treatment-emergent ADA based on ADA and mADA assay results (overall subject classification) by hypersensitivity reaction

Table sorted by hypersensitivity reaction category (see 9.4.5) and treatment group. The table will present the incidence of different overall subject classifications (no derived sets). Population: safety population.

### Table 14.3.4.7: Immunogenicity: ADA incidence over time by pre-Ab population

Incidence of positive ADA samples at each time point by pre-Ab population and treatment group (see 9.4.6). NA & NR samples will be excluded from the incidence calculation.

Population: Safety population.

### Table 14.3.4.8: Immunogenicity: NAb incidence over time

Incidence of positive NAb samples (reported or imputed) at each time point by treatment group. NA & NR samples will be excluded from the incidence calculation.

ALX0061-C203 – Statistical Analysis Plan – Final 1.0 – 4 OCT 2018



Population: Safety population

# Table 14.3.4.9: Immunogenicity: ADA/mADA log10(Titer) over time by pre-Ab population

Descriptive statistics at each time point of titer values by pre-Ab population and treatment group. Within the pre-Ab negative population, only ADA log10(titers) will be available to calculate descriptive statistics. For the pre-Ab positive population, table will be subdivided in ADA and mADA log10(titer) results.

Population: Safety population.

# Table 14.3.4.10: Immunogenicity: NAb response ratio over time of NAb positive samples

Descriptive statistics at each time point of NAb response ratio by treatment group.

Population: Safety population.

## 14 INDEX OF FIGURES

#### Figure 14.2.1.1.1: ACR response - ACR20 response

Line plot of the percentage of subjects with ACR20 response at each time point, including SE bars, with one line per treatment group.

Population: ITO.

### Figure 14.2.1.1.2: ACR response - ACR50 response

Line plot of the percentage of subjects with ACR50 response at each time point, including SE bars, with one line per treatment group.

Population: ITO.

#### Figure 14.2.1.1.3: ACR response - ACR70 response

Line plot of the percentage of subjects with ACR70 response at each time point, including SE bars, with one line per treatment group.

Population: ITO.

### Figure 14.2.1.1.4: ACR response - ACR-N index of improvement

Line plot of the mean ACR-N index at each time point, including SE bars, with one line per treatment group.

Population: ITO.

### Figure 14.2.1.2.1: DAS28 Score – Actual values

Line plot of the mean DAS28(CRP) and the DAS28(ESR) score at each time point, including SE bars, with one line per treatment group. Separate graphs will be created for the DAS28(CRP) and the DAS28(ESR) score.

Population: ITO.

#### Figure 14.2.1.2.2: DAS28 Score – EULAR (using CRP and using ESR) response

Line plot of the percentage of subjects with EULAR good response at each time point, including SE bars, with one line per treatment group. Separate graphs will be created for EULAR response based on the DAS28(CRP) and on the DAS28(ESR).



### Figure 14.2.1.2.3: DAS28 Score – Disease activity

Line plot of the percentage of subjects with disease remission at each time point, including SE bars, with one line per treatment group. Separate graphs will be created for remission based on the DAS28(ESR) and for the DAS28(CRP)<2.6 category. The graphs will be repeated for percentage of subjects with LDA/disease remission.

Population: ITO.

#### Figure 14.2.1.3.1: Boolean disease remission definition

Line plot of the percentage of subjects with disease remission based on the Boolean definition at each time point, including SE bars, with one line per treatment group.

Population: ITO.

#### Figure 14.2.1.4.1: CDAI Score – Actual values

Line plot of the mean CDAI score at each time point, including SE bars, with one line per treatment group.

Population: ITO.

#### Figure 14.2.1.4.2: CDAI Score – Disease activity

Line plot of the percentage of subjects with disease remission based on the CDAI score at each time point, including SE bars, with one line per treatment group.

Population: ITO.

#### Figure 14.2.1.5.1: SDAI Score – Actual values

Line plot of the mean SDAI score at each time point, including SE bars, with one line per treatment group.

Population: ITO.

#### Figure 14.2.1.5.2: SDAI Score – Disease activity

Line plot of the percentage of subjects with disease remission based on the SDAI score at each time point, including SE bars, with one line per treatment group.

Population: ITO.

### Figure 14.2.1.6.1: HAQ-DI Score – Actual values

Line plot of the mean HAQ-DI score at each time point, including SE bars, with one line per treatment group.

Population: ITO.

#### Figure 14.2.1.6.2: HAQ-DI Score – Clinically meaningful improvement

Line plot of the percentage of subjects with HAQ-DI response at each time point, including SE bars, with one line per treatment group.

Population: ITO.

### Figure 14.2.1.6.3: HAQ-DI Score – Normal physical function

Line plot of the percentage of subjects with normal physical function, based on the HAQ-DI score at each time point, including SE bars, with one line per treatment group.



### Figure 14.2.1.7.1: SF-36 – Physical and mental component scores – Actual values

Line plot of the mean physical and mental component score at each time point, including SE bars, with one line per treatment group. Separate graphs will be created for the physical and mental component score.

Population: ITO.

#### Figure 14.2.1.8.1: FACIT-F – Actual values

Line plot of the mean FACIT-F total score and scores of subscales at each time point, including SE bars, with one line per treatment group.

Population: ITO.

#### Figure 14.2.1.9.1: Duration of morning stiffness – Actual values

Line plot of the mean duration of morning stiffness at each time point, including SE bars, with one line per treatment group.

Population: ITO.

#### Figure 14.2.1.10.1: VAS scales – Actual values

Line plot of the mean patient's assessment of pain VAS, patient's global assessment of disease activity VAS and the physician's global assessment of disease activity VAS, including SE bars, with one line per treatment group. Separate graphs will be created for the patient's assessment of pain VAS, patient's global assessment of disease activity VAS and the physician's global assessment of disease activity VAS.

Population: ITO.

#### Figure 14.2.1.11.1: CRP and ESR – Actual values

Line plot of the mean CRP and ESR concentrations, including SE bars, with one line per treatment group. Separate graphs will be created for CRP and ESR concentrations.

Population: ITO.

## Figure 14.2.1.12.1: TJC and SJC - Actual values

Line plot of the mean TJC and SJC, including SE bars, with one line per treatment group. Separate graphs will be created for TJC and SJC.

Population: ITO.

#### Figure 14.2.1.13.1: PK: Mean drug concentrations

Line plot of the mean drug concentrations, including SE bars, with one line per treatment group. Plots will be created with both linear and semi-logarithmic PK profiles. Both graphs will be displayed on the same page.

Population: PK population.

# Figure 14.2.1.13.2: PK: Mean drug concentrations (geometric mean)

Line plot of the geometric mean drug concentrations, including geometric SD bars, with one line per treatment group. Plots will be created with both linear and semi-logarithmic PK profiles. Both graphs will be displayed on the same page.

Population: PK population.



# Figure 14.2.1.13.3: Immunogenicity: Individual line plot of ADA log10(titer), mADA log10(titer), NAb response, PK concentration, DAS 28 Score and ACR50 over time

For all subjects, line plot of ADA titer, mADA titer, NAb response ratio, PK, DAS28(CRP), and ACR50 vs. time (incl. parent screening & baseline visit). Different responses can be plotted against separate Y-axes above each other, but scale of time-axis should be identical for each plotted response. Note that for parent screening and baseline visit and OLE baseline visit, NAb response will be indicated by a flag (pos="Y" or neg="N") above the corresponding ADA titer. For PK and DAS28(CRP), a treatment group average over time plot will be added with each of the individual plot.

Population: safety population.

#### Figure 14.3.1.1: Laboratory – box plots of parameters of interest

Longitudinal box plots per treatment group of neutrophils, platelets, ALT, AST and cholesterol ratio. Separate graphs will be created for each parameter.

Population: ITO.

### 15 INDEX OF LISTINGS

### 15.1 General

### Listing 16.2.1.1: Subject disposition

Listing of subject numbers, parent trial, dose in parent trial, population indicators, investigator and country.

Population: ITO population.

### Listing 16.2.1.2: Trial visits

Listing of all visits, including the visit date and study day.

Population: ITO population.

### Listing 16.2.1.3: Subject disposition: First and last contact in the trial

List with the following 3 dates:

- Date of the first signature on (C203) trial ICF
- Last visit date (all visits; including unscheduled visits)
- Last date of contact in the study with any subject.

Population: all screened population.

#### **Listing 16.2.1.4: Trial termination**

Listing of completion/discontinuation, the reason for discontinuation and the number of days since first study treatment administration at trial termination. In case the discontinuation was due to AE, the AE will be presented in this listing. If there is another explanation on the discontinuation reason collected in the CRF, this will also be presented in this listing.

Population: ITO population.



### Listing 16.2.1.5: Trial termination for adverse event

Same as previous listing for subjects with primary reason for study discontinuation adverse event.

Population: ITO population.

#### Listing 16.2.1.6: Major protocol deviations

Listing of all major protocol deviations.

Population: ITO population.

### Listing 16.2.1.7: No-treatment subjects

Listing of all subjects that were not treated, including the screening failures. The trial termination reason and/or the reason for being a no-treatment subject will be listed, whichever is available.

Population: all screened population, minus the safety population.

#### Listing 16.2.2.1: Demographic data

Listing of all demographic parameters. Country will be presented on this listing as well.

Population: ITO population.

### Listing 16.2.2.2: Baseline disease characteristics

Listing of all baseline disease characteristics parameters which are not listed in the efficacy section.

Population: ITO population.

### Listing 16.2.2.3: Concomitant therapies

Listing of all data on concomitant therapies, including coding information.

Population: ITO population.

#### Listing 16.2.2.4: Exposure to study medication: Actual data

Listing of all data collected in the CRF related to the use of study medication.

Population: safety population.

### Listing 16.2.2.5: Exposure to study medication: Derived data

Listing of all derived data related to the use of study medication.

Population: safety population.

#### Listing 16.2.2.6: Comments

Listing of remarks and comments written in the CRF.

Population: ITO population.

#### 15.2 Efficacy

#### Listing 16.2.3.1: ACR response

Listing per subject and visit of ACR20, ACR50 and ACR70 response and ACR-N index Population: ITO.



#### Listing 16.2.3.2: TJC and SJC

Listing per subject and visit of TJC and SJC actual values, changes and percentage changes from baseline

Population: ITO.

#### Listing 16.2.3.3: DAS28

Listing per subject and visit of TJC28, SJC28, CRP, ESR, DAS28(ESR), DAS28(CRP), EULAR response, DAS28(ESR) disease activity, DAS28(CRP) disease activity, VASPA and Boolean remission.

Population: ITO.

#### Listing 16.2.3.4: CDAI and SDAI

Listing per subject and visit of CDAI actual values, changes from baseline, disease activity and of SDAI actual values, changes from baseline, disease activity.

Population: ITO.

### **Listing 16.2.3.5: HAQ-DI**

Listing per subject and visit of HAQ-DI actual values, changes from baseline, percentage changes from baseline, response (clinically meaningful improvement) and normal physical function.

Population: ITO.

#### Listing 16.2.3.6: SF-36

Listing per subject and visit of the actual values and changes from baseline for the physical and mental component scores and for the 8 subscales (original scores).

Population: ITO.

#### Listing 16.2.3.7: FACIT-F and duration of morning stiffness

Listing per subject and visit of the actual values and changes from baseline for FACIT-F total score and subscales and of the actual values and changes from baseline for duration of morning stiffness.

Population: ITO.

#### Listing 16.2.3.8: VAS scales

Listing per subject and visit of the actual values, percentage changes from baseline and changes from baseline for VAS, VASPA and VASPHA.

Population: ITO.

#### Listing 16.2.3.9: CRP and ESR

Listing per subject and visit of the actual values, percentage changes from baseline and changes from baseline for CRP and ESR concentrations.

Population: ITO.

#### 15.3 Pharmacokinetics

#### Listing 16.2.4.1: PK: Study drug concentrations

Listing of all individual study drug concentrations.

Population: PK population.



### Listing 16.2.4.2: PK: Sampling times

Listing of nominal sampling times, actual sampling times and sampling time deviations. In case the actual sampling time deviates more than allowed per study protocol from the nominal time, the time point will be flagged.

Population: PK population.

### 15.4 Safety

#### Listing 16.2.7.1: Adverse events

Listing of all adverse events (started or ongoing in the C203 study) of the following:

- AE verbatim
- AE preferred term (flagging serious TEAEs with an asterisk \*)
- AE start and end
- AE onset day
- AE duration
- AE severity
- AE drug relatedness: relation to study drug, to MTX (C201 subjects only), to folic acid and to study procedure
- AE outcome
- AE action taken related to study drug
- Concomitant therapy started (yes/no)

Population: safety population.

#### Listing 16.2.7.2: Serious adverse events

Same as the previous listing, but only selecting SAEs. Additionally, the reason(s) for SAE will be listed as well.

Population: safety population.

#### **Listing 16.2.7.3: Treatment-related adverse events**

Same as the previous listing, but only selecting treatment-related TEAEs.

Population: safety population.

# Listing 16.2.7.4: Adverse events leading to discontinuation of the study or the study medication

Same as the previous listing, but only selecting TEAEs that lead to a stop of trial medication, or of the trial itself.



#### Listing 16.2.7.5: Adverse events leading to death

Same as the previous listing, but only selecting TEAEs that lead to death.

#### Listing 16.2.7.6: Severe/Serious hypersensitivity adverse events

Listing of severe/serious hypersensitivity adverse events, including ADA/mADA log10(titer) and biomarker test results (tryptase, total complement (CH50) and circulating immune complexes).

Population: safety population.

#### Listing 16.2.7.7: Physical examinations: Abnormalities

Listing of all abnormal findings, including the clinically significance status.

Population: safety population.

### Listing 16.2.7.8: Pregnancy tests

Listing of all pregnancy test results, for women of childbearing potential only.

Population: ITO population.

### Listing 16.2.8.1: Laboratory data: Full listing

Listing of raw laboratory data and changes, including a fasted (Y/N) flag, an abnormality L/H flag, the test's normal range and a clinical relevance flag.

Population: safety population.

#### Listing 16.2.8.2: Laboratory data: Abnormalities

Listing similar to 16.2.8.1, but only consisting of data scored as out-of-normal-range or clinically significant, plus also the baseline reference time point.

Population: safety population.

# Listing 16.2.8.3: Laboratory data: Abnormalities for key hematology and biochemistry parameters

Listing of ALT, AST, total bilirubin, gamma-glutamyltransferase, leukocytes, neutrophils, thrombocytes, fibrinogen and lipids scored as at least CTCAE toxicity grade 1, plus also the baseline reference time point.

Population: safety population.

#### **Listing 16.2.8.4: Laboratory data: Comments**

Listing of all comments. This listing will be linked to the full listing and the abnormalities listings via numbered entries like "[C13]".

Population: safety population.

#### Listing 16.2.9.1: Vital signs: Full listing

Listing of all parameters: raw values, changes from baseline, and flagging clinically significant results.

Population: safety population.

#### Listing 16.2.9.2: Vital signs: Abnormalities

Listing of all data scored as clinically significant, plus also the baseline reference time point.



### 15.5 Immunogenicity

### Listing 16.2.10.1: Immunogenicity: Full listing

Listing of all immunogenicity parameters (ADA log10(titer), ADA subject classification, mADA log10(titer), mADA subject classification, overall subject classification, NAb result ("yes"/"no" for data obtained from parent trial; ratio for OLE post-baseline visits) and nAb subject classification at each time point (parent trial screening and/or baseline sample results, the "C203 baseline" results and Week 12, Week 24, Week 36, Week 48, Week 60, Week 72, Week 84, Week 96, Week 104 and FU or ET visit).



# **16 APPENDICES**

16.1 Appendix 1: Schedule of assessments



| Study Period | Screening/E | Screening/Baseline, Treatment and Assessment period (weeks) | | | | | | | | Early Termination <sup>c</sup> (weeks) | Follow-up<br>(weeks) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Visit <sup>D</sup> | Screening/<br>Baseline <sup>B</sup> | 4 | 8 | 12 | 24 | 36 | 48 | 60 | 72 | 84 | 96 | 104 | 2 (after last study<br>drug<br>administration) | 12 (after last<br>study drug<br>dosing) |
| Visit Number | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | | 13 |
| Ambulatory visit | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Written informed consent | Х | | | | | | | | | | | | | |
| Review of entry criteria | Х | | | | | | | | | | | | | |
| Smoking history | Х | | | | | | | | | | | | | |
| Study drug injection card dispensation | Х | | | | | | | | | | | | | |
| Study drug administration (via interactive web response system [IWRS]) E | Х | Inje | | ns to c | continu | ie eve | ry 2 w | eeks ( | up to a | and inc | cluding | g week | | |
| Physical examination | XΒ | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Vital signs <sup>F</sup> | ΧB | Х | Х | Χ | Х | Х | Χ | Х | Х | Х | Х | Х | X | Х |
| Tuberculosis (TB) evaluation (questioning) | ΧB | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Routine clinical laboratory analyses <sup>H</sup> | ΧB | Х | Х | Х | | Х | | Х | | Х | Х | | | Х |
| Extended clinical laboratory analyses (including fasting serum lipids) <sup>1</sup> | ХВ | | | | Х | | Х | | Х | | | Х | Х | |
| Pregnancy test (urine) for females of childbearing potential only | XΒ | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Morning stiffness duration | ΧB | | | | | | | | | | | Х | Х | |
| Joint assessment (66/68-joint count) | ΧB | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| IWRS notification of tender & swollen joint counts | X <sup>B</sup> | | | Х | Х | Х | Х | Х | Х | Х | Х | | | |



| Patient pain visual analogue scale (VAS) | ΧB | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Health Assessment Questionnaire – Disability Index (HAQ-DI) | X <sup>B</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Short Form (36) Health Survey (SF-36) | X <sup>B</sup> | | Х | | Х | | Х | | | Х | Х | |
| Functional Assessment of Chronic Illness<br>Therapy – | X <sup>B</sup> | | Х | | Х | | Х | | | Х | Х | |
| Fatigue (FACIT-Fatigue) | | | | | | | | | | | | |
| Physician and Patient global assessment of disease activity | X <sup>B</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Concomitant medication | X <sup>B</sup> | <u> </u> | 1 | 1 | | | | 1 | | | | <b>—</b> |
| Adverse events (AEs) <sup>J</sup> | X <sup>B</sup> | | | | | | | | | | | <b>—</b> |
| Pharmacokinetic (PK) samples <sup>K</sup> | X <sup>B</sup> | Х | Х | Х | Х | Х | Х | Х | Х | Х | X | |
| Immunogenicity samples | ΧB | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |

- A. All assessments are to be completed prior to the study drug administration, except for subjects who discontinue study drug injections. The order of assessments if more than 1 assessment is planned at the same time should be performed according to the following principles: vital signs should be assessed prior to blood sampling; patient reported outcomes should occur prior to the physician's joint evaluation, independent joint assessment should occur prior to physician's global assessment, and study drug should be dosed after all other assessments have been performed.
- B. The Baseline Visit will coincide with the 24-week End of Treatment Visit of the preceding Study ALX0061-C201, or with the 12-week End of Treatment Visit of Study ALX0061-C202. The results from the End of Treatment Visit assessments for these studies do not have to be repeated at baseline for this study, and include physical examination, vital signs, TB evaluation (questioning), routine/extended clinical laboratory analyses (at Week 22 in Study ALX0061-C201 or at Week 10 in Study ALX0061-C202), pregnancy test (urine), morning stiffness duration, joint assessment (66/68-joint count), patient pain VAS, HAQ-DI, SF-36, FACIT-F, physician and patient global assessment, concomitant medication, AEs, PK blood samples, and immunogenicity.
- c. The Early Termination Visit is to be performed 2 weeks after the last study drug dosing for subjects who discontinue from the trial for other reasons than described in the efficacy discontinuation criteria (see section 3.2.3.2), unless they discontinue during a study visit, in which case that becomes their Early Termination Visit. For subjects who will meet the efficacy discontinuation criteria at Week 12, 24, 36, 48, 60, 72, 84 or 96, the visit at which subjects will meet these discontinuation criteria is defined as the Early Termination Visit.
- D. All post baseline visits may occur at the indicated week  $\pm$  3 days throughout the trial.
- E. At the study visits at Weeks 0, 4, 8, 12, 24, 36, 48, 60, 72, 84, and 96, study drug is to be administered s.c. at the study site. At all other time points, subjects are allowed to self-administer away from the clinic. Subjects unable to have injections administered away from the study site will be required to return to the site every 2 weeks for administration of study drug by an authorized health professional.

# Ablynx

- F. Vital signs (assessment after 5 minutes in supine position) will include weight, blood pressure, pulse, and temperature. A height measurement is not required (data available from the preceding study). In case blood sampling is to be performed at the same visit, the vital signs assessment is to be performed prior to the blood sampling.
- G. If TB is suspected at any time during the study, chest x-ray and interferon-gamma release assay (IGRA) should be performed.
- H. Samples for routine clinical laboratory analyses will be collected predose, and include blood chemistry, hematology, acute phase proteins (C-reactive protein [CRP], erythrocyte sedimentation rate [ESR], fibrinogen) and urinalysis (urinalysis at Weeks 48 and 104). For subjects on warfarin, international normalized ratio (INR) will be performed at Weeks 0, 4, 8, 12, 24, 36, 48, 60, 72, 84, and 96, or at the Early Termination Visit.
- I. At the indicated visits, samples for extended clinical laboratory analyses, including fasting serum lipids on top of the routine clinical laboratory analyses, will be performed predose. Extended clinical laboratory samples will be taken predose after the subject has been fasting for at least 10 h.
- J. AEs will be recorded from the time the informed consent form is signed through the Follow-up Visit. The Investigator must follow-up on all SAEs and AEs until the events have subsided, returned to baseline, or the subject's condition has stabilized in cases of permanent impairment. In case of acute or delayed severe/serious hypersensitivity reactions, an additional serum sample should be collected as soon as possible after the start of the event (blood volume: 5 mL).
- к. PK and immunogenicity samples will be taken predose.



# 16.2 Appendix 2: Prednisolone equivalent dose chart

| | Approx. equivalent dose (mg/day)* | Conversion factor |
|--------------------|-----------------------------------|-------------------|
| Cortisone | 25 | 0.20 |
| Hydrocortisone | 20 | 0.25 |
| Methylprednisolone | 4 | 1.25 |
| Prednisolone | 5 | 1.00 |
| Prednisone | 5 | 1.00 |
| Triamcinolone | 4 | 1.25 |
| Betamethasone | 0.70 | 7.15 |
| Dexamethasone | 0.75 | 6.67 |
| Deflazacort | 6 | 0.83 |

<sup>\*</sup> Based on Prednisolone dose of 5 mg/day.

### References:

Dixon JS (1991), Meikle AW and Tyler FH (1977), Webb R, Singer M. and Nayal S et al. (2005)



# 16.3 Appendix 3: CTCAE grades (version 4.03 14JUN2010)

| | | Investigations | • | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Activated partial thromboplastin<br>time prolonged | >ULN - 1.5 x ULN | >1.5 - 2.5 x ULN | >2.5 x ULN; hemorrhage | - | - |
| | | romboplastin time is found to be g<br>s and disorders, both primary and | | possible indicator of coagulopat | hy, a prolonge |
| Alanine aminotransferase | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| | oratory test results that indicate a | n increase in the level of alanine a | ।<br>minotransferase (ALT or SGPT) ir | the blood specimen. | <u> </u> |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the level of alkaline p | hosphatase in a blood specimen. | | |
| Aspartate aminotransferase<br>increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the level of aspartate | aminotransferase (AST or SGOT | ) in a blood specimen. | |
| Blood antidiuretic hormone<br>abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding based on lab | oratory test results that indicate al | bnormal levels of antidiuretic horm | one in the blood specimen. | | |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 10.0 x ULN | >10.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n abnormally high level of bilirubin | in the blood. Excess bilirubin is as | ssociated with jaundice. | |
| Blood corticotrophin decreased | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Hospitalization indicated | - | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of corticotroph | nin in a blood specimen. | | |
| Blood gonadotrophin abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | - |
| Definition: A finding based on lab | ı | ı<br>bnormal levels of gonadotrophin h | ormone in a blood specimen. | ı | 1 |
| Blood prolactin abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; limiting instrumental ADL | - | - | - |
| Definition: A finding based on lab | ļ. | ।<br>bnormal levels of prolactin hormon | l<br>le in a blood specimen. | I | Ţ |
| Carbon monoxide diffusing | | 6 - 8 units below LLN; for follow- | Asymptomatic decrease of >8 | - | _ |
| capacity decreased | up, a decrease of 3 - 5 units<br>(ml/min/mm Hg) below the<br>baseline value | up, an asymptomatic decrease<br>of >5 - 8 units (ml/min/mm Hg)<br>below the baseline value | units drop; >5 units drop along<br>with the presence of pulmonary<br>symptoms (e.g., >Grade 2<br>hypoxia or >Grade 2 or higher<br>dyspnea) | | |
| Definition: A finding based on lun | g function test results that indicate | a decrease in the lung capacity | to absorb carbon monoxide. | ı | |
| Cardiac troponin I increased | Levels above the upper limit of<br>normal and below the level of<br>myocardial infarction as defined<br>by the manufacturer | - | Levels consistent with<br>myocardial infarction as defined<br>by the manufacturer | - | - |
| · | | of cardiac troponin I in a biological | T . | T | 1 |
| Cardiac troponin T increased | Levels above the upper limit of<br>normal and below the level of<br>myocardial infarction as defined<br>by the manufacturer | - | Levels consistent with myocardial infarction as defined by the manufacturer | - | - |
| Definition: A laboratory test result | t which indicates increased levels | of cardiac troponin T in a biologica | al specimen. | | |
| CD4 lymphocytes decreased | <lln -="" 0.5="" 500="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <500 - 200/mm3; <0.5 - 0.2 x<br>10e9 /L | <200 - 50/mm3; <0.2 x 0.05 -<br>10e9 /L | <50/mm3; <0.05 x 10e9 /L | - |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of CD4 lymph | ocytes in a blood specimen. | | |
| Cholesterol high | >ULN - 300 mg/dL; >ULN - 7.75<br>mmol/L | >300 - 400 mg/dL; >7.75 - 10.34<br>mmol/L | >400 - 500 mg/dL; >10.34 -<br>12.92 mmol/L | >500 mg/dL; >12.92 mmol/L | - |
| Definition: A finding based on lab | oratory test results that indicate hi | igher than normal levels of cholest | erol in a blood specimen. | | |
| CPK increased | >ULN - 2.5 x ULN | >2.5 x ULN - 5 x ULN | >5 x ULN - 10 x ULN | >10 x ULN | - |

| | | Investigations | 3 | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| reatinine increased | >1 - 1.5 x baseline; >ULN - 1.5<br>x ULN | >1.5 - 3.0 x baseline; >1.5 - 3.0 x ULN | >3.0 baseline; >3.0 - 6.0 x ULN | >6.0 x ULN | - |
| efinition: A finding based on la | boratory test results that indicate in | ncreased levels of creatinine in a b | lological specimen. | | |
| jection fraction decreased | - | Resting ejection fraction (EF) 50<br>- 40%; 10 - 19% drop from<br>baseline | Resting ejection fraction (EF) 39<br>- 20%; >20% drop from baseline | | - |
| Definition: The percentage compontraction. | outed when the amount of blood ej | ected during a ventricular contract | ion of the heart is compared to the | amount that was present prior to | the |
| Electrocardiogram QT corrected<br>nterval prolonged | QTc 450 - 480 ms | QTc 481 - 500 ms | QTc >= 501 ms on at least two<br>separate ECGs | QTc >= 501 or >60 ms change<br>from baseline and Torsade de<br>pointes or polymorphic<br>ventricular tachycardia or<br>signs/symptoms of serious<br>arrhythmia | - |
| efinition: A finding of a cardiac | dysrhythmia characterized by an a | abnormally long corrected QT Inter | val. | | |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25% decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50% decrease from baseline | <0.5 - 0.25 x LLN or 50 - <75%<br>decrease from baseline | <0.25 x LLN or 75% decrease<br>from baseline or absolute value<br><50 mg/dL | - |
| efinition: A finding based on la | boratory test results that indicate a | n decrease in levels of fibrinogen | in a blood specimen. | T | |
| Forced expiratory volume<br>decreased | FEV1% (percentages of<br>observed FEV1 and FVC<br>related to their respective<br>predicted values) 99 - 70%<br>predicted | FEV1 60 - 69% | 50 - 59% | <= 49% | - |
| efinition: A finding based on te | st results that indicate a relative de | crease in the fraction of the force | vital capacity that is exhaled in a | specific number of seconds. | |
| GGT Increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | - CO ODD WILLIAM | | |
| | -024 - 2.0 x 0214 | >2.5 - 5.0 X OLIN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| Definition: A finding based on lai | boratory test results that indicate h | igher than normal levels of the en | ı<br>zyme gamma-glutamyltransferase | In the blood specimen. GGT (gam | ima- |
| Definition: A finding based on lai<br>plutamyltransferase ) catalyzes ( | boratory test results that indicate h<br>the transfer of a gamma glutamyl g | igher than normal levels of the en-<br>group from a gamma glutarnyl pepi<br>T | ı<br>zyme gamma-glutamyltransferase | In the blood specimen. GGT (gam | ima- |
| Definition: A finding based on lai | boratory test results that indicate h | igher than normal levels of the en | ı<br>zyme gamma-glutamyltransferase | In the blood specimen. GGT (gam | rma- |
| efinition: A finding based on lai<br>ilutamyltransferase ) catalyzes i<br>srowth hormone abnormal | boratory test results that indicate h<br>the transfer of a gamma glutamyl of<br>Asymptomatic; clinical or<br>diagnostic observations only; | igher than normal levels of the en-<br>group from a gamma glutamyl pepi<br>Symptomatic; medical<br>Intervention indicated; limiting<br>Instrumental ADL | yyme gamma-gjutamyltransferase<br>tide to another peptide, amino acid | In the blood specimen. GGT (gam | -<br>Ima- |
| efinition: A finding based on lai<br>lutamytransferase ) catalyzes i<br>crowth hormone abnormal<br>definition: A finding based on lai | boratory test results that indicate he<br>the transfer of a gamma glutamyl of<br>Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | igher than normal levels of the en-<br>group from a gamma glutamyl pepi<br>Symptomatic; medical<br>Intervention indicated; limiting<br>Instrumental ADL | yyme gamma-gjutamyltransferase<br>tide to another peptide, amino acid | In the blood specimen. GGT (gam | -<br>nma-<br> - |
| Definition: A finding based on lai<br>ilutamyttransferase ) catalyzes i<br>Frowth hormone abnormal<br>Definition: A finding based on lai<br>daptoglobin decreased | boratory test results that indicate he<br>the transfer of a gamma glutamyi g<br>Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated<br>boratory test results that indicate a | igher than normal levels of the en-<br>group from a gamma glutamyl pepi<br>Symptomatic; medical<br>Intervention indicated; limiting<br>Instrumental ADL<br>bnormal levels of growth hormone | yyme gamma-glutamyitransferase<br>tide to another peptide, amino acid<br>-<br>-<br>ln a biological specimen. | In the blood specimen. GGT (gam | -<br>ima-<br>- |
| Definition: A finding based on lai<br>liutamyttransferase ) catalyzes (<br>Growth hormone abnormal<br>Definition: A finding based on lai<br>saptoglobin decreased<br>Definition: A finding based on lai | boratory test results that indicate he transfer of a gamma glutamyl gray Asymptomatic; clinical or diagnostic observations only; intervention not indicated boratory test results that indicate a LLN boratory test results that indicate a | igher than normal levels of the en-<br>group from a gamma glutamyl pepi<br>Symptomatic; medical<br>Intervention indicated; limiting<br>Instrumental ADL<br>bnormal levels of growth hormone | zyme gamma-glutamyitransferase<br>tide to another peptide, amino acid<br>-<br>-<br>In a biological specimen.<br>-<br>In in a blood specimen. | In the blood specimen. GGT (gam | -<br> ma-<br> -<br> - |
| Definition: A finding based on lai<br>jutamyttransferase ) catalyzes (<br>Growth hormone abnormal<br>Definition: A finding based on lai<br>Haptoglobin decreased<br>Definition: A finding based on lai<br>Hemoglobin increased | boratory test results that indicate in the transfer of a gamma glutamyl graph of diagnostic observations only; intervention not indicated boratory test results that indicate a LLN boratory test results that indicate a increase in >0 - 2 gm/dL above ULN or above baseline if | igher than normal levels of the engroup from a gamma glutamyl pepi Symptomatic; medical intervention indicated; limiting instrumental ADL bhoormal levels of growth hormone - n decrease in levels of haptoglobil increase in >2 - 4 gm/dL above ULN or above baseline if baseline is above ULN | in a blood specimen. Increase in >4 gm/dL above ULN or above baseline if baseline is above ULN | In the blood specimen. GGT (gam | |
| efinition: A finding based on ial<br>lutamytransferase ) catalyzes to<br>crowth hormone abnormal<br>definition: A finding based on ial<br>laptoglobin decreased<br>definition: A finding based on ial<br>demoglobin increased<br>definition: A finding based on ial<br>definition: A finding based on ial<br>definition: A finding based on ial | boratory test results that indicate he transfer of a gamma glutamyl glasmyn glutamyl glasmyn glutamyl glasmyn | igher than normal levels of the engroup from a gamma glutamyl pepi Symptomatic; medical intervention indicated; limiting instrumental ADL bhoormal levels of growth hormone - n decrease in levels of haptoglobil increase in >2 - 4 gm/dL above ULN or above baseline if baseline is above ULN | in a blood specimen. Increase in >4 gm/dL above ULN or above baseline if baseline is above ULN | In the blood specimen. GGT (gam | |
| lefinition: A finding based on lai<br>lutamytransferase ) catalyzes to<br>prowth hormone abnormal<br>definition: A finding based on lai<br>daptoglobin decreased<br>definition: A finding based on lai<br>demoglobin increased<br>definition: A finding based on lai<br>definition: A finding based on lai | boratory test results that indicate in the transfer of a gamma glutamyl graph of diagnostic observations only; intervention not indicated boratory test results that indicate a lincrease in >0 - 2 gm/dL above ULN or above baseline if baseline is above ULN boratory test results that indicate in >1 - 1.5 x ULN; >1 - 1.5 times above baseline if on | igher than normal levels of the engroup from a gamma glutamyl pepi Symptomatic; medical intervention indicated; limiting instrumental ADL bhoormal levels of growth hormone - n decrease in levels of haptoglobi increase in >2 - 4 gm/dL above ULN or above baseline if baseline is above ULN creased levels of hemoglobin in a >1.5 - 2.5 x ULN; >1.5 - 2.5 times above baseline if on anticoagulation | in a blood specimen. Increase in >4 gm/dL above ULN or above baseline if baseline is above ULN blological specimen. >2.5 x ULN; >2.5 times above baseline if on anticoagulation | In the blood specimen. GGT (gam is or water | |
| efinition: A finding based on ial<br>lutamytransferase ) catalyzes to<br>irrowth hormone abnormal<br>efinition: A finding based on ial<br>laptoglobin decreased<br>lefinition: A finding based on ial<br>lemoglobin increased<br>lefinition: A finding based on ial<br>NR increased<br>lefinition: A finding based on ial<br>NR increased | boratory test results that indicate in the transfer of a gamma glutamyl gampa glutamyl glutam | igher than normal levels of the engroup from a gamma glutamyl pepi Symptomatic; medical intervention indicated; limiting instrumental ADL bhoormal levels of growth hormone - n decrease in levels of haptoglobi increase in >2 - 4 gm/dL above ULN or above baseline if baseline is above ULN creased levels of hemoglobin in a >1.5 - 2.5 x ULN; >1.5 - 2.5 times above baseline if on anticoagulation | in a blood specimen. Increase in >4 gm/dL above ULN or above baseline if baseline is above ULN blological specimen. >2.5 x ULN; >2.5 times above baseline if on anticoagulation | In the blood specimen. GGT (gam is or water | |
| efinition: A finding based on ial<br>lutamytransferase ) catalyzes to<br>irrowth hormone abnormal<br>efinition: A finding based on ial<br>laptoglobin decreased<br>lefinition: A finding based on ial<br>lemoglobin increased<br>lefinition: A finding based on ial<br>IR increased<br>lefinition: A finding based on ial<br>lipase increased | boratory test results that indicate he transfer of a gamma glutamyl glutamyl gamma glutamyl glutamy | igher than normal levels of the engroup from a gamma glutamyl pepi symptomatic; medical intervention indicated; limiting instrumental ADL bnormal levels of growth hormone - n decrease in levels of haptoglobil increase in > 2 - 4 gm/dL above ULN or above baseline if baseline is above ULN acreased levels of hemoglobin in a > 1.5 - 2.5 x ULN; > 1.5 - 2.5 times above baseline if on anticoagulation in increase in the ratio of the patier > 1.5 - 2.0 x ULN | tyme gamma-glutamyttransferase tide to another peptide, amino acid - In a biological specimen. Increase in >4 gm/dL above ULN or above baseline if baseline is above ULN biological specimen. >2.5 x ULN; >2.5 times above baseline if on anticoagulation int's prothrombin time to a control since it is prothrombin time to a c | In the blood specimen. GGT (gam is or water. | |
| efinition: A finding based on ial<br>lutamytransferase ) catalyzes is<br>crowth hormone abnormal<br>efinition: A finding based on ial<br>laptoglobin decreased<br>lefinition: A finding based on ial<br>lemoglobin increased<br>lefinition: A finding based on ial<br>liR increased<br>lefinition: A finding based on ial<br>lipase increased<br>lefinition: A finding based on ial<br>lipase increased<br>lefinition: A finding based on ial<br>lipase increased | boratory test results that indicate he transfer of a gamma glutamyl of Asymptomatic; clinical or diagnostic observations only; intervention not indicated boratory test results that indicate a location of the same of the sa | igher than normal levels of the engroup from a gamma glutamyl pepi symptomatic; medical intervention indicated; limiting instrumental ADL bnormal levels of growth hormone - in decrease in levels of haptoglobil increase in >2 - 4 gm/dL above ULN or above baseline if baseline is above ULN increased levels of hemoglobin in a >1.5 - 2.5 x ULN; >1.5 - 2.5 times above baseline if on anticoagulation in increase in the ratio of the patier >1.5 - 2.0 x ULN in increase in the level of lipase in | tyme gamma-glutamyttransferase tide to another peptide, amino acid - In a biological specimen. Increase in >4 gm/dL above ULN or above baseline if baseline is above ULN biological specimen. >2.5 x ULN; >2.5 times above baseline if on anticoagulation int's prothrombin time to a control since it is prothrombin time to a c | In the blood specimen. GGT (gam is or water. | |
| efinition: A finding based on ial lutamytransferase ) catalyzes to contain the contained of | boratory test results that indicate he transfer of a gamma glutamyl of Asymptomatic; clinical or diagnostic observations only; intervention not indicated boratory test results that indicate a location of the same of the sa | igher than normal levels of the en; proup from a gamma glutamyl pepi symptomatic; medical intervention indicated; limiting instrumental ADL bnormal levels of growth hormone - n decrease in levels of haptoglobi increase in >2 - 4 gm/dL above ULN or above baseline if baseline is above ULN ncreased levels of hemoglobin in a >1.5 - 2.5 x ULN; >1.5 - 2.5 times above baseline if on anticoagulation in increase in the ratio of the patier >1.5 - 2.0 x ULN in lincrease in the level of lipase in <800 - 500/mm3; <0.8 - 0.5 x 10e9 /L | tyme gamma-glutamyttransferase tide to another peptide, amino acid - In a biological specimen. Increase in >4 gm/dL above ULN or above baseline if baseline is above ULN biological specimen. >2.5 x ULN; >2.5 times above baseline if on anticoagulation hts prothrombin time to a control so >2.0 - 5.0 x ULN a biological specimen. >2.5 x ULN; >2.5 times above baseline if on anticoagulation | In the blood specimen. GGT (gam is or water. | |
| refinition: A finding based on lai lutamytransferase ) catalyzes is crowth hormone abnormal refinition: A finding based on lai laptoglobin decreased refinition: A finding based on lai lemoglobin increased refinition: A finding based on lai lai lapse increased refinition: A finding based on lai layer passed refinition: A finding based on lai layer passed refinition: A finding based on lai layer phocyte count decreased refinition: A finding based on lai layer phocyte count decreased refinition: A finding based on lai layer phocyte count decreased refinition: A finding based on lai layer phocyte count decreased refinition: A finding based on lai | Asymptomatic; clinical or diagnostic observations only; intervention not indicated boratory test results that indicate a cLLN boratory test results that indicate a lincrease in >0 - 2 gm/dL above ULN or above ULN boratory test results that indicate in >1 - 1.5 x ULN; >1 - 1.5 times above baseline if on anticoagulation boratory test results that indicate a >ULN - 1.5 x ULN; >1 - 1.5 times above baseline and conditional or above baseline and conditional or allowed by the conditional or anticoagulation boratory test results that indicate a >ULN - 1.5 x ULN boratory test results that indicate a <iln -="" 0.8="" 10e9="" 800="" <iln="" l<="" mm3;="" td="" x=""><td>igher than normal levels of the en; proup from a gamma glutamyl pepi symptomatic; medical intervention indicated; limiting instrumental ADL bnormal levels of growth hormone - n decrease in levels of haptoglobi increase in &gt;2 - 4 gm/dL above ULN or above baseline if baseline is above ULN ncreased levels of hemoglobin in a &gt;1.5 - 2.5 x ULN; &gt;1.5 - 2.5 times above baseline if on anticoagulation in increase in the ratio of the patier &gt;1.5 - 2.0 x ULN in lincrease in the level of lipase in &lt;800 - 500/mm3; &lt;0.8 - 0.5 x 10e9 /L</td><td>tyme gamma-glutamyttransferase tide to another peptide, amino acid - In a biological specimen. Increase in &gt;4 gm/dL above ULN or above baseline if baseline is above ULN biological specimen. &gt;2.5 x ULN; &gt;2.5 times above baseline if on anticoagulation hts prothrombin time to a control so &gt;2.0 - 5.0 x ULN a biological specimen. &gt;2.5 x ULN; &gt;2.5 times above baseline if on anticoagulation</td><td>In the blood specimen. GGT (gam is or water. </td><td></td></iln> | igher than normal levels of the en; proup from a gamma glutamyl pepi symptomatic; medical intervention indicated; limiting instrumental ADL bnormal levels of growth hormone - n decrease in levels of haptoglobi increase in >2 - 4 gm/dL above ULN or above baseline if baseline is above ULN ncreased levels of hemoglobin in a >1.5 - 2.5 x ULN; >1.5 - 2.5 times above baseline if on anticoagulation in increase in the ratio of the patier >1.5 - 2.0 x ULN in lincrease in the level of lipase in <800 - 500/mm3; <0.8 - 0.5 x 10e9 /L | tyme gamma-glutamyttransferase tide to another peptide, amino acid - In a biological specimen. Increase in >4 gm/dL above ULN or above baseline if baseline is above ULN biological specimen. >2.5 x ULN; >2.5 times above baseline if on anticoagulation hts prothrombin time to a control so >2.0 - 5.0 x ULN a biological specimen. >2.5 x ULN; >2.5 times above baseline if on anticoagulation | In the blood specimen. GGT (gam is or water. | |
| efinition: A finding based on lai<br>lutamyttransferase ) catalyzes to<br>irrowth hormone abnormal<br>efinition: A finding based on lai<br>laptoglobin decreased<br>lefinition: A finding based on lai<br>lemoglobin increased<br>lefinition: A finding based on lai<br>lipase increased<br>lefinition: A finding based on lai<br>lipase increased<br>lefinition: A finding based on lai<br>lymphocyte count decreased<br>lefinition: A finding based on lai<br>lymphocyte count decreased<br>lefinition: A finding based on lai<br>lymphocyte count increased | Asymptomatic; clinical or diagnostic observations only; intervention not indicated boratory test results that indicate a cLLN boratory test results that indicate a lincrease in >0 - 2 gm/dL above ULN or above ULN boratory test results that indicate in >1 - 1.5 x ULN; >1 - 1.5 times above baseline if on anticoagulation boratory test results that indicate a >ULN - 1.5 x ULN; >1 - 1.5 times above baseline and conditional or above baseline and conditional or allowed by the conditional or anticoagulation boratory test results that indicate a >ULN - 1.5 x ULN boratory test results that indicate a <iln -="" 0.8="" 10e9="" 800="" <iln="" l<="" mm3;="" td="" x=""><td>igher than normal levels of the en; proup from a gamma glutamyl pepi symptomatic; medical intervention indicated; limiting instrumental ADL bnormal levels of growth hormone - in decrease in levels of haptoglobi increase in &gt;2 - 4 gm/dL above ULN or above baseline if baseline is above ULN orceased levels of hemoglobin in a &gt;1.5 - 2.5 x ULN; &gt;1.5 - 2.5 times above baseline if on anticoagulation in increase in the ratio of the patter &gt;1.5 - 2.0 x ULN increase in the ratio of the patter &gt;1.5 - 2.0 x ULN increase in the level of lipase in &lt;800 - 500/mm3; &lt;0.8 - 0.5 x 10e9 /L decrease in number of lymphocyt &gt;4000/mm3 - 20,000/mm3</td><td>eyme gamma-glutamyttransferase tide to another peptide, amino acid In a biological specimen. Increase in &gt;4 gm/dL above ULN or above baseline if baseline is above ULN I biological specimen. &gt;2.5 x ULN; &gt;2.5 times above baseline if on anticoagulation t's prothrombin time to a control s &gt;2.0 - 5.0 x ULN a biological specimen. &lt;500 - 200/mm3; &lt;0.5 - 0.2 x 10e9 /L es in a biood specimen. &gt;20,000/mm3</td><td>In the blood specimen. GGT (gam is or water. ample in the blood. &gt;5.0 x ULN &lt;200/mm3; &lt;0.2 x 10e9 /L</td><td>-</td></iln> | igher than normal levels of the en; proup from a gamma glutamyl pepi symptomatic; medical intervention indicated; limiting instrumental ADL bnormal levels of growth hormone - in decrease in levels of haptoglobi increase in >2 - 4 gm/dL above ULN or above baseline if baseline is above ULN orceased levels of hemoglobin in a >1.5 - 2.5 x ULN; >1.5 - 2.5 times above baseline if on anticoagulation in increase in the ratio of the patter >1.5 - 2.0 x ULN increase in the ratio of the patter >1.5 - 2.0 x ULN increase in the level of lipase in <800 - 500/mm3; <0.8 - 0.5 x 10e9 /L decrease in number of lymphocyt >4000/mm3 - 20,000/mm3 | eyme gamma-glutamyttransferase tide to another peptide, amino acid In a biological specimen. Increase in >4 gm/dL above ULN or above baseline if baseline is above ULN I biological specimen. >2.5 x ULN; >2.5 times above baseline if on anticoagulation t's prothrombin time to a control s >2.0 - 5.0 x ULN a biological specimen. <500 - 200/mm3; <0.5 - 0.2 x 10e9 /L es in a biood specimen. >20,000/mm3 | In the blood specimen. GGT (gam is or water. ample in the blood. >5.0 x ULN <200/mm3; <0.2 x 10e9 /L | - |
| Definition: A finding based on iai ijutamytransferase ) catalyzes (a prowith hormone abnormal definition: A finding based on iai daptoglobin decreased definition: A finding based on iai demoglobin increased definition: A finding based on iai demoglobin increased definition: A finding based on iai demoglobin: A finding based on ia | boratory test results that indicate he the transfer of a gamma glutamyl of Asymptomatic; clinical or diagnostic observations only; intervention not indicated boratory test results that indicate a substitution of a substitution of a linerase in >0 - 2 gm/dL above ULN or above baseline if baseline is above ULN boratory test results that indicate in a linerase in >0 - 2 gm/dL above ULN or above baseline if baseline is above ULN boratory test results that indicate in anticoagulation boratory test results that indicate a substitution of a lineratory test results that indicate a lineratory test results th | igher than normal levels of the en; proup from a gamma glutamyl pepi symptomatic; medical intervention indicated; limiting instrumental ADL bnormal levels of growth hormone - in decrease in levels of haptoglobil increase in >2 - 4 gm/dL above ULN or above baseline if baseline is above ULN orceased levels of hemoglobin in a >1.5 - 2.5 x ULN; >1.5 - 2.5 times above baseline if on anticoagulation in increase in the ratio of the patter >1.5 - 2.0 x ULN increase in the level of lipase in 10e9 /L decrease in number of lymphocyt >4000/mm3 - 20,000/mm3 in abnormal increase in the number of intervention. | eyme gamma-glutamyttransferase tide to another peptide, amino acid In a biological specimen. Increase in >4 gm/dL above ULN or above baseline if baseline is above ULN I biological specimen. >2.5 x ULN; >2.5 times above baseline if on anticoagulation t's prothrombin time to a control s >2.0 - 5.0 x ULN a biological specimen. <500 - 200/mm3; <0.5 - 0.2 x 10e9 /L es in a biood specimen. >20,000/mm3 | In the blood specimen. GGT (gam is or water. | - |
| Definition: A finding based on lai illutamytransferase ) catalyzes is crowth hormone abnormal definition: A finding based on lai itaptoglobin decreased definition: A finding based on lai illutans and the complete of the co | Asymptomatic; clinical or diagnostic observations only; intervention not indicated boratory test results that indicate a subserved in the server of the serv | igher than normal levels of the en; proup from a gamma glutamyl pepi symptomatic; medical intervention indicated; limiting instrumental ADL bnormal levels of growth hormone - in decrease in levels of haptoglobil increase in >2 - 4 gm/dL above ULN or above baseline if baseline is above ULN orceased levels of hemoglobin in a >1.5 - 2.5 x ULN; >1.5 - 2.5 times above baseline if on anticoagulation in increase in the ratio of the patien >1.5 - 2.0 x ULN increased levels of lipase in levels of lipase in levels of lipase in levels of lipase in the ratio of the patien >1.5 - 2.0 x ULN increase in the level of lipase in levels | eyme gamma-glutamyttransferase tide to another peptide, amino acid In a biological specimen. Increase in >4 gm/dL above ULN or above baseline if baseline is above ULN Ibiological specimen. >2.5 x ULN; >2.5 times above baseline if on anticoagulation 1's prothrombin time to a control s >2.0 - 5.0 x ULN a biological specimen. <500 - 200/mm3; <0.5 - 0.2 x 10e9 /L es in a biood specimen. >20,000/mm3 or of lymphocytes in the blood, effur <1000 - 500/mm3; <1.0 - 0.5 x 10e9 /L | In the blood specimen. GGT (gam is or water. | - |



| | | Investigations | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Platelet count decreased | <lln -="" -<="" 75,000="" <lln="" mm3;="" td=""><td>&lt;75,000 - 50,000/mm3; &lt;75.0 -</td><td>&lt;50,000 - 25,000/mm3; &lt;50.0 -</td><td>&lt;25,000/mm3; &lt;25.0 x 10e9 /L</td><td>-</td></lln> | <75,000 - 50,000/mm3; <75.0 - | <50,000 - 25,000/mm3; <50.0 - | <25,000/mm3; <25.0 x 10e9 /L | - |
| | 75.0 x 10e9 /L | 50.0 x 10e9 /L | 25.0 x 10e9 /L | | |
| Definition: A finding based on lab | oratory test results that indicate a | decrease in number of platelets in | a blood specimen. | | |
| Serum amylase Increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 - 5.0 x ULN | >5.0 x ULN | - |
| Definition: A finding based on lab | coratory test results that indicate a | n increase in the levels of amylase | In a serum specimen. | | |
| Urine output decreased | - | - | Oliguria (<80 ml in 8 hr) | Anuria (<240 ml in 24 hr) | - |
| Definition: A finding based on tes | ,<br>st results that indicate urine produc | tion is less relative to previous ou | tput. | | • |
| Vital capacity abnormal | 90 - 75% of predicted value | <75 - 50% of predicted value; | <50% of predicted value; | - | - |
| | | limiting instrumental ADL | limiting self care ADL | | |
| Definition: A finding based on pu value. | imonary function test results that in | ndicate an abnormal vital capacity | (amount of exhaled after a maxim | um Inhalation) when compared to | the predicted |
| Weight gain | 5 - <10% from baseline | 10 - <20% from baseline | >=20% from baseline | - | - |
| Definition: A finding characterize | d by an increase in overall body w | eight; for pediatrics, greater than t | he baseline growth curve. | | |
| Weight loss | 5 to <10% from baseline; | 10 - <20% from baseline; | >=20% from baseline; tube | - | - |
| | Intervention not indicated | nutritional support Indicated | feeding or TPN indicated | | |
| Definition: A finding characterize | d by a decrease in overall body we | eight; for pediatrics, less than the b | paseline growth curve. | | |
| White blood cell decreased | <lln -="" 3.0="" 3000="" <lln="" mm3;="" td="" x<=""><td>&lt;3000 - 2000/mm3; &lt;3.0 - 2.0 x</td><td>&lt;2000 - 1000/mm3; &lt;2.0 - 1.0 x</td><td>&lt;1000/mm3; &lt;1.0 x 10e9 /L</td><td>-</td></lln> | <3000 - 2000/mm3; <3.0 - 2.0 x | <2000 - 1000/mm3; <2.0 - 1.0 x | <1000/mm3; <1.0 x 10e9 /L | - |
| | 10e9 /L | 10e9 /L | 10e9 /L | | |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in number of white blo | od cells in a blood specimen. | | - |
| Investigations - Other, specify | Asymptomatic or mild | Moderate; minimal, local or | Severe or medically significant | Life-threatening consequences; | Death |
| | symptoms; clinical or diagnostic | noninvasive intervention | but not immediately life- | urgent Intervention Indicated | |
| | observations only; intervention | Indicated; limiting age- | threatening; hospitalization or | | |
| | not indicated | appropriate instrumental ADL | prolongation of existing | | |
| | | | hospitalization indicated; | | |
| | 1 | I | disabiling; limiting self care ADL | | I |

# 16.4 Appendix 4: FACIT-F Scoring Guidelines (version 4)

Instructions:\*

- 1. Record answers in "item response" column. If missing, mark with an X
- 2. Perform reversals as indicated, and sum individual items to obtain a score.
- 3. Multiply the sum of the item scores by the number of items in the subscale, then divide by the

number of items answered. This produces the subscale score.

- 4. Add subscale scores to derive total scores (TOI, FACT-G & FACIT-F).
- 5. The higher the score, the better the QOL.

| Subscale | Item Code | Reverse item? | Item response | Item Score |
|-------------------|-----------|---------------|---------------|------------|
| PHYSICAL | GP1<br>= | 4 | | |
| WELL-BEING | GP2<br>= | 4 | | |
| (PWB) | GP3<br>= | 4 | | |
| Score range: 0-28 | GP4<br>= | 4 | - | |
| <b>3</b> | GP5<br>= | 4 | | |
| | GP6<br>= | 4 | | |
| | GP7<br>= | 4 | | |

| | | | Sum individual item scores: | | | | |
|---|---|---|---|---|---|---|---|
| | | | Multiply by 7: | | | | |
| = <u>PWB subs</u> | cale score | Divid | le by | number | of | items | answered: |
| SOCIAL/FAMILY | GS1 | 0 | + | | | = | |
| WELL-BEING | GS2 | 0 | + | | | = | |
| (SWB) | GS3 | 0 | + | | | = | |
| | GS4 | 0 | + | | | = | |
| Score range: 0-28 | GS5 | 0 | + | | | = | |
| | GS6 | 0 | + | | | = | |



| | GS7 | | 0 | + | <del></del> | | = | : |
|---|---|---|---|---|---|---|---|---|
| | | | | Sum | individual i | item s | cores: _ | |
| | | | | | Multi | iply b | y 7: | <del></del> |
| =SWB subs | cale score | | Divide | by | number | of | items | answered: |
| EMOTIONAL | GE1 | 4 | - | | | | = | |
| WELL-BEING | GE2 | 0 | + | | | | = | |
| (EWB) | GE3 | 4 | - | | | | = | |
| | GE4 | 4 | - | | | | = | |
| Score range: 0-24 | GE5 | 4 | - | | | | = | |
| | GE6 | 4 | - | | | | = | |
| | | | | Sum | individual i | item s | cores: _ | |
| | | | | | Multi | iply b | y 6: | |
| = <u>EWB subs</u> | cale score | | Divide | by | | | | answered: |
| FUNCTIONAL | GF1 | | 0 | + | | | = | : |
| WELL-BEING | GF2 | | 0 | + | | | | : |
| (FWB) | GF3 | | 0 | + | | | = | : |
| | GF4 | | 0 | + | | | = | |
| Score range: 0-28 | GF5 | | 0 | + | | | = | |
| Georg range: 0-20 | GF6 | | 0 | + | | | = | : |
| | GF7 | | 0 | + | | | = | : |
| | | | | Sum | individual i | item s | cores: _ | |
| | | | | | Multi | iply b | y 7: | |
| =FWB subs | cale score | | Divide | by | number | of | items | answered: |

| <u>Subscale</u> | Item Code | Reverse item? | Item response | <u>ltem</u> |
|-----------------|-----------|---------------|---------------|-------------|
| <u>Score</u> | | | | |



| FATIGUE | HI7 | 4 | - | | = | |
|---|---|---|---|---|---|---|
| SUBSCALE | HI12 | 4 | - | | = | |
| (FS) | An1 | 4 | - | | = | |
| | An2 | 4 | - | | = | |
| Score range: 0-52 | An3 | 4 | - | | = | |
| 30010 Tango. 0 02 | An4 | 4 | - | | = | |
| | An5 | 0 | + | | = | |
| | An7 | 0 | + | | = | |
| | An8 | 4 | - | | = | |
| | An12 | 4 | - | | = | |
| | An14 | 4 | - | | = | |
| | An15 | 4 | - | | = | |
| | An16 | 4 | - | | = | |
| Subscale score To derive a FACIT-F Score range: 0-108 | To derive a FACIT-F Trial Outcome Index (TOI): | | | | | |
| <b>To Derive a FACT-G</b><br>Score range: 0-108 | total score: | | + | | + | + |
| | | | = <b>FA</b> | CT-G Total score | | - |
| | (PWE | score) | (SWB s | score) (EWB score) | (FWB score) | |



| To Der | ive a FA | CIT-F total score: | | | |
|---|---|---|---|---|---|
| Score | range: | 0- | | | |
| | = | +<br>=FACIT-F Total score | _ + | + | + |
| | | (PWB score) (SWB score) | (EWB score) | (FWB score) | ( <b>FS</b> score) |

\*For guidelines on handling missing data and scoring options, please refer to the Administration and Scoring Guidelines in the manual or on-line at www.facit.org.



### 16.5 Appendix 5: Search criteria for adverse events of special interest

Search criteria for AESIs are either MedDRA PT clusters or SMQs. The SMQs and the individual PTs for the PT clusters are provided below. The MedDRA version used for the data coding is v21.0.

#### Infections

Abdominal abscess Acarodermatitis Acute sinusitis

Abdominal hernia Acid fast bacilli infection Adenoiditis

gangrenous Acinetobacter Adenopathy syphilitic

Abdominal infection bacteraemia Adenoviral conjunctivitis
Abdominal Acinetobacter infection

lymphadenopathy

Acinetobacter infection

Adenoviral

haemorrhagic cystitis

Abdominal sepsis positive Adenoviral hepatitis

Abdominal wall abscess Acne pustular

Abdominal wall abscess Acne pustular Adenoviral upper
Abdominal wall infection Acquired respiratory infection

Abortion infected immunodeficiency syndrome Adenovirus encephalomyeloradiculit

Abscess Acrodermatitis chronica is

Abscess bacterial atrophicans Adenovirus infection

Abscess fungal Actinomyces test positive Adenovirus test

Abscess jaw
Abscess limb
Actinomycosis
Actinomycotic
abdominal infection
Adenovirus test positive
Adiponectin increased
Administration site

Abscess neck
Actinomycotic
Abscess of external
Actinomycotic
pulmonary infection
Administration site

auditory meatus

Actinomycotic skin

Abscess of eyelid

Actinomycotic skin

Administration site

Abscess of salivary

Acute endocarditis

Acute endocarditis

gland Acute focal bacterial Adrenal gland abscess
Abscess oral nephritis Adrenal gland

Abscess rupture

Abscess rupture

Acute haemorrhagic

Conjunctivitis

Adrenal gland

tuberculosis

Adrenalitis

Abscess sweat gland Acute hepatitis B Aeromonas infection

Acanthamoeba infection Acute hepatitis C Aeromonas test positive

Acanthamoeba keratitis Acute HIV infection African trypanosomiasis

Acariasis

Acute pulmonary

AlDS cholangiopathy
histoplasmosis

ALX0061-C203 – Statistical Analysis Plan – Final 1.0 – 4 OCT 2018
Anal abscess


Application site AIDS related complex Angina gangrenous folliculitis AIDS related Angiostrongylus complication infection Application site infection AIDS retinopathy Anicteric leptospirosis Application site pustules

Air-borne transmission **Anisakiasis** Arachnoiditis Alcaligenes infection Anogenital warts Arboviral infection Allescheriosis Anorectal cellulitis Arbovirus test positive Alopecia syphilitic Anorectal human Arenaviral haemorrhagic

papilloma virus infection fever Alpha haemolytic streptococcal infection Anorectal infection Arenavirus test positive Alphaviral infection Anorectal infection Argentine haemorrhagic

bacterial fever Alphavirus test Anthrax Arteriosclerotic

Alphavirus test positive gangrene Anthrax sepsis Alternaria infection

Arteriovenous fistula site Antifungal treatment Alveolar osteitis infection

Antimicrobial American Arteriovenous graft site susceptibility test trypanosomiasis abscess

Antimicrobial Amniotic cavity infection Arteriovenous graft site susceptibility test infection Amniotic infection intermediate

syndrome of Blane Arteritis infective Antimicrobial Amoeba test susceptibility test Arthritis bacterial

resistant Amoeba test positive Arthritis fungal Antimicrobial Amoebiasis

Arthritis gonococcal susceptibility test Amoebic brain abscess Arthritis helminthic sensitive

Amoebic colitis Arthritis infective Aortic aneurysm syphilitic Amoebic dysentery Arthritis reactive Aortitis salmonella Amoebic lung abscess Arthritis rubella

Aortitis syphilitic Amoebic skin ulcer Arthritis salmonella Aphthovirus test positive

Apical granuloma Anal candidiasis Arthropod infestation

Appendiceal abscess Anal chlamydia infection Arthropod-borne disease

**Appendicitis** Anal fistula infection Appendicitis perforated **Ascariasis** Anal fungal infection Application site abscess Aspergilloma Anal infection

Application site cellulitis Aspergillosis oral Anal tinea

Arthritis viral


Aspergillus infection Bacterial disease carrier Bifidobacterium infection Aspergillus test Bacterial food poisoning Bifidobacterium test positive Aspergillus test positive Bacterial infection Bile culture Astrovirus test positive **Bacterial** iritis Bile culture positive Asymptomatic Bacterial labyrinthitis bacteriuria Biliary abscess Bacterial pericarditis Asymptomatic HIV Biliary sepsis Bacterial prostatitis infection Biliary tract infection Bacterial pyelonephritis Asymptomatic viral Biliary tract infection Bacterial rhinitis hepatitis bacterial Bacterial sepsis Atypical mycobacterial Biliary tract infection infection Bacterial test cryptosporidial Atypical mycobacterial Bacterial test positive Biliary tract infection lower respiratory tract fungal Bacterial toxaemia infection Biliary tract infection Bacterial tracheitis Atypical mycobacterial helminthic lymphadenitis Bacterial translocation Biliary tract infection Atypical mycobacterial Bacterial vaginosis viral pneumonia Bacterial vulvovaginitis BK virus infection Atypical mycobacterium Bacteriuria pericarditis Black piedra Bacteriuria in pregnancy Atypical mycobacterium Bladder candidiasis test positive **Bacteroides** Bladder diverticulitis bacteraemia Atypical pneumonia Blastocystis infection Bacteroides infection Avian influenza Blastomycosis Bacteroides test positive Babesiosis **Blebitis** Balamuthia infection Bacillary angiomatosis Blepharitis Balanitis candida Bacillus bacteraemia Blister infected Balanoposthitis Bacillus infection Blood bactericidal Balanoposthitis infective Bacillus test positive activity Balantidiasis Blood beta-D-glucan Bacteraemia abnormal Bartholin's abscess **Bacterascites** Blood beta-D-glucan Bartonella test positive Bacterial abscess decreased central nervous system Bartonellosis Blood beta-D-glucan Bacterial allergy Bed bug infestation increased Bacterial dacryocystitis Beta haemolytic Blood culture streptococcal infection Bacterial diarrhoea

Blood culture positive


Blood HIV RNA Bronchitis haemophilus Campylobacter gastroenteritis

Blood HIV RNA below assay limit Bronchitis

Campylobacter gastroenteritis

Campylobacter infection

Blood HIV RNA pneumococcal Campylobacter sepsis decreased Bronchitis viral Campylobacter test

Blood HIV RNA Bronchoalveolar lavage abnormal positive Candida cervicitis

Body tinea Bronchopulmonary Candida

Bolivian haemorrhagic aspergillosis endophthalmitis fever

Bronchopulmonary Candida infection

Bone abscess aspergillosis allergic Candida nappy rash

Bone tuberculosis Bronchoscopy abnormal

Borderline leprosy

Brucella sepsis

Candida osteomyelitis

Candida pneumonia

Bordetella infection Brucella test Candida retinitis

Bordetella test Brucella test positive Candida sepsis

Bordetella test positive Brucellosis Candida test

Borrelia infection Bubonic plague Candida test positive

Borrelia test
Bulbar poliomyelitis
Candiduria
Borrelia test positive
Bullous impetigo
Capillariasis
Botryomycosis
Burkholderia cepacia

Bottyonycosis Burkholderia cepacia Capillaritis

Complex infection Capnocytophaga

Boutonneuse fever

Burkholderia cepacia complex sepsis

Burkholderia cepacia infection

Bovine pustular stomatitis virus infection Burkholderia gladioli positive Capnocytophaga test

Bovine tuberculosis infection infection Carbuncle

Brain abscess

Burkholderia mallei

Brain empyema

Brain empyema

Cardiac granuloma

Cardiac infection

Cardiac infection

Breast abscess Burkholderia Cardiac valve abscess

Breast cellulitis pseudomallei infection Cardiac valve

Breast discharge infected Burkholderia test vegetation positive Cardiovascular syphilis

Bronchiectasis Burn infection Carditis

Bronchiolitis

Bursitis infective
Cat scratch disease
Bursitis infective
staphylococcal
Catheter culture

Bronchitis bacterial Calicivirus test positive

Bronchitis fungal Catheter culture positive

Catheter site abscess

ALX0061-C203 – Statistical Analysis Plan – Final 1.0 – 4 OCT 2018 Page 75/111


Catheter site cellulitis Cervicitis gonococcal Chronic recurrent multifocal osteomyelitis Catheter site infection Cervicitis human papilloma virus Chronic sinusitis Catheter site pustule Cervicitis mycoplasmal Chronic tonsillitis Catheter site warmth Cervicitis streptococcal Citrobacter infection Cavernous sinus thrombosis Cervicitis trichomonal Citrobacter sepsis Cellulitis Cervix warts Citrobacter test positive Cellulitis enterococcal Cestode infection Clitoris abscess Chancroid Clonorchiasis Cellulitis gangrenous Cellulitis laryngeal Chest wall abscess Clostridial infection Cellulitis of male Chikungunya virus Clostridial sepsis external genital organ infection Clostridium bacteraemia Cellulitis orbital Chlamydia test Clostridium colitis Cellulitis pasteurella Chlamydia test positive Clostridium difficile Cellulitis pharyngeal Chlamydial cervicitis colitis Cellulitis staphylococcal Chlamydial infection Clostridium difficile infection Cellulitis streptococcal Chlamydial pelvic inflammatory disease Clostridium test Central nervous system Cholangitis infective abscess Clostridium test positive Central nervous system Cholecystitis infective CNS ventriculitis enteroviral infection Cholera Coccidioides Central nervous system encephalitis Cholesteatoma fungal infection Coccidioidomycosis Cholesterol granuloma Central nervous system Colitis herpes Choriomeningitis infection lymphocytic Colon gangrene Central nervous system Chorioretinitis Colonic abscess inflammation Choroid tubercles Colorado tick fever Central nervous system viral infection Choroiditis Colorado tick fever virus test positive Cerebral aneurysm Chromoblastomycosis ruptured syphilitic Colostomy infection Chronic gastritis Cerebral aspergillosis Community acquired Chronic hepatitis Cerebral fungal infection infection Chronic hepatitis B Condyloma latum Cerebral malaria Chronic hepatitis C Congenital condyloma Cerebral septic infarct

Cerebral toxoplasmosis

Chronic pulmonary

histoplasmosis


Congenital cytomegalovirus infection

Congenital hepatitis B

infection

Congenital herpes simplex infection

Congenital HIV infection

Congenital infection

Congenital malaria

Congenital pneumonia

Congenital rubella

infection

Congenital syphilis

Congenital syphilitic

encephalitis

Congenital syphilitic

meningitis

Congenital syphilitic osteochondritis

Congenital toxoplasmosis

Congenital tuberculosis

Congenital varicella

infection

Congo-Crimean haemorrhagic fever

Conjunctivitis

Conjunctivitis bacterial

Conjunctivitis chlamydial

Conjunctivitis

gonococcal neonatal

Conjunctivitis tuberculous

Conjunctivitis viral

Corneal abscess

Corneal endotheliitis

Corneal infection

Corona virus infection

Coronavirus test

positive

Corynebacterium

infection

Corynebacterium sepsis

Corynebacterium test

Corynebacterium test

positive

Cow pox

Coxiella infection

Coxiella test positive

Coxsackie carditis

Coxsackie endocarditis

Coxsackie myocarditis

Coxsackie pericarditis

Coxsackie viral disease

of the newborn

Coxsackie viral infection

Coxsackie virus test

Coxsackie virus test

positive

Cranial nerve infection

Creutzfeldt-Jakob

disease

Cronobacter

bacteraemia

Cronobacter infection

Cronobacter necrotising

enterocolitis

Cronobacter test

positive

Cross infection

Croup infectious

Cryptococcal cutaneous

infection

Cryptococcal fungaemia

Cryptococcosis

Cryptococcus test

Cryptococcus test

positive

Cryptosporidiosis

infection

CSF culture

CSF culture positive

CSF immunoglobulin G

index

CSF

leukocyte/erythrocyte

ratio

CSF

leukocyte/erythrocyte

ratio increased

CSF measles antibody

positive

CSF virus identified

CSF virus no organisms

observed

Culture

Culture cervix

Culture cervix positive

Culture positive

Culture stool

Culture stool positive

Culture throat

Culture throat positive

Culture tissue specimen

Culture tissue specimen

positive

Culture urine

Culture urine positive

Culture wound

Culture wound positive

Cutaneous anthrax


Cutaneous Cytomegalovirus Dental fistula coccidioidomycosis gastroenteritis Dental gangrene Cutaneous larva Cytomegalovirus Dermatitis infected gastrointestinal infection migrans Dermatomyositis Cutaneous Cytomegalovirus leishmaniasis hepatitis Dermatophytosis Dermo-hypodermitis Cutaneous Cytomegalovirus sporotrichosis infection Device related infection Cutaneous tuberculosis Cytomegalovirus Device related sepsis mononucleosis Cyclitis Diabetic foot infection Cytomegalovirus Cyclosporidium infection Diabetic gangrene mucocutaneous ulcer Cystitis Diaphragmatic hernia Cytomegalovirus Cystitis bacterial myelomeningoradiculitis gangrenous Diarrhoea infectious Cystitis erosive Cytomegalovirus myocarditis Diarrhoea infectious Cystitis escherichia neonatal Cytomegalovirus Cystitis glandularis oesophagitis Diphtheria Cystitis gonococcal Cytomegalovirus Diphtheria carrier Cystitis haemorrhagic pancreatitis Diphyllobothriasis Cystitis helminthic Cytomegalovirus Direct infection pericarditis Cystitis interstitial transmission Cytomegalovirus Cystitis klebsiella Disseminated syndrome Cystitis noninfective cryptococcosis Cytomegalovirus test Cystitis pseudomonal Disseminated Cytomegalovirus test cytomegaloviral Cystitis radiation positive infection Cystitis ulcerative Cytomegalovirus urinary Disseminated tract infection Cystitis viral tuberculosis Cytomegalovirus Cytomegalovirus Diverticulitis viraemia chorioretinitis Douglas' abscess Dacryoadenitis acquired Cytomegalovirus colitis Dracunculiasis Dacryocanaliculitis Cytomegalovirus Dural abscess duodenitis **Dacryocystitis** Dysentery Cytomegalovirus Deltaretrovirus test enteritis Ear infection positive Ear infection bacterial Cytomegalovirus **Demodicidosis** enterocolitis

Cytomegalovirus

gastritis

Dengue fever

Dental caries

Ear infection fungal


Ear infection Encephalitis brain stem Endocarditis staphylococcal Encephalitis california Encephalitis california

Ear infection viral Encephalitis Endocarditis gonococcal

Ear lobe infection cytomegalovirus Endocarditis
Ear tuberculosis Encephalitis eastern Endocarditis

Ebola disease equine Endocarditis helminthic

Ebola Reston virus Encephalitis enteroviral Endocarditis histoplasma Encephalitis fungal

Ebola virus test positive Encephalitis Endocarditis meningococcal

Echinococciasis

Echo virus infection

Encephalitis influenzal

Endocarditis pseudomonal

Echovirus test Encephalitis Japanese Endocarditis Q fever

Echovirus test positive Encephalitis lethargica Endocarditis rheumatic

Ecthyma Encephalitis Eczema herpeticum Encephalitis staphylococcal

Eczema impetiginous Encephalitis mumps Endocarditis syphilitic Endocarditis viral

Eczema infected Encephalitis post immunisation Endometritis

Eczema vaccinatum Endometritis

Ehrlichia test

Encephalitis post
varicella

Endometritis bacterial

Ehrlichia test positive Encephalitis protozoal Endometritis decidual

Elephantiasis nostras

Encephalitis protozoal

Endometritis gonococcal

Encephalitis rickettsial

verrucosa Encephalitis rickettsiai Endophthalmitis
Embolic pneumonia Encephalitis toxic Endotoxaemia

Empedobacter brevis Encephalitis venezuelan equine Endotoxic shock

Empedobacter test

Encephalitis viral

Enteritis infectious

Enteritis necroticans

positive Encephalitis western equine Enterobacter

cholecystitis Encephalomyelitis bacteraemia

Enterobacter infection

Emphysematous rubella Enterobacter pyelonephritis End stage AIDS Enterobacter

Empyema Endemic syphilis Enterobacter sepsis

Encephalitis Endocarditis Enterobacter test

Encephalitis allergic Endocarditis bacterial Enterobacter

Encephalitis australia Endocarditis candida positive

Enterobacter tracheobronchitis

ALX0061-C203 – Statistical Analysis Plan – Final 1.0 – 4 OCT 2018 Page 79/111


Enterobiasis Epiglottitis obstructive Escherichia urinary tract

Enterococcal Epstein-Barr viraemia infection

bacteraemia Epstein-Barr virus Escherichia vaginitis

Enterococcal infection antibody Eubacterium infection
Enterococcal sepsis Epstein-Barr virus Exanthema subitum

Enterococcus test antibody positive Exserohilum infection

positive Epstein-Barr virus External ear cellulitis
Enterocolitis AIDS External ear cellulitis

Enterocolitis AIDS

Enterocolitis bacterial

Extradural abscess

Enterocolitis fungal associated lymphoma Extrapulmonary tuberculosis

Enterocolitis helminthic associated Eye abscess

Enterocolitis infectious lymphoproliferative Eye infection

disorder Enterocolitis viral Eye infection bacterial

Epstein-Barr virus

Enterovirus infection

Epstein-Barr virus

Eye infection bacterial

Eye infection chlamydial

Enterovirus test Epstein-Barr virus test Eye infection fungal

Enterovirus test positive Epstein-Barr virus test Eye infection

Eosinophilia myalgia positive gonococcal

syndrome Erosive balanitis Eye infection helminthic

Eosinophilic cystitis Eruptive Eye infection intraocular

Ependymitis pseudoangiomatosis Eye infection staphylococcal

Epidemic polyarthritis Erysipeloid Eye infection syphilitic

Epidemic typhus Erysipelothrix infection Eye infection toxoplasmal

Erysipeiotinix test positive Eye infection viral

Epididymitis Erythema induratum Eyelid boil

Epididymitis Erythema infectiosum Eyelid folliculitis blastomyces Erythema migrans Eyelid infection

Epididymitis mumps Erythrasma Faecal-oral transmission

Epididymitis tuberculous Escherichia of infection

Epididymitis bacteraemia Fallopian tube abscess

ureaplasmalEscherichia infectionFascial infectionEpididymo-orchitisEscherichiaFascioliasisgonococcalpyelonephritisFasciolopsiasisEpiglottitisEscherichia sepsisFasciolopsiasis

Epiglottitis Febrile infection
Epiglottitis haemophilus Escherichia test positive


Female genital tract tuberculosis

luberculosis

Femoral hernia gangrenous

**Filariasis** 

Filariasis lymphatic

Filovirus infection

Filovirus test positive

Flavivirus infection

Flavivirus test positive

Flavobacterium infection

Flavobacterium test

positive

Flea infestation

**Folliculitis** 

Foot and mouth disease

Francisella test positive

Fungaemia

Fungal abscess central

nervous system

Fungal cystitis

Fungal endocarditis

Fungal infection

Fungal labyrinthitis

Fungal oesophagitis

Fungal paronychia Fungal peritonitis

Fungal retinitis

Fungal rhinitis

Fungal sepsis

Fungal skin infection

Fungal test

Fungal test positive

Fungal tracheitis

Fungating wound

Funisitis

**Furuncle** 

Fusarium infection

Fusobacterium test

Fusobacterium infection

positive

Gallbladder abscess

Gallbladder empyema

Gangrene

Gangrene neonatal

Gangrenous balanitis

Gardnerella infection

Gardnerella test positive

Gas gangrene

Gastric infection

Gastric ulcer

helicobacter

Gastritis bacterial

Gastritis fungal

Gastritis helminthic

Gastritis herpes

Gastritis viral

Gastroenteritis

Gastroenteritis adenovirus

Gastroenteritis

aerobacter

Gastroenteritis aeromonas

Gastroenteritis astroviral

Gastroenteritis bacillus

Castrocritoritis bacillas

Gastroenteritis bacterial

Gastroenteritis caliciviral

Gastroenteritis

clostridial

Gastroenteritis cryptococcal

Gastroenteritis

cryptosporidial

Gastroenteritis enteroviral

Gastroenteritis

Escherichia coli

Gastroenteritis norovirus

Gastroenteritis

paracolon bacillus

Gastroenteritis proteus

Gastroenteritis

pseudomonas

Gastroenteritis rotavirus

Gastroenteritis

salmonella Gastroenteritis

sapovirus

Gastroenteritis shigella

Gastroenteritis

staphylococcal

Gastroenteritis vibrio

Gastroenteritis viral

Gastroenteritis yersinia

Gastrointestinal anthrax

Gastrointestinal

bacterial infection

Gastrointestinal

bacterial overgrowth

Gastrointestinal

candidiasis

Gastrointestinal fungal

infection

Gastrointestinal

gangrene

Gastrointestinal

infection


Gastrointestinal Gerstmann Straussler Haemophilus sepsis mucosal necrosis Scheinker syndrome Haemophilus test Gastrointestinal Gianotti-Crosti positive necrosis syndrome Haemorrhagic fever Gastrointestinal Giardia test Haemorrhagic fever with protozoal infection Giardia test positive renal syndrome Gastrointestinal viral Giardiasis Haemorrhoid infection infection Gingival abscess Hand-foot-and-mouth Generalised vaccinia disease Gingivitis Genital abscess Hantaviral infection Gliosis Genital candidiasis Hantavirus pulmonary Gnathostomiasis Genital herpes infection Gonococcal pelvic Genital herpes simplex Hantavirus test positive inflammatory disease Genital herpes zoster **HBV-DNA** polymerase Gonorrhoea increased Genital infection Gradenigo's syndrome Helicobacter gastritis Genital infection Graft infection bacterial Helicobacter infection Gram stain Genital infection female Helicobacter sepsis Gram stain positive Genital infection fungal Helicobacter test Granuloma inquinale Genital infection Helicobacter test Granulomatous helminthic positive dermatitis Genital infection male Helminthic infection Granulomatous liver Genital infection viral Henipavirus test positive disease Genital tract Hepatic amoebiasis Granulomatous inflammation pneumonitis Hepatic candidiasis Genitourinary chlamydia Groin abscess Hepatic cyst infection infection Groin infection Hepatic echinococciasis Genitourinary tract gonococcal infection Group B streptococcus Hepatic infection neonatal sepsis Genitourinary tract Hepatic infection Guillain-Barre syndrome bacterial infection Gynaecological Hepatic infection fungal Genotype drug resistance test chlamydia infection Hepatic infection helminthic H1N1 influenza Genotype drug resistance test abnormal Haematoma infection Hepatic infiltration eosinophilic Genotype drug Haemophilus

bacteraemia

Haemophilus infection

resistance test positive

Geotrichum infection

Hepatic necrosis

Hepatitis


| Hepatitis A | Hepatitis B e antigen | Hepatitis D antigen positive |
|---|---|---|
| Hepatitis A antibody | Hepatitis B e antigen | • |
| Hepatitis A antibody | positive D aurita a | Hepatitis D RNA |
| abnormal Hepatitis A antibody | Hepatitis B surface antibody | Hepatitis D RNA positive |
| positive | Hepatitis B surface | Hepatitis D virus test |
| Hepatitis A antigen positive | antibody positive Hepatitis B surface | Hepatitis D virus test positive |
| Hepatitis A virus test | antigen | Hepatitis E |
| Hepatitis A virus test positive | Hepatitis B surface antigen positive | Hepatitis E antibody |
| Hepatitis acute | Hepatitis B virus test | Hepatitis E antibody abnormal |
| Hepatitis B | Hepatitis B virus test | Hepatitis E antibody |
| • | positive | positive |
| Hepatitis B antibody | Hepatitis C | Hepatitis E antigen |
| Hepatitis B antibody abnormal | Hepatitis C antibody | Hepatitis E antigen |
| Hepatitis B antibody | Hepatitis C antibody | positive |
| positive | positive | Hepatitis E virus test |
| Hepatitis B antigen | Hepatitis C RNA | positive |
| Hepatitis B antigen<br>positive | Hepatitis C RNA decreased | Hepatitis F |
| | | Hepatitis fulminant |
| Hepatitis B core | Hepatitis C RNA fluctuation | Hepatitis G |
| Intibody<br>Hepatitis B core<br>Intibody positive | Hepatitis C RNA | Hepatitis H |
| | increased | Hepatitis infectious |
| Hepatitis B core antigen | Hepatitis C RNA | mononucleosis |
| Hepatitis B core antigen | positive | Hepatitis mumps |
| positive | Hepatitis C virus test | Hepatitis neonatal |
| Hepatitis B DNA assay | Hepatitis C virus test | Hepatitis non-A non-B |
| Hepatitis B DNA assay | positive | Hepatitis non-A non-B |
| positive | Hepatitis chronic active | non-C |
| Hepatitis B DNA decreased | Hepatitis chronic persistent | Hepatitis post transfusion |
| Hepatitis B DNA | Hepatitis D | Hepatitis syphilitic |
| increased | Hepatitis D antibody | Hepatitis toxoplasmal |
| Hepatitis B e antibody | Hepatitis D antibody | Hepatitis viral |
| Hepatitis B e antibody | positive | Hepatitis viral |
| positive | Hepatitis D antigen | Hepatitis viral test |


Herpes simplex test HIV associated Hepatitis viral test positive nephropathy Herpes simplex test Hepatitis viruspositive HIV cardiomyopathy associated nephropathy Herpes simplex virus HIV carrier Hepatobiliary infection conjunctivitis neonatal HIV enteropathy Hepatosplenic Herpes simplex visceral HIV infection candidiasis Herpes virus infection HIV infection CDC Hernia gangrenous Herpes zoster category A Herpangina Herpes zoster HIV infection CDC Herpes dermatitis cutaneous disseminated category B Herpes oesophagitis Herpes zoster HIV infection CDC disseminated category C Herpes ophthalmic Herpes zoster infection HIV infection CDC Herpes pharyngitis neurological Group I Herpes sepsis Herpes zoster HIV infection CDC Herpes simplex meningitis Group II Herpes simplex colitis Herpes zoster **HIV infection CDC** meningoencephalitis Group III Herpes simplex encephalitis Herpes zoster **HIV infection CDC** meningomyelitis group IV Herpes simplex gastritis **HIV infection CDC** Herpes zoster Herpes simplex hepatitis Group IV subgroup A necrotising retinopathy Herpes simplex **HIV infection CDC** Herpes zoster oticus meningitis Group IV subgroup B Herpes zoster Herpes simplex pharyngitis **HIV infection CDC** meningoencephalitis Group IV subgroup C1 Heterophyiasis Herpes simplex HIV infection CDC meningomyelitis Hirudiniasis Group IV subgroup C2

Histiocytic necrotising

necrotising retinopathy

Herpes simplex
oesophagitis

Histoplasmosis
cutaneous
externa

Histoplasmosis
disseminated

Herpes simplex

pharyngitis

HIV antibody
Herpes simplex
pneumonia
HIV antibody positive
HIV antipody positive
HIV antipody

Herpes simplex sepsis

HIV antigen positive

HIV infection CDC

**HIV infection CDC** 

HIV infection WHO

HIV infection WHO

HIV infection WHO

clinical stage I

clinical stage II

clinical stage III

Group IV subgroup D

Group IV subgroup E

## Áblynx


HIV infection WHO Human polyomavirus Induced abortion clinical stage IV infection infection HIV peripheral Human rhinovirus test Infantile septic granulomatosis neuropathy positive HIV test Human T-cell Infected bite lymphocytic virus type II Infected bunion HIV test positive infection HIV tropism test Infected cyst Human T-cell HIV wasting syndrome lymphotropic virus Infected dermal cyst infection HIV-associated Infected fistula neurocognitive disorder Human T-cell Infected lymphocele lymphotropic virus type I Hookworm infection Infected naevus infection Hordeolum Infected neoplasm Hydrocele male infected HTLV test positive Infected seroma Hymenolepiasis HTLV-1 carrier Infected skin ulcer Hypopyon HTLV-1 test positive Infected varicose vein latrogenic infection HTLV-2 test positive Infection lleal gangrene Human anaplasmosis Infection in an Immune reconstitution Human ehrlichiosis inflammatory syndrome host associated tuberculosis Human herpes virus 6 serology Infection masked **Impetigo** Human herpes virus 6 Infection parasitic Implant site abscess serology positive Infection protozoal Implant site cellulitis Human herpes virus 8 Infection reactivation Implant site infection test positive Infection susceptibility Implant site pustules Human herpesvirus 6 increased infection Incision site abscess Human herpesvirus 7 Incision site cellulitis via personal contact infection Incisional hernia

Human herpesvirus 8 infection

Human

immunodeficiency virus

transmission

Human papilloma virus

test

Human papilloma virus

test positive

gangrenous

Inclusion body myositis

Inclusion conjunctivitis

Inclusion conjunctivitis

neonatal

Indeterminate leprosy

Indirect infection transmission

immunocompromised

Infection transmission

Infection via vaccinee

Infectious colitis

Infectious crystalline

keratopathy

Infectious disease

carrier

Infectious iridocyclitis

Infectious mononucleosis


Infectious pleural Influenza C virus test Joint abscess effusion positive Joint tuberculosis Infectious thyroiditis Influenza virus test Kaposi's sarcoma AIDS Infective aneurysm Influenza virus test related positive Infective aortitis Kaposi's varicelliform Infusion site abscess eruption Infective chondritis Kawasaki's disease Infusion site cellulitis Infective corneal ulcer Infusion site infection Keratitis Infective episcleritis Keratitis bacterial Infusion site pustule Infective exacerbation of bronchiectasis Inguinal hernia Keratitis fungal gangrenous Infective exacerbation of Keratitis interstitial chronic obstructive Injection site abscess Keratitis viral airways disease Injection site cellulitis Keratoconjunctivitis Infective Injection site infection measles gastroduodenitis Injection site joint Keratosis gonococcal Infective glossitis infection Kerion Infective iritis Injection site pustule Kidney infection Infective mesenteric Instillation site abscess Klebsiella bacteraemia panniculitis Instillation site infection Klebsiella infection Infective myositis Instillation site pustules Infective periostitis Klebsiella sepsis Intervertebral discitis Klebsiella test positive Infective pulmonary Intestinal fistula infection exacerbation of cystic Kuru fibrosis Intestinal gangrene Kyasanur Forest Infective spondylitis disease Intestinal tuberculosis Infective tenosynovitis Intrauterine infection Labyrinthitis Infective thrombosis Iridocyclitis Lacrimal sac cellulitis Infective uveitis **Iritis** Lactobacillus infection Infestation Isosporiasis Lactobacillus test Influenza positive Japanese spotted fever Influenza A virus test Laryngitis JC polyomavirus test Influenza A virus test Laryngitis bacterial JC polyomavirus test positive positive Laryngitis fungal Influenza B virus test JC virus granule cell Laryngitis viral Influenza B virus test neuronopathy Laryngotracheitis positive JC virus infection obstructive

Jejunal gangrene

Lassa fever


Latent syphilis Lung abscess Mastoid empyema Latent tuberculosis Lung infection Mastoiditis Legionella infection Lung infection Measles pseudomonal Legionella test Measles antibody Lupus encephalitis Legionella test positive Measles antibody Lupus vulgaris positive Leishmaniasis Lyme disease Measles post vaccine Lemierre syndrome Lymph gland infection Mediastinal abscess Lentivirus test positive Mediastinitis Lymph node abscess Lepromatous leprosy Lymph node Meibomian gland Leprosy tuberculosis discharge Leptospira test positive Meibomianitis Lymphadenitis bacterial Leptospirosis Lymphadenitis fungal Meningitis Leptotrichia infection Lymphadenitis Meningitis aseptic Leuconostoc infection helminthic Meningitis aspergillus Lice infestation Lymphadenitis viral Meningitis bacterial Ligneous conjunctivitis Lymphangitis Meningitis borrelia Lineal gingival erythema Lymphogranuloma Meningitis candida venereum Lip infection Meningitis chemical Lyssavirus test positive Listeria encephalitis Meningitis coccidioides Malaria Listeria sepsis Meningitis coxsackie Malaria antibody test Listeria test positive viral Malaria antibody test Listeriosis Meningitis cronobacter positive Liver abscess Meningitis cryptococcal Malarial myocarditis Localised infection Meningitis echo viral Male genital tract Lochial infection Meningitis enterococcal tuberculosis Louping ill Malignant syphilis Meningitis enteroviral Lower respiratory tract Marburg disease Meningitis eosinophilic infection Marburg virus test Meningitis exserohilum Lower respiratory tract positive Meningitis fungal infection bacterial Mastitis Meningitis gonococcal Lower respiratory tract Mastitis bacterial infection fungal Meningitis haemophilus Mastitis fungal Lower respiratory tract Meningitis herpes infection viral Mastitis postpartum Meningitis histoplasma Ludwig angina Mastoid abscess

ALX0061-C203 – Statistical Analysis Plan – Final 1.0 – 4 OCT 2018

Meningitis leptospiral


Meningitis listeria

Meningitis meningococcal

Meningitis mumps Meningitis neonatal

Meningitis pneumococcal

Meningitis salmonella

Meningitis staphylococcal

Meningitis streptococcal

Meningitis toxoplasmal

Meningitis trypanosomal

Meningitis tuberculous

Meningitis viral

Meningococcal bacteraemia

Meningococcal carditis

Meningococcal infection

Meningococcal sepsis

Meningoencephalitis

amoebic

Meningoencephalitis

bacterial

Meningoencephalitis

helminthic

Meningoencephalitis herpes simplex neonatal

Meningoencephalitis

herpetic

Meningoencephalitis

viral

Meningomyelitis herpes

Mesenteric abscess

Mesenteritis

Metagonimiasis

Metapneumovirus

infection

Methylobacterium

infection

Microbiology test

Microbiology test

abnormal

Micrococcal sepsis

Micrococcus infection

Micrococcus test

positive

Microsporidia infection

Microsporum infection

Middle ear operation

Middle East respiratory

syndrome

Miliary pneumonia

Milker's nodules

Minimum inhibitory concentration

Molluscipoxvirus test

positive

Molluscum contagiosum

Monkeypox

Mononucleosis heterophile test

Mononucleosis

heterophile test positive

Mononucleosis

syndrome

Moraxella infection

Moraxella test positive

Morbillivirus test positive

Morganella infection

Morganella test positive

Mucocutaneous

candidiasis

Mucocutaneous leishmaniasis

Mucormycosis

Mucosal infection

Mumps

Mumps antibody test

Mumps antibody test

positive

Mumps deafness

Murine typhus

Murray Valley encephalitis

Muscle abscess

Muscular sarcoidosis

Mycetoma mycotic

Mycobacterial disease

carrier

Mycobacterial infection

Mycobacterial peritonitis

Mycobacterium abscessus infection

Mycobacterium avium complex immune

Mycobacterium avium complex infection

restoration disease

Mycobacterium chelonae infection

Mycobacterium fortuitum infection

Mycobacterium kansasii

infection

Mycobacterium leprae

test positive

Mycobacterium marinum infection

Mycobacterium test


Mycobacterium test positive

Mycobacterium tuberculosis complex

Mycobacterium tuberculosis complex test positive

test

Mycobacterium ulcerans infection

Mycoplasma genitalium infection

Mycoplasma infection

Mycoplasma test

Mycoplasma test positive

Mycoplasmal postabortal fever

Mycoplasmal postpartum fever

Mycotic corneal ulcer

Mycotic endophthalmitis

Mycotoxicosis

Myelitis

Myelitis transverse

Myiasis

Myocardiac abscess

Myocarditis

Myocarditis bacterial

Myocarditis helminthic

Myocarditis infectious

Myocarditis meningococcal

Myocarditis mycotic

Myocarditis post

infection

Myocarditis septic

Myocarditis syphilitic

Myocarditis toxoplasmal

Myometritis Myositis

Myositis ossificans

Myositis-like syndrome

Myringitis

Naegleria infection
Nail bed infection
Nail bed infection

bacterial

Nail bed infection viral

Nail candida

Nail infection

Nairovirus test positive

Nasal abscess

Nasal candidiasis

Nasal discharge discolouration

Nasal herpes

Nasal vestibulitis Nasopharyngitis

Natural killer cell count

Natural killer cell count

decreased

Natural killer cell count

increased

Natural killer T cell

count

Natural killer T cell count decreased

Natural killer T cell count increased

Necrobacillosis

Necrotising fasciitis

Necrotising fasciitis

fungal

Necrotising fasciitis staphylococcal

Necrotising fasciitis streptococcal

Necrotising herpetic

retinopathy

Necrotising myositis Necrotising retinitis Necrotising ulcerative gingivostomatitis

Necrotising ulcerative

periodontitis

Neisseria infection

Neisseria test positive

Nematodiasis

Neonatal candida

infection

Neonatal infection

Neonatal infective

mastitis

Neonatal

mucocutaneous herpes

simplex

Neonatal pneumonia

Neuroborreliosis

Neurocryptococcosis Neurocysticercosis

Neurological infection
Neurosarcoidosis

Neurosyphilis

Neutropenic infection Neutropenic sepsis Newcastle disease

Newcastle disease virus

test positive


Oral candidiasis Nipah virus infection Osteomyelitis salmonella Nipple infection Oral fungal infection Osteomyelitis viral Nipple inflammation Oral hairy leukoplakia Otitis externa Oral helminthic infection Nocardia sepsis Otitis externa bacterial Nocardia test positive Oral herpes Otitis externa candida Nocardiosis Oral infection Otitis externa fungal Norovirus test positive Oral pustule Otitis externa viral North Asian tick typhus Oral viral infection Otitis media Nosocomial infection Orbital infection Otitis media acute Obstetric infection Orbivirus infection Otitis media bacterial Oculoglandular Orbivirus test positive Otitis media chronic syndrome **Orchitis** Oesophageal Otitis media fungal Orchitis mumps candidiasis Otitis media Orf Oesophageal infection haemophilus Organic dust toxic Oesophageal Otitis media moraxella syndrome tuberculosis Otitis media post Oro-pharyngeal Oesophagitis bacterial measles aspergillosis **Omphalitis** Otitis media viral Oropharyngeal Omsk haemorrhagic candidiasis Otorrhoea fever Oropharyngeal Otosalpingitis Onchocerciasis gonococcal infection Ovarian abscess Oncovirus test positive Oropharyngitis fungal Ovarian bacterial Onychomycosis Orthobunyavirus test infection positive **Oophoritis** Overgrowth bacterial Orthopox virus infection Ophthalmia neonatorum **Pachymeningitis** Orthopoxvirus test Pancreas infection Ophthalmic herpes positive simplex Pancreatic abscess Osler's nodes Ophthalmic herpes Pancreatitis bacterial zoster Osteomyelitis Pancreatitis fungal **Opisthorchiasis** Osteomyelitis acute Pancreatitis helminthic Opportunistic infection Osteomyelitis bacterial Pancreatitis mumps Osteomyelitis Optic neuritis Pancreatitis viral blastomyces Optic neuritis

Osteomyelitis chronic

Osteomyelitis fungal

meningococcal

Oral bacterial infection

**Panencephalitis** 

**Panophthalmitis** 

Parasitic oesophagitis


Pantoea agglomerans Parasitic test Peptostreptococcus test infection positive Parasitic test positive Pantoea agglomerans Perianal streptococcal Paraspinal abscess test positive infection Parathyroid gland Papilloma viral infection Pericarditis amoebic abscess **Paracoccidioides** Pericarditis fungal Paratyphoid fever infection Pericarditis gonococcal Paravaccinia **Paragonimiasis** Pericarditis helminthic Paravaccinia virus test Parainfluenzae viral Pericarditis histoplasma positive laryngotracheobronchitis Pericarditis infective Parechovirus infection Parainfluenzae virus infection Paronychia Pericarditis meningococcal Parametric abscess Parophthalmia Pericarditis Parotid abscess **Parametritis** mycoplasmal **Parotitis** Paraoesophageal Pericarditis rheumatic abscess Parvovirus B19 test Pericarditis syphilitic Parapox virus infection Parvovirus B19 test Pericarditis tuberculous positive Parapoxvirus test Perichondritis positive Parvovirus infection Pericoronitis Parasite allergy Pasteurella infection Parasite blood test Perihepatic abscess Pasteurella test positive Parasite blood test Perihepatitis Pathogen resistance positive Perihepatitis gonococcal Peliosis hepatis Parasite cervical Perinatal HBV infection Pelvic abscess specimen test positive Perinatal HIV infection Pelvic infection Parasite DNA test Perineal abscess Parasite DNA test Pelvic inflammatory disease Perineal infection positive Pelvic inflammatory Parasite stool test Perinephric abscess disease mycoplasmal Periodontal destruction Parasite stool test Pelvic sepsis positive Periodontal Parasite tissue Penicillium infection inflammation specimen test positive Penile abscess Periodontitis Parasite urine test Penile infection Periorbital abscess positive Penile wart Periorbital cellulitis Parasitic encephalitis Peptic ulcer helicobacter Periorbital infection Parasitic gastroenteritis Peptostreptococcus Peripheral nerve

infection

ALX0061-C203 – Statistical Analysis Plan – Final 1.0 – 4 OCT 2018

infection


Pharyngoconjunctival

fever of children

abscess

Pharyngolaryngeal


**Periporitis** Pharyngotonsillitis Pneumonia anthrax staphylogenes Phlebitis infective Pneumonia bacterial Perirectal abscess Phlebotomus fever Pneumonia blastomyces Peritoneal abscess Phlebovirus test positive Pneumonia bordetella Peritoneal candidiasis Pneumonia chlamydial Pilonidal cyst Peritoneal chlamvdia Pneumonia cryptococcal Pilonidal cyst congenital infection **Pingueculitis** Pneumonia Peritoneal tuberculosis cytomegaloviral Pinta Peritonitis Pneumonia escherichia Pitted keratolysis Peritonitis bacterial Pneumonia fungal Plague Peritonitis gonococcal Pneumonia Plague sepsis Peritonitis helminthic haemophilus Plasma cell mastitis Peritonitis Pneumonia helminthic Plasmodium falciparum pneumococcal Pneumonia herpes viral infection Peritonitis syphilitic Pneumonia influenzal Plasmodium malariae Peritonitis viral infection Pneumonia klebsiella Peritonsillar abscess Plasmodium ovale Pneumonia legionella Peritonsillitis infection Pneumonia measles Plasmodium vivax Periumbilical abscess Pneumonia moraxella infection Persistent generalised Pneumonia lymphadenopathy Pleural fluid analysis mycoplasmal **Pertussis** Pleural infection Pneumonia necrotising Petrositis Pleural infection Pneumonia bacterial Phaehyphomycosis parainfluenzae viral Pleurisy viral Pharyngeal abscess Pneumonia Pneumococcal pneumococcal Pharyngeal chlamydia bacteraemia infection Pneumonia Pneumococcal infection pseudomonal **Pharyngitis** Pneumococcal sepsis Pneumonia respiratory Pharyngitis bacterial syncytial viral Pneumocystis jirovecii **Pharyngitis** infection Pneumonia salmonella mycoplasmal Pneumocystis jirovecii Pneumonia Pharyngitis pneumonia staphylococcal streptococcal Pneumocystis test Pneumonia

positive

ALX0061-C203 – Statistical Analysis Plan – Final 1.0 – 4 OCT 2018

Pneumonia

Pneumonia adenoviral

streptococcal

Pneumonia toxoplasmal


Pneumonia tularaemia


Pneumonia viral Post viral fatique **Prostatitis** syndrome Pneumonic plague Prostatitis Escherichia Postoperative abscess coli Pneumovirus test positive Postoperative wound Prostatitis gonococcal infection Pogosta disease Prostatitis trichomonal Postoperative wound Polioencephalitis Prostatitis tuberculous infection **Poliomyelitis** Prostatovesiculitis Postpartum sepsis Poliovirus test Proteus infection Potassium hydroxide Poliovirus test positive preparation Proteus test positive Polymerase chain Protozoal corneal ulcer Potassium hydroxide reaction preparation positive Pseudallescheria infection **Polymyositis** Presumed ocular histoplasmosis Polyneuropathy mumps Pseudallescheria sepsis syndrome Polyomavirus test Pseudofolliculitis barbae Primary syphilis positive Pseudomembranous Primary transmission Polyomaviruscolitis associated nephropathy Prion agent test positive Pseudomonal Pontiac fever bacteraemia Proctitis bacterial Porphyromonas Pseudomonal sepsis Proctitis chlamydial infection Pseudomonas Proctitis fungal Porphyromonas test aeruginosa meningitis Proctitis gonococcal positive Pseudomonas **Proctitis herpes** Portal pyaemia bronchitis Proctitis infectious Portal tract inflammation Pseudomonas infection Proctitis monilial Post abortion infection Pseudomonas test Proctitis mycoplasmal positive Post herpetic neuralgia Progressive massive **Psittacosis** Post polio syndrome fibrosis Psoas abscess Post procedural cellulitis Progressive multifocal **Psorospermiasis** Post procedural leukoencephalopathy infection Puerperal infection Progressive vaccinia Post procedural Puerperal pyrexia Propionibacterium pneumonia infection **Pulmonary** Post procedural sepsis echinococciasis Propionibacterium test Post streptococcal positive Pulmonary mycosis

Prostate infection

Prostatic abscess

glomerulonephritis

Post vaccination

autoinoculation

Pulmonary sepsis

Pulmonary syphilis


Pulmonary Rabies Retinitis trichosporonosis Raoultella ornithinolytica Retinitis histoplasma Pulmonary tuberculoma infection Retinitis viral Pulmonary tuberculosis Raoultella test positive Retroperitoneal abscess Pulpitis dental Rash pustular Retroperitoneal infection Punctate keratitis Recrudescent typhus Retroviral infection Puncture site abscess Rectal abscess Retroviral rebound Rectovaginal septum Puncture site discharge syndrome abscess Puncture site infection Reye's syndrome Reiter's syndrome Puncture site oedema Rheumatic fever Relapsing fever Purulence Rheumatic heart Renal abscess disease Purulent discharge Renal cyst infection Rhinitis Purulent pericarditis Renal syphilis Rhinolaryngitis Purulent synovitis Renal tuberculosis Rhinoscleroma **Pyelocystitis** Respiratory moniliasis Rhinosporidiosis **Pyelonephritis** Respiratory papilloma Rhinotracheitis Pyelonephritis acute Respiratory syncytial Rhinovirus infection Pyelonephritis chronic virus bronchiolitis Rhodococcus infection Pyelonephritis fungal Respiratory syncytial Rhodococcus test **Pyelonephritis** virus bronchitis positive mycoplasmal Respiratory syncytial Rickettsialpox Pyelonephritis viral virus infection Rickettsioses not tick Pyloric abscess Respiratory syncytial borne virus test Pvoderma Rickettsiosis Respiratory syncytial Pyoderma streptococcal Rift Valley fever virus test positive Pyometra Rocky mountain spotted Respiratory tract **Pyomyositis** infection fever **Pyonephrosis** Root canal infection Respiratory tract infection bacterial Pyopneumothorax Roseola Respiratory tract Pyospermia Roseolovirus test infection fungal positive Pythium insidiosum Respiratory tract infection

Queensland tick typhus Rubella

positive

infection viral

Respirovirus test

ALX0061-C203 – Statistical Analysis Plan – Final 1.0 – 4 OCT 2018

Pyuria

Q fever


Rotavirus infection

Rotavirus test positive

Rotavirus test


Rubella antibody Secondary syphilis Serratia test positive positive Secondary transmission Severe acute respiratory Rubella antibody test syndrome Seminal vesicular Rubella immunity infection Severe invasive confirmed streptococcal infection Seminal vesiculitis Rubella in pregnancy Sexual transmission of Seminal vesiculitis infection Rubella infection gonococcal neurological Sexually transmitted Sepsis disease Rubivirus test positive Sepsis neonatal Sexually transmitted Rubulavirus test positive Sepsis pasteurella disease carrier Salmonella bacteraemia Sepsis syndrome Shigella infection Salmonella sepsis Septic arthritis Shigella sepsis Salmonella test positive haemophilus Shigella test positive Salmonellosis Septic arthritis neisserial Shunt infection Salpingitis Septic arthritis Sialoadenitis staphylococcal Salpingitis gonococcal Silicotuberculosis Septic arthritis Salpingitis tuberculous streptobacillus Sinobronchitis Salpingo-oophoritis Septic arthritis Sinusitis Sapovirus test positive streptococcal Sinusitis aspergillus Sarcocystis infection Septic embolus Sinusitis bacterial Scarlet fever Septic encephalopathy Sinusitis fungal Scedosporium infection Septic necrosis Skin bacterial infection Schistosoma test Septic phlebitis Skin candida Schistosoma test Septic rash Skin graft infection positive Septic shock Skin infection **Schistosomiasis** Septic vasculitis Skin infection helminthic Schistosomiasis bladder Seroconversion test Slit-lamp tests abnormal Schistosomiasis Seroconversion test cutaneous Slow virus infection positive Schistosomiasis liver Small intestine Serology abnormal gangrene Scrotal abscess Serology positive Smallpox Scrotal gangrene Serology test Snowshoe hare virus Scrotal infection

Scrub typhus

infection

Sebaceous gland

Serratia bacteraemia

Serratia infection

Serratia sepsis

infection

Soft tissue infection


Spermatic cord Staphylococcal parotitis Streptococcal funiculitis endocarditis Staphylococcal Spermatic cord pharyngitis Streptococcal impetigo inflammation Staphylococcal scalded Streptococcal infection Sphingomonas skin syndrome Streptococcal sepsis paucimobilis infection Staphylococcal sepsis Streptococcal urinary Spinal cord abscess Staphylococcal skin tract infection Spinal cord infection infection Streptococcus test Spirillary fever Staphylococcal Streptococcus test toxaemia Spirillum test positive positive Staphylococcus test Spirochaetal infection Strongyloidiasis Staphylococcus test Subacute endocarditis Spleen tuberculosis positive Splenic abscess Subacute sclerosing Stenotrophomonas panencephalitis Splenic candidiasis infection Subarachnoid abscess Splenic infection Stenotrophomonas Subcutaneous abscess sepsis Splenic infection bacterial Stenotrophomonas test Subdiaphragmatic abscess positive Splenic infection fungal Sternitis Subglottic laryngitis Splenic infection helminthic Subperiosteal abscess Stitch abscess Splenic infection viral Stoma site abscess Superinfection Sporotrichosis Stoma site candida Superinfection bacterial Spotted fever rickettsia Stoma site cellulitis Superinfection fungal test positive Stoma site infection Superinfection Sputum culture mycobacterial Stomach granuloma Sputum culture positive Superinfection viral Stomatococcal infection Sputum purulent Suspected transmission Stomatococcus test of an infectious agent St. Louis encephalitis positive via product Staphylococcal abscess Strawberry tongue Sweat gland infection Staphylococcal Streptobacillary fever Sweating fever bacteraemia Streptobacillus infection Sycosis barbae Staphylococcal impetigo Streptobacillus test **Syphilis** Staphylococcal infection positive Syphilis anal Staphylococcal Streptococcal abscess mediastinitis Syphilis genital Streptococcal Staphylococcal bacteraemia Syphilis musculoskeletal

osteomyelitis


Syphilitic endocarditis of Tonsillitis fungal **Trichomoniasis** heart valve intestinal Tonsillitis streptococcal Systemic candida Trichophytic granuloma Tooth abscess Systemic mycosis Trichophytosis Tooth infection **Taeniasis** Trichosporon infection Torulopsis infection Tertiary syphilis Trichostrongyliasis Toxic shock syndrome Testicular abscess Trichuriasis Toxic shock syndrome Tetanus staphylococcal **Trigonitis** Tetanus neonatorum Toxic shock syndrome Tropical eosinophilia streptococcal Thornwaldt disease Tropical infectious **Toxocariasis** disease Thrombophlebitis septic Toxoplasma serology Tropical spastic paresis Thymus abscess Toxoplasma serology Tropical ulcer Thyroglossal cyst positive infection Trypanosoma serology Toxoplasmosis positive Thyroid echinococciasis **Tracheitis** Trypanosomiasis Thyroid gland abscess Tracheitis obstructive Tuberculin test Thyroid tuberculosis Tracheobronchitis Tuberculin test positive Thyroiditis subacute Tracheobronchitis Tuberculoid leprosy Tick-borne fever mycoplasmal Tuberculoma of central Tick-borne viral Tracheobronchitis viral nervous system encephalitis Tracheostomy infection **Tuberculosis** Tinea barbae Tuberculosis bladder Trachoma Tinea blanca Transmission of an **Tuberculosis** Tinea capitis infectious agent via gastrointestinal Tinea cruris product Tuberculosis liver Tinea faciei Transplant abscess Tuberculosis of central Tinea imbricata Trematode infection nervous system Tinea infection Trench fever Tuberculosis of eye Tinea manuum Tuberculosis of Treponema test genitourinary system Tinea nigra Treponema test false

Treponema test positive

**Trichiniasis** 

**Trichomoniasis** 

positive

intrathoracic lymph nodes

Tuberculosis of

Tuberculosis of

peripheral lymph nodes

Tuberculosis ureter

ALX0061-C203 – Statistical Analysis Plan – Final 1.0 – 4 OCT 2018

Tinea pedis

**Tonsillitis** 

Tinea versicolour

Tongue abscess

Tonsillitis bacterial


Tuberculous abscess Ureteritis Uterine abscess central nervous system Urethral abscess Uterine infection **Tuberculous** Urethral carbuncle Uveitis endometritis Urethral stricture post Vaccination site Tuberculous laryngitis infection abscess Tuberculous pleurisy Urethritis Vaccination site cellulitis **Tuberculous** Urethritis chlamydial Vaccination site tenosynovitis discharge Urethritis gonococcal Tubo-ovarian abscess Vaccination site Urethritis mycoplasmal Tularaemia infection Urethritis trichomonal Type 1 lepra reaction Vaccination site pallor Urethritis ureaplasmal Type 2 lepra reaction Vaccination site pustule Urinary bladder abscess Typhoid carrier Vaccine associated Urinary tract abscess paralytic poliomyelitis Typhoid fever Urinary tract infection Vaccine breakthrough **Typhus** infection Urinary tract infection Typhus rickettsia test bacterial Vaccine virus shedding Typhus rickettsia test Urinary tract infection Vaccinia test positive positive enterococcal Vaccinia virus infection Ulcerative keratitis Urinary tract infection Vaginal abscess Umbilical hernia fungal gangrenous Vaginal cellulitis Urinary tract infection Umbilical sepsis neonatal Vaginal infection Upper aerodigestive Urinary tract infection Vaginitis chlamydial tract infection pseudomonal Vaginitis gardnerella Upper respiratory fungal Urinary tract infection Vaginitis viral staphylococcal infection Variant Creutzfeldt-Upper respiratory tract Urinary tract infection Jakob disease infection viral Varicella Upper respiratory tract Urinary tract infection bacterial inflammation Varicella post vaccine Varicella virus test Upper respiratory tract Urogenital infection infection helminthic bacterial Varicella virus test positive Urachal abscess Urogenital infection fungal Varicella zoster gastritis Ureaplasma infection Urogenital Varicella zoster Ureaplasma test trichomoniasis positive oesophagitis Urosepsis Varicella zoster Ureter abscess

pneumonia

Viral myelitis


Vector-borneViral sepsisVulvovaginitistransmission of infectionViral sinusitisstreptococcalVeillonella infectionViral skip infectionVulvovaginitis

Veillonella infection

Viral skin infection

Viral skin infection

Viral skin infection

Viral skin infection

Viral skin infection

Viral skin infection

Virgitiest Waterhouse-

transmission Viral test positive Friderichsen syndrome

Vessel puncture site Viral titre Weil's disease

infection Viral titre decreased West Nile viral infection

Vestibular neuronitisViral titre increasedWhipple's diseaseVestibulitisViral tonsillitisWithdrawal hepatitis

Vibrio test positive Viral tracheitis Wound abscess

Viraemia Viral upper respiratory Wound contamination

Viral cardiomyopathy

Viral corneal ulcer

tract infection

Viral uveitis

Wound infection

Wound infection

Viral diarrhoea Viral vasculitis bacterial

Viral epiglottitis Virologic failure Wound infection fungal

Viral haemorrhagic

Visceral larva migrans

Wound infection helminthic

cystitis Visceral leishmaniasis

Viral hepatitis carrier

Vitreous abscess

Vitreous abscess

Vitritis

Wound infection pseudomonas

Viral infection

Viral labyrinthitis

Wound infection

Vorticella infection

staphylococcal

Viral load Vulval abscess Wound infection viral

Viral load decreased Vulval cellulitis Wound sepsis

Viral load increased Vulvitis Yaws

Viral mastitis

Vulvovaginal candidiasis

Yaws of bone

Viral mutation identified

Vulvovaginal human

papilloma virus infection

Yaws of skin

Viral myocarditis

Vulvovaginal mycotic

Yellow fever vaccine-

Viral myositis infection associated neurotropic

Viral myosius

Vulvovaginal warts

disease

Viral oesophagitis

Vulvovaginitis

Yellow fever vaccine-

Viral parotitis

Vulvovaginitis

Yellow fever vaccineassociated viscerotropic

Viral pericarditis chlamydial disease

Viral pharyngitisVulvovaginitisYersinia bacteraemiaViral rashgonococcalYersinia infectionViral rhinitisVulvovaginitis helminthicYersinia sepsis

Yellow fever




Yersinia test Young's syndrome Zoonotic bacterial

Yersinia test positive Zoonosis infection

#### Serious infections

Any events like this will be listed under cluster = Infections, and can be identified based on AESER = Y

### Opportunistic infections (excluding TB)

Aeromonas infection Candida Cytomegalovirus Aeromonas test positive endophthalmitis chorioretinitis

Allescheriosis Candida osteomyelitis Cytomegalovirus colitis

Alternaria infection Candida pneumonia Cytomegalovirus

Aspergilloma Candida retinitis duodenitis

Candida sepsis

Candida sepsis

Aspergillosis oral enteritis

Aspergillus infection Capnocytophaga Cytomegalovirus

Aspergillus test Capnocytophaga test enterocolitis

Aspergillus test positive positive Cytomegalovirus gastritis

Atypical mycobacterial Cerebral aspergillosis Cytomegalovirus

infection Cerebral fungal infection gastroenteritis

Attraced mycobacterial Cerebral toxoplasmosis Cytomegalovirus

Atypical mycobacterial pneumonia Chronic pulmonary Cytomegalovirus gastrointestinal infection

Atypical mycobacterium histoplasmosis Cytomegalovirus gastrointestinal ulcer

Bacillary angiomatosis encephalitis Cytomegalovirus

Bacillary angiomatosis

Coccidioidomycosis

hepatitis

BK virus infection

Coccidiolidomycosis

Cytomegalovirus

Cottis herpes

Bronchopulmonary infection aspergillosis Cryptococcal cutaneous

Burkholderia cepacia infection Cytomegalovirus mucocutaneous ulcer

complex infection Cryptococcal fungaemia Cytomegalovirus

Burkholderia cepacia Cryptococcosis myelomeningoradiculitis complex sepsis Cryptococcus test Cytomegalovirus

Burkholderia gladioli Cryptococcus test myocarditis infection

Burkholderia infection positive Cytomegalovirus oesophagitis

Burkholderia test coccidioidomycosis Cytomegalovirus positive pancreatitis

Fungal tracheitis

Gastritis fungal

Gastritis herpes

Fusarium infection


Gastroenteritis Herpes zoster Cytomegalovirus pericarditis cryptococcal meningoencephalitis Cytomegalovirus Genital herpes zoster Herpes zoster syndrome meningomyelitis Hepatic candidiasis Cytomegalovirus test Herpes zoster Hepatic infection fungal necrotising retinopathy Cytomegalovirus test Hepatitis toxoplasmal Herpes zoster oticus positive Hepatosplenic Cytomegalovirus urinary Herpes zoster candidiasis tract infection pharyngitis Herpes oesophagitis Cytomegalovirus Histoplasmosis viraemia Herpes sepsis cutaneous Herpes simplex colitis Disseminated Histoplasmosis cryptococcosis disseminated Herpes simplex encephalitis Infection in an Disseminated cytomegaloviral immunocompromised Herpes simplex gastritis infection host Herpes simplex hepatitis Encephalitis JC polyomavirus test Herpes simplex cytomegalovirus JC polyomavirus test meningitis Encephalitis fungal positive Herpes simplex **Endocarditis** JC virus granule cell meningoencephalitis histoplasma neuronopathy Herpes simplex Enterocolitis fungal JC virus infection meningomyelitis Exserohilum infection Kaposi's sarcoma AIDS Herpes simplex related Exserohilum test necrotising retinopathy Kaposi's varicelliform Exserohilum test Herpes simplex eruption oesophagitis positive Listeria encephalitis Eye infection Herpes simplex toxoplasmal pneumonia Listeria sepsis Herpes simplex sepsis Fungaemia Listeria test positive Herpes simplex visceral Lymphadenitis fungal Fungal abscess central nervous system Herpes zoster Meningitis aspergillus Fungal oesophagitis cutaneous disseminated Meningitis candida Fungal retinitis Herpes zoster Meningitis coccidioides disseminated Fungal sepsis Meningitis cryptococcal

Herpes zoster infection

neurological

meningitis

Herpes zoster

Meningitis exserohilum

Meningitis fungal

Meningitis herpes


| Meningitis | histoplasma |
|------------|-------------|

Meningitis listeria

Meningitis toxoplasmal

Meningomyelitis herpes

Methylobacterium

infection

Miliary pneumonia

Mucocutaneous candidiasis

Mucormycosis

Mycobacterium avium complex immune restoration disease

Mycobacterium avium complex infection

Mycobacterium chelonae infection

Mycobacterium fortuitum infection

Mycobacterium kansasii

infection

Myocarditis toxoplasmal

Necrotising herpetic

retinopathy

Neurocryptococcosis

Neutropenic infection

Neutropenic sepsis

Nocardia sepsis

Nocardia test positive

Nocardiosis Oesophageal

candidiasis

Ophthalmic herpes

zoster

Opportunistic infection

Oral candidiasis

Oral fungal infection

Oral hairy leukoplakia

Oro-pharyngeal aspergillosis

Oropharyngeal

candidiasis

Oropharyngitis fungal

Otitis media fungal

Pancreatitis fungal

Penicillium infection

Pericarditis fungal

Pericarditis histoplasma

Phaehyphomycosis

Pneumocystis jirovecii

infection

Pneumocystis jirovecii

pneumonia

Pneumocystis test

positive

Pneumonia cryptococcal

Pneumonia cytomegaloviral

Pneumonia herpes viral

Pneumonia toxoplasmal

Polyomavirus-

associated nephropathy

Presumed ocular histoplasmosis syndrome

Proctitis herpes

Progressive multifocal leukoencephalopathy

Progressive vaccinia

Pseudallescheria

infection

Pseudallescheria sepsis

Pyelonephritis fungal

Respiratory moniliasis

Retinitis histoplasma

Retinitis viral

Rhodococcus infection

Rhodococcus test

positive

Scedosporium infection

Sepsis pasteurella

Sinusitis aspergillus

Sinusitis fungal

Splenic candidiasis

Splenic infection fungal

Stomatococcal infection

Stomatococcus test

positive

Strongyloidiasis

Systemic candida

Systemic mycosis

Tonsillitis fungal

Upper respiratory fungal

infection

Varicella zoster gastritis

Varicella zoster oesophagitis

Varicella zoster pneumonia

Varicella zoster virus

infection

Viral oesophagitis

Yersinia sepsis

Active TB


Adrenal gland Male genital tract Tuberculosis liver tuberculosis tuberculosis Tuberculosis of central Bone tuberculosis Meningitis tuberculous nervous system Choroid tubercles Oesophageal Tuberculosis of eye tuberculosis Congenital tuberculosis Tuberculosis of Pericarditis tuberculous genitourinary system Conjunctivitis tuberculous Peritoneal tuberculosis Tuberculosis of intrathoracic lymph Cutaneous tuberculosis Prostatitis tuberculous nodes Disseminated Pulmonary tuberculoma Tuberculosis of tuberculosis Pulmonary tuberculosis peripheral lymph nodes Ear tuberculosis Renal tuberculosis Tuberculosis ureter Epididymitis tuberculous Salpingitis tuberculous Tuberculous abscess Erythema induratum central nervous system Silicotuberculosis Exposure to Tuberculous Spleen tuberculosis communicable disease endometritis Thyroid tuberculosis Extrapulmonary Tuberculous laryngitis tuberculosis Tuberculoma of central Tuberculous pleurisy nervous system Female genital tract Tuberculous tuberculosis **Tuberculosis** tenosynovitis

### Latent TB

Lymph node tuberculosis

Joint tuberculosis

Latent tuberculosis Mycobacterium Tuberculin test false tuberculosis complex negative Mycobacterium test test positive positive Tuberculin test positive

Tuberculosis bladder

**Tuberculosis** 

gastrointestinal

Herpes zoster infection

Herpes virus infection

Colitis herpes Herpes zoster Herpes zoster meningoencephalitis Gastritis herpes Herpes zoster cutaneous disseminated Herpes zoster Genital herpes zoster meningomyelitis Herpes zoster Herpes oesophagitis disseminated Herpes zoster Herpes ophthalmic necrotising retinopathy Herpes zoster infection Herpes pharyngitis neurological Herpes zoster oticus Herpes sepsis Herpes zoster Herpes zoster meningitis pharyngitis

ALX0061-C203 – Statistical Analysis Plan – Final 1.0 – 4 OCT 2018


Meningitis herpes

Meningomyelitis herpes

Ophthalmic herpes zoster

Pneumonia herpes viral

Proctitis herpes

Varicella zoster gastritis

Varicella zoster oesophagitis

Varicella zoster pneumonia

Varicella zoster virus infection

### **Malignancies**

Malignancies standardized MedDRA query (SMQ) (Narrow)

### Hypersensitivity reactions (including anaphylaxis and angioedema)

Anaphylactic reaction SMQ (Narrow)

Angioedema SMQ (Narrow)

Hypersensitivity SMQ (Narrow)

### Gastrointestinal (GI) perforation

Gastrointestinal perforation SMQ (Narrow)

### **Demyelinating disorders**

Demyelination SMQ (Narrow)

### Major adverse cardiac events (MACE)

Cardiac failure SMQ (Narrow)

Cerebrovascular disorders SMQ (Narrow)

Ischemic heart disease SMQ (Narrow)

# Your Health and Well-Being

This survey asks for your views about your health. This information will help keep track of how you feel and how well you are able to do your usual activities. *Thank you for completing this survey!* 

For each of the following questions, please mark an  $\boxtimes$  in the one box that best describes your answer.

1. In general, would you say your health is:



2. <u>Compared to one week ago</u>, how would you rate your health in general <u>now</u>?

| Much better<br>now than one<br>week ago | Somewhat<br>better<br>now than one<br>week ago | About the same as one week ago | Somewhat<br>worse<br>now than one<br>week ago | Much worse<br>now than one<br>week ago |
|---|---|---|---|---|
| <b>V</b> □ 1 | ₩eek age | <b>▼</b> | ₩CGR ago | |


3. The following questions are about activities you might do during a typical day. Does <u>your health now limit you</u> in these activities? If so, how much?

| | | Yes,<br>limited<br>a lot | Yes,<br>limited<br>a little | No, not limited at all |
|---|---|---|---|---|
| a | <u>Vigorous activities</u> , such as running, lifting heavy objects, participating in strenuous sports | 1 | 2 | 3 |
| b | Moderate activities, such as moving a table, pushing a vacuum cleaner, bowling, or playing golf | 1 | 2 | 3 |
| c | Lifting or carrying groceries | 1 | 2 | 3 |
| d | Climbing several flights of stairs | 1 | 2 | 3 |
| e | Climbing one flight of stairs | 1 | 2 | 3 |
| f | Bending, kneeling, or stooping | 1 | 2 | 3 |
| g | Walking more than a mile | 1 | 2 | 3 |
| h | Walking several hundred yards | 1 | 2 | 3 |
| i | Walking one hundred yards | 1 | 2 | 3 |
| i | Bathing or dressing yourself | | 2 | 3 |


4. During the <u>past week</u>, how much of the time have you had any of the following problems with your work or other regular daily activities <u>as a result of your physical health?</u>

| | | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
|---|---|---|---|---|---|---|
| a | Cut down on the <u>amount of</u> <u>time</u> you spent on work or other activities | 1 | 2 | 3 | 4 | 5 |
| b | Accomplished less than you would like | 1 | 2 | 3 | 4 | 5 |
| c | Were limited in the <u>kind</u> of work or other activities | 1 | 2 | 3 | 4 | 5 |
| d | Had <u>difficulty</u> performing the work or other activities (for example, it took extra effort) | 🗌 1 | 2 | 3 | | 5 |
| 5. | During the <u>past week</u> , ho following problems with <u>result of any emotional panxious</u> )? | your work | or other re | egular daily | activities <u>:</u> | |
| | | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
| a | Cut down on the amount of time you spent on work or other activities | 1 | ···· 2 ···· | 3 | 4 | 5 |
| b | Accomplished less than you would like | 1 | 2 | 3 | 4 | 5 |
| c | Did work or other activities | | | | | |



6. During the <u>past week</u>, to what extent has your physical health or emotional problems interfered with your normal social activities with family, friends, neighbors, or groups?



7. How much bodily pain have you had during the past week?



8. During the <u>past week</u>, how much did <u>pain</u> interfere with your normal work (including both work outside the home and housework)?

| Not at all | A little bit | Moderately | Quite a bit | Extremely |
|------------|--------------|------------|-------------|-----------|
| | 2 | 3 | 4 | 5 |



9. These questions are about how you feel and how things have been with you <u>during the past week</u>. For each question, please give the one answer that comes closest to the way you have been feeling. How much of the time during the <u>past week</u>...

| | | All of the time | Most of the time | Some of the time | A little of the time | None of the time |
|---|---|---|---|---|---|---|
| a | Did you feel full of life? | 1 | 2 | 3 | 4 | 5 |
| b | Have you been very nervous? | 1 | 2 | 3 | 4 | 5 |
| c | Have you felt so down in the dumps that nothing could cheer you up? | 1 | 2 | 3 | 4 | 5 |
| d | Have you felt calm and peaceful? | 1 | 2 | 3 | 4 | 5 |
| e | Did you have a lot of energy? | 1 | 2 | 3 | 4 | 5 |
| f | Have you felt downhearted and depressed? | 1 | 2 | 3 | 4 | 5 |
| g | Did you feel worn out? | 1 | 2 | 3 | 4 | 5 |
| h | Have you been happy? | 1 | 2 | 3 | 4 | 5 |
| i | Did you feel tired? | 1 | 2 | 3 | 4 | 5 |

10. During the <u>past week</u>, how much of the time has your <u>physical health</u> <u>or emotional problems</u> interfered with your social activities (like visiting with friends, relatives, etc.)?

| All of the time | Most of the time | Some of the time | A little of the time | None of the time |
|---|---|---|---|---|
| <b>▼</b> | <b>▼</b> | <b>▼</b> 3 | <b>▼</b> | <b>▼</b> |


### 11. How TRUE or FALSE is each of the following statements for you?

| | | Definitely true | Mostly true | Don't know | Mostly false | Definitely false |
|---|---|---|---|---|---|---|
| a | I seem to get sick a little easier than other people | 1 | 2 | 3 | 4 | 5 |
| b | I am as healthy as<br>anybody I know | 1 | 2 | 3 | 4 | 5 |
| c | I expect my health to get worse | 1 | 2 | 3 | 4 | 5 |
| d | My health is excellent | 1 | 2 | 3 | 4 | 5 |

### Thank you for completing these questions!

SF-36v2 $^{\circ}$  Health Survey  $^{\circ}$  1992, 1996, 2000 Medical Outcomes Trust and QualityMetric Incorporated. All rights reserved. SF-36 $^{\circ}$  is a registered trademark of Medical Outcomes Trust.

(SF-36v2® Health Survey Acute, United States (English))